CLINICAL TRIAL: NCT03231943
Title: A Double-Blind (Sponsor Unblinded), Randomized, Placebo-Controlled, Single and Repeated Dose Escalation Study to Investigate the Safety, Tolerability and Pharmacokinetics of GSK3640254 in Healthy Participants
Brief Title: GSK3640254 First Time in Human (FTIH) Study in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 207187; 2017-001367-21 (EudraCT Number)
Record Dates: First submitted 2017-07-24; First posted 2017-07-27 (Actual); Results first posted 2019-10-18 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-05

CONDITIONS: Infection, Human Immunodeficiency Virus; HIV Infections
Keywords: FTIH; Healthy; Tolerability; Dose-escalation; HIV-1; Safety; PK; GSK3640254; Maturation inhibitor
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome; HIV Infections | interventions — GSK3640254

STUDY DESIGN:
Intervention Model Description: This is a dose-escalation study and dose will be escalated based on the safety data of the initial dose.
Who Masked: Participant, Investigator
Masking Description: This will be a double-blind study with subjects and the site-staff blinded and sponsor unblinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Subjects in cohort 1-2: Part 1 (Experimental): Eligible subjects will participate in cohort 1 or 2 and each of these two cohorts will contain up to four escalating doses of GSK3640254. In each cohort, 6 subjects will be randomized to receive single oral dose of GSK3640254 and 2 subjects will be randomized to receive placebo. Hence, each subject in cohort 1 and 2 will receive up to 3 escalating doses of GSK3640254 and one placebo in crossover manner.
  Interventions: Drug: GSK3640254; Drug: Placebo
- GSK3640254 receivers (cohort 3-6 and expansion): Part 2 (Experimental): Eligible subjects will participate in one of the 4 cohorts (3,4,5,6). In each cohort, 6 subjects will be randomized to receive a once-daily oral dose of GSK3640254 for 14 days. After the safety data of cohort 3-6 is available, 18 eligible subjects will be randomized to receive once daily oral dose of GSK3640254 for 14 days in expansion cohort.
  Interventions: Drug: GSK3640254
- Subjects receiving placebo (cohort 3-6): Part 2 (Placebo Comparator): Eligible subjects will participate in one of the 4 cohorts (3,4,5,6). In each cohort, 2 subjects will be randomized to receive a once-daily oral dose of placebo for 14 days. After the safety data of cohort 3-6 is available, 6 eligible subjects will be randomized to receive once daily oral dose of placebo for 14 days in expansion cohort.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK3640254 — GSK3640254 is a capsule available in 1 milligram (mg), 10 mg and 100 mg dosing strength. GSK3640254 capsule will be given via oral route during each dosing day with approximately 240 mL of water.
  Arms: GSK3640254 receivers (cohort 3-6 and expansion): Part 2; Subjects in cohort 1-2: Part 1
Drug: Placebo — Placebo capsule matching to the study treatment will be given via oral route during each dosing day with approximately 240 mL of water.
  Arms: Subjects in cohort 1-2: Part 1; Subjects receiving placebo (cohort 3-6): Part 2

SUMMARY:
Human immuno deficiency virus 1 (HIV-1) infections continues to be a serious health threat throughout the world and development of medicines with new mechanism of action have an important role to play. GSK3640254 is a maturation inhibitor (MI) and can be effective in HIV-1 treatment. This randomized, 2-part, single and repeat increasing dose study will collect information on safety, tolerability and drug levels in the body of in healthy subjects for GSK3640254. The information collected in this study will help in further clinical development of GSK3640254, including a Phase IIA Proof of Concept (PoC) study in HIV-infected subjects. Approximately 16 healthy subjects will be randomized to receive single oral dose of GSK3640254 and placebo in Part 1 and approximately 56 healthy subjects will be randomized to receive repeat oral dose of GSK3640254 or placebo in Part 2. All doses will be given immediately after a moderate fat meal. Maximum duration of study participation will be approximately 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 18 to 55 years of age inclusive, at the time of signing the informed consent.
* Subjects who are overtly healthy as determined by medical evaluation including medical history and psychiatric history, physical examination, laboratory tests, and 24 hour Holter monitoring.
* Body weight >=50.0 kilogram (kg) (110 pounds) for men and 45.0kg (99 pounds) for women and body mass index (BMI) within the range 18.5-32.0 kg per meter square (kg/m^2) (inclusive).
* Male or female subjects. A male subject must agree to use contraception during the treatment period and for at least 14 weeks following the last dose, corresponding to the time needed to eliminate study treatment for potential genotoxic and teratogenic study treatments plus an additional 90 days (spermatogenesis cycle). In addition, male subjects must refrain from donating sperm during this period. A female subject is eligible to participate if she is not a woman of childbearing potential (WOCBP).
* Capable of giving signed informed consent.

Exclusion Criteria:

* Alanine transaminase (ALT) >1.5 into upper limit of normal (ULN).
* Bilirubin >1.5 into ULN (isolated bilirubin >1.5 into ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities.
* Pre-existing clinically relevant, in the opinion of the primary investigator (PI), gastro-intestinal pathology or diagnosis - example irritable bowel syndrome, inflammatory bowel disease, and/or significant Baseline signs and symptoms.
* Medical history of cardiac arrhythmias or cardiac disease or a family or personal history of long QT syndrome.
* Any known or suspected pre-existing psychiatric condition.
* Any other clinical condition (including but not limited to active substance use) or prior therapy that, in the opinion of the Investigator, would make the subject unsuitable for the study; unable to comply with dosing requirements; or unable to comply with study visits; or a condition that could affect the absorption, distribution, metabolism or excretion of the drug.
* Unable to refrain from the use of prescription or non-prescription drugs (with the exception of paracetamol), including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication and for the duration of the study, unless in the opinion of the Investigator and ViiV Healthcare Sponsor and medical monitor, the medication will not interfere with the study medications, procedures, or compromise subject safety.
* Unwillingness to abstain from ingestion of any food or drink containing grapefruit and grapefruit juice, Seville oranges, blood oranges, or pomelos within 7 days prior to the first dose of study treatment(s) or until the end of the study.
* Participation in another concurrent clinical study or prior clinical study (with the exception of imaging trials) prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Where participation in the study would result in donation of blood or blood products in excess of 500 milliliter (mL) within 56 days.
* Presence of hepatitis B surface antigen (HBsAg), or positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment.
* A positive pre-study drug/alcohol screen.
* A positive test for a diagnostic HIV-1 polymerase chain reaction (PCR).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Exclusion criteria for screening ECG: Heart rate <45 or >100 beats per minute (bpm) for males and <50 or >100 bpm for females; PR interval <120 or >220 millisecond (msec); QRS duration <70 or >120 msec; the Fridericia's QT correction formula (QTcF) interval >450 msec.
* Evidence of previous myocardial infarction (does not include ST segment changes associated with re-polarization).
* Any conduction abnormality (including but not specific to left or right complete bundle branch block, Atrioventricular block [2nd degree or higher], Wolff-Parkinson-White [WPW] syndrome).
* Sinus Pauses >3 seconds.
* Any significant arrhythmia which, in the opinion of the Investigator or GlaxoSmithKline/ViiV medical monitor, will interfere with the safety for the individual subject.
* Non-sustained or sustained ventricular tachycardia (3 consecutive ventricular ectopic beats).
* History of regular alcohol consumption within 6 months of the study defined as: an average weekly intake of >14 units. One unit is equivalent to 8 gram of alcohol: a half-pint approximately 240 mL of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* Regular use of tobacco- or nicotine-containing products within 3 months prior to screening.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the Investigator or medical monitor, contraindicates their participation.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2017-09-19 (Actual); Primary Completion 2018-09-09 (Actual); Study Completion 2018-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study is available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (copy the URL below to your browser)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20826

REFERENCES:
- [Background] Joshi SR, Fernando D, Igwe S, McKenzie L, Krishnatry AS, Halliday F, Zhan J, Greene TJ, Xu J, Ferron-Brady G, Lataillade M, Min S. Phase I evaluation of the safety, tolerability, and pharmacokinetics of GSK3640254, a next-generation HIV-1 maturation inhibitor. Pharmacol Res Perspect. 2020 Dec;8(6):e00671. doi: 10.1002/prp2.671. PMID 33200887

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted to evaluate safety, tolerability and pharmacokinetic (PK) of GSK3640254 in healthy participants at one center in United Kingdom from 19-September-2017 to 09-September-2018
Pre-assignment Details: Total 78 participants were enrolled in the study. This was a two part study, Part 1 was single ascending dose (SAD) and Part 2 was multiple ascending dose (MAD).
Groups:
- Part 1: Placebo Followed by GSK3640254 10mg/100mg/400mg: Participants received single dose placebo followed by GSK3640254 10 milligram (mg) followed by GSK3640254 100 mg followed by GSK3640254 400 mg oral dose on Day 1
- Part 1: GSK3640254 1mg/ Placebo /100 mg/400 mg: Participants received single dose GSK3640254 1mg followed by placebo followed by GSK3640254 100 mg followed by GSK3640254 400 mg oral dose on Day 1
- Part 1: GSK3640254 1mg/10mg/Placebo /400mg: Participants received single dose GSK3640254 1mg followed by GSK3640254 10 mg followed by placebo followed by GSK3640254 400 mg oral dose on Day 1
- Part 1: GSK3640254 1mg/10mg/100mg/Placebo: Participants received single dose GSK3640254 1mg followed by GSK3640254 10 mg followed by GSK3640254 100 mg followed by placebo as oral dose on Day 1
- Part 1: Placebo/ GSK3640254 30mg/200 mg/700 mg: Participants received single dose placebo followed by GSK3640254 30mg followed by GSK3640254 200 mg followed by GSK3640254 700 mg as oral dose on Day 1
- Part1:GSK3640254 3mg/Placebo/200mg/700mg: Participants received single dose GSK3640254 3mg followed by placebo followed by GSK3640254 200 mg followed by GSK3640254 700 mg as oral dose on Day 1
- Part 1:GSK3640254 3mg/30mg/Placebo/GSK3640254 700mg: Participants received single dose GSK3640254 3 mg followed by GSK3640254 30 mg followed by placebo followed by GSK3640254 700 mg as oral dose on Day 1
- Part 1:GSK3640254 3mg/30mg/GSK3640254 200mg/Placebo: Participants received single dose GSK3640254 3mg followed by GSK3640254 30mg followed by GSK3640254 200mg followed by placebo as oral dose on Day 1
- Part 2: Repeated Dose GSK3640254 50 mg: Participants received repeated dose of GSK3640254 50 mg once daily up to 14 days
- Part 2: Repeated Dose GSK3640254 100mg: Participants received repeated dose of GSK3640254 100 mg once daily up to 14 days
- Part 2: GSK3640254 200mg + Expansion: Participants received repeated dose of GSK3640254 200 mg once daily up to 14 days
- Part 2: Repeated Dose GSK3640254 320mg: Participants received repeated dose of GSK3640254 320 mg once daily up to 14 days
- Part 2: Repeated Dose Placebo: Participants received repeated dose of matching placebo once daily up to 14 days
Period: Part 1, Period 1 (up to Day 15)
Arm/Group | Part 1: Placebo Followed by GSK3640254 10mg/100mg/400mg | Part 1: GSK3640254 1mg/ Placebo /100 mg/400 mg | Part 1: GSK3640254 1mg/10mg/Placebo /400mg | Part 1: GSK3640254 1mg/10mg/100mg/Placebo | Part 1: Placebo/ GSK3640254 30mg/200 mg/700 mg | Part1:GSK3640254 3mg/Placebo/200mg/700mg | Part 1:GSK3640254 3mg/30mg/Placebo/GSK3640254 700mg | Part 1:GSK3640254 3mg/30mg/GSK3640254 200mg/Placebo | Part 2: Repeated Dose GSK3640254 50 mg | Part 2: Repeated Dose GSK3640254 100mg | Part 2: GSK3640254 200mg + Expansion | Part 2: Repeated Dose GSK3640254 320mg | Part 2: Repeated Dose Placebo
Started | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1, Period 2 (up to Day 30)
Arm/Group | Part 1: Placebo Followed by GSK3640254 10mg/100mg/400mg | Part 1: GSK3640254 1mg/ Placebo /100 mg/400 mg | Part 1: GSK3640254 1mg/10mg/Placebo /400mg | Part 1: GSK3640254 1mg/10mg/100mg/Placebo | Part 1: Placebo/ GSK3640254 30mg/200 mg/700 mg | Part1:GSK3640254 3mg/Placebo/200mg/700mg | Part 1:GSK3640254 3mg/30mg/Placebo/GSK3640254 700mg | Part 1:GSK3640254 3mg/30mg/GSK3640254 200mg/Placebo | Part 2: Repeated Dose GSK3640254 50 mg | Part 2: Repeated Dose GSK3640254 100mg | Part 2: GSK3640254 200mg + Expansion | Part 2: Repeated Dose GSK3640254 320mg | Part 2: Repeated Dose Placebo
Started | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 0 (Two participants withdrawn were replaced) | 1 (One participant withdrawn was replaced) | 2 | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1, Period 3 (up to Day 45)
Arm/Group | Part 1: Placebo Followed by GSK3640254 10mg/100mg/400mg | Part 1: GSK3640254 1mg/ Placebo /100 mg/400 mg | Part 1: GSK3640254 1mg/10mg/Placebo /400mg | Part 1: GSK3640254 1mg/10mg/100mg/Placebo | Part 1: Placebo/ GSK3640254 30mg/200 mg/700 mg | Part1:GSK3640254 3mg/Placebo/200mg/700mg | Part 1:GSK3640254 3mg/30mg/Placebo/GSK3640254 700mg | Part 1:GSK3640254 3mg/30mg/GSK3640254 200mg/Placebo | Part 2: Repeated Dose GSK3640254 50 mg | Part 2: Repeated Dose GSK3640254 100mg | Part 2: GSK3640254 200mg + Expansion | Part 2: Repeated Dose GSK3640254 320mg | Part 2: Repeated Dose Placebo
Started | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Completed | 1 (One participant withdrawn was replaced) | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1 Period 4 (up to Day 60)
Arm/Group | Part 1: Placebo Followed by GSK3640254 10mg/100mg/400mg | Part 1: GSK3640254 1mg/ Placebo /100 mg/400 mg | Part 1: GSK3640254 1mg/10mg/Placebo /400mg | Part 1: GSK3640254 1mg/10mg/100mg/Placebo | Part 1: Placebo/ GSK3640254 30mg/200 mg/700 mg | Part1:GSK3640254 3mg/Placebo/200mg/700mg | Part 1:GSK3640254 3mg/30mg/Placebo/GSK3640254 700mg | Part 1:GSK3640254 3mg/30mg/GSK3640254 200mg/Placebo | Part 2: Repeated Dose GSK3640254 50 mg | Part 2: Repeated Dose GSK3640254 100mg | Part 2: GSK3640254 200mg + Expansion | Part 2: Repeated Dose GSK3640254 320mg | Part 2: Repeated Dose Placebo
Started | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2
Arm/Group | Part 1: Placebo Followed by GSK3640254 10mg/100mg/400mg | Part 1: GSK3640254 1mg/ Placebo /100 mg/400 mg | Part 1: GSK3640254 1mg/10mg/Placebo /400mg | Part 1: GSK3640254 1mg/10mg/100mg/Placebo | Part 1: Placebo/ GSK3640254 30mg/200 mg/700 mg | Part1:GSK3640254 3mg/Placebo/200mg/700mg | Part 1:GSK3640254 3mg/30mg/Placebo/GSK3640254 700mg | Part 1:GSK3640254 3mg/30mg/GSK3640254 200mg/Placebo | Part 2: Repeated Dose GSK3640254 50 mg | Part 2: Repeated Dose GSK3640254 100mg | Part 2: GSK3640254 200mg + Expansion | Part 2: Repeated Dose GSK3640254 320mg | Part 2: Repeated Dose Placebo
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 25 | 7 | 14
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 24 | 6 | 14
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part 1: Cohort 1: Participants received GSK3640254 1mg, GSK3640254 10 mg, GSK3640254 100mg, GSK3640254 400mg as ascending single dose on Day 1 of each period, each participant received placebo in one of the four periods
- Part 1: Cohort 2: Participants received GSK3640254 3mg, GSK3640254 30 mg, GSK3640254 200mg, GSK3640254 700mg as ascending single dose on Day 1 of each period, each participant received placebo in one of the four periods
- Part 2: Repeated Dose GSK3640254 100 mg: Participants received repeated dose of GSK3640254 100 mg once daily up to 14 days
- Part 2: Repeated Dose GSK3640254 200 mg + Expansion: Participants received repeated dose of GSK3640254 200 mg once daily up to 14 days
- Part 2: Repeated Dose GSK3640254 320 mg: Participants received repeated dose of GSK3640254 320 mg once daily up to 14 days
- Total: Total of all reporting groups
Arm/Group | Part 1: Cohort 1 | Part 1: Cohort 2 | Part 2: Repeated Dose GSK3640254 50 mg | Part 2: Repeated Dose GSK3640254 100 mg | Part 2: Repeated Dose GSK3640254 200 mg + Expansion | Part 2: Repeated Dose GSK3640254 320 mg | Part 2: Repeated Dose Placebo | Total
Number analyzed (Participants) | 12 | 8 | 6 | 6 | 25 | 7 | 14 | 78
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 12 | 8 | 6 | 6 | 25 | 7 | 14 | 78
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 12 | 8 | 6 | 6 | 25 | 7 | 14 | 78
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  ASIAN - CENTRAL/SOUTH ASIAN HERITAGE | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 3
  BLACK OR AFRICAN AMERICAN | 1 | 1 | 1 | 1 | 4 | 0 | 2 | 10
  WHITE-WHITE/CAUCASIAN/EUROPEAN HERITAGE | 9 | 6 | 5 | 5 | 20 | 5 | 11 | 61
  MULTIPLE | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  ASIAN - EAST ASIAN HERITAGE | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  ASIAN - SOUTH EAST ASIAN HERITAGE | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  WHITE - ARABIC/NORTH AFRICAN HERITAGE | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Part 1:Number of Participants With Adverse Events (AEs) and Serious AEs (SAEs)
Description: An AE is any untoward medical occurrence in a subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect or any other situation according to medical or scientific judgment will be categorized as SAE. Results are presented treatment wise.
Time Frame: Up to Day 15
Population: Safety Population. It is comprised of all participants who received at least one dose of a study treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1: GSK3640254 1 mg: Participants received single dose of GSK3640254 1 mg following a moderate fat meal on Day 1
- Part 1: GSK3640254 3 mg: Participants received single dose of GSK3640254 3 mg following a moderate fat meal on Day 1
- Part 1: GSK3640254 10 mg: Participants received single dose of GSK3640254 10 mg following a moderate fat meal on Day 1
- Part 1: GSK3640254 30mg: Participants received single dose of GSK3640254 30 mg following a moderate fat meal on Day 1
- Part 1: GSK3640254 100 mg: Participants received single dose of GSK3640254 100 mg following a moderate fat meal on Day 1
- Part 1: GSK3640254 200 mg: Participants received single dose of GSK3640254 200 mg following a moderate fat meal on Day 1
- Part 1: GSK3640254 400 mg: Participants received single dose of GSK3640254 400 mg following a moderate fat meal on Day 1
- Part 1: GSK3640254 700 mg: Participants received single dose of GSK3640254 700 mg following a moderate fat meal on Day 1
- Part 1: Single Dose Placebo: Participants received single dose of matching placebo following a moderate fat meal on Day 1
Arm/Group | Part 1: GSK3640254 1 mg | Part 1: GSK3640254 3 mg | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 30mg | Part 1: GSK3640254 100 mg | Part 1: GSK3640254 200 mg | Part 1: GSK3640254 400 mg | Part 1: GSK3640254 700 mg | Part 1: Single Dose Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16
Participants
  AE | 3 | 2 | 4 | 3 | 3 | 4 | 4 | 1 | 7
  SAE | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Part 1: Change From Baseline in Hematology Parameters: Basophils, Eosinophils, Leukocytes, Lymphocytes, Monocytes, Neutrophils, Platelets.
Description: Blood samples were collected to analyze the hematology parameters: basophils, eosinophils, leukocytes, lymphocytes, monocytes, neutrophils and platelets. Day -2 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value. Results are presented treatment wise.
Time Frame: Baseline (Day -2), 24 hours, 48 hours, 96 hours and Follow up (Day 15)
Population: Safety Population. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Measure: Mean (Standard Deviation); unit: 10^9 cells /Liter
Arm/Group | Part 1: GSK3640254 1 mg | Part 1: GSK3640254 3 mg | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 30mg | Part 1: GSK3640254 100 mg | Part 1: GSK3640254 200 mg | Part 1: GSK3640254 400 mg | Part 1: GSK3640254 700 mg | Part 1: Single Dose Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16
10^9 cells /Liter
  Basophils, 24 hours, n=6,6,6,6,6,6,5,6,16: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 6 | 16
  Basophils, 24 hours, n=6,6,6,6,6,6,5,6,16 | -0.002 (0.0075) | -0.002 (0.0147) | 0.005 (0.0084) | -0.002 (0.0075) | -0.007 (0.0103) | 0.002 (0.0098) | -0.002 (0.0148) | -0.007 (0.0121) | 0.001 (0.0106)
  Basophils, 48 hours, n=6,6,5,6,6,6,6,6,16: number analyzed (Participants) | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 16
  Basophils, 48 hours, n=6,6,5,6,6,6,6,6,16 | -0.002 (0.0098) | 0.012 (0.0117) | 0.010 (0.0187) | -0.007 (0.0103) | -0.005 (0.00550) | 0.007 (0.0082) | 0.000 (0.0167) | 0.000 (0.0110) | 0.005 (0.0115)
  Basophils, 96 hours, n=6,6,6,6,6,6,6,6,15: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 15
  Basophils, 96 hours, n=6,6,6,6,6,6,6,6,15 | 0.003 (0.0103) | 0.000 (0.0155) | -0.003 (0.0103) | -0.002 (0.0147) | -0.005 (0.0152) | 0.002 (0.0098) | -0.007 (0.0052) | -0.002 (0.0147) | 0.004 (0.0118)
  Basophils, Day 15,n=6,6,6,6,6,6,6,6,16 | 0.002 (0.0133) | 0.012 (0.0117) | 0.000 (0.0110) | 0.002 (0.0098) | -0.007 (0.0082) | 0.010 (0.0063) | -0.005 (0.0207) | -0.005 (0.0084) | 0.007 (0.0178)
  Eosinophils, 24 hours, n=6,6,6,6,6,6,5,6,16: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 6 | 16
  Eosinophils, 24 hours, n=6,6,6,6,6,6,5,6,16 | -0.022 (0.1876) | 0.012 (0.0376) | 0.005 (0.0650) | 0.015 (0.0489) | 0.008 (0.0508) | -0.017 (0.0186) | -0.032 (0.0642) | 0.023 (0.0266) | 0.005 (0.0648)
  Eosinophils, 48 hour, 6,6,5,6,6,6,6,6,16: number analyzed (Participants) | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 16
  Eosinophils, 48 hour, 6,6,5,6,6,6,6,6,16 | -0.032 (0.1982) | 0.018 (0.0731) | 0.008 (0.0497) | 0.010 (0.0544) | 0.010 (0.0544) | 0.020 (0.0346) | -0.030 (0.0443) | 0.012 (0.0796) | 0.037 (0.0266)
  Eosinophils, 96 hours, n=6,6,6,6,6,6,6,6,15: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 15
  Eosinophils, 96 hours, n=6,6,6,6,6,6,6,6,15 | -0.052 (0.1970) | 0.035 (0.0575) | -0.012 (0.0591) | 0.003 (0.0602) | 0.013 (0.0207) | -0.018 (0.0382) | 0.028 (0.0861) | 0.022 (0.0256) | 0.013 (0.0656)
  Eosinophils, FU (Day 15), n=6,6,6,6,6,6,6,6,16 | -0.023 (0.1328) | 0.012 (0.0534) | 0.000 (0.0335) | 0.020 (0.0921) | 0.018 (0.0542) | 0.012 (0.0471) | -0.032 (0.0960) | -0.012 (0.0354) | -0.015 (0.0791)
  Leukocytes, 24 hours, n=6,6,6,6,6,6,5,6,16: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 6 | 16
  Leukocytes, 24 hours, n=6,6,6,6,6,6,5,6,16 | 0.592 (0.9839) | 0.877 (0.7228) | -0.910 (1.1691) | 0.058 (0.8437) | 0.132 (0.8528) | -0.742 (2.2552) | -0.088 (0.4219) | 0.078 (0.6916) | 0.079 (0.8700)
  Leukocytes, 48 hours, n=6,6,5,6,6,6,6,6,16: number analyzed (Participants) | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 16
  Leukocytes, 48 hours, n=6,6,5,6,6,6,6,6,16 | 0.603 (1.3012) | 0.388 (0.8506) | -0.878 (1.2611) | -0.292 (0.9476) | 0.307 (1.1555) | -0.673 (1.8656) | 1.220 (2.6559) | 0.312 (0.6725) | 0.104 (0.8442)
  Leukocytes 96 hours, n=6,6,6,6,6,6,6,6,15: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 15
  Leukocytes 96 hours, n=6,6,6,6,6,6,6,6,15 | 0.693 (1.1514) | 0.953 (0.8659) | -0.897 (0.9192) | -0.107 (0.9821) | 0.503 (1.1885) | -0.458 (2.3501) | 0.390 (1.3833) | 0.557 (0.5838) | 0.272 (0.8542)
  Leukocytes, FU (Day 15), n=6,6,6,6,6,6,6,6,16 | 0.348 (1.0652) | 0.502 (1.2216) | -0.113 (1.8444) | -0.007 (1.0958) | 0.292 (0.6240) | -0.835 (1.6488) | -0.142 (1.5163) | 0.327 (0.9991) | -0.111 (0.7964)
  Lymphocytes, 24 hours, n=6,6,6,6,6,6,5,6,16: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 6 | 16
  Lymphocytes, 24 hours, n=6,6,6,6,6,6,5,6,16 | 0.073 (0.3189) | 0.243 (0.1888) | -0.248 (0.3124) | -0.140 (0.2305) | -0.188 (0.3172) | -0.158 (0.1659) | -0.124 (0.0727) | -0.005 (0.2375) | 0.027 (0.2972)
  Lymphocytes, 48 hours, n=6,6,5,6,6,6,6,6,16: number analyzed (Participants) | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 16
  Lymphocytes, 48 hours, n=6,6,5,6,6,6,6,6,16 | 0.082 (0.3344) | 0.320 (0.2909) | -0.244 (0.4865) | -0.238 (0.2739) | -0.050 (0.2748) | -0.110 (0.2873) | -0.303 (0.4113) | 0.082 (0.2490) | 0.164 (0.3759)
  Lymphocytes, 96 hours, n=6,6,6,6,6,6,6,6,15: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 15
  Lymphocytes, 96 hours, n=6,6,6,6,6,6,6,6,15 | 0.142 (0.2643) | 0.207 (0.2388) | -0.215 (0.3661) | -0.035 (0.1747) | 0.000 (0.3509) | -0.143 (0.1766) | -0.093 (0.3449) | 0.285 (0.2741) | 0.181 (0.4474)
  Lymphocytes, FU (Day 15), n=6,6,6,6,6,6,6,6,16 | -0.027 (0.4607) | 0.082 (0.2491) | -0.165 (0.6984) | -0.012 (0.4303) | -0.067 (0.4020) | -0.097 (0.4866) | -0.232 (0.3513) | -0.130 (0.3107) | 0.005 (0.3483)
  Monocytes, 24 hours, n=6,6,6,6,6,6,5,6,16: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 6 | 16
  Monocytes, 24 hours, n=6,6,6,6,6,6,5,6,16 | 0.017 (0.0755) | 0.040 (0.0846) | -0.107 (0.1405) | -0.045 (0.0505) | -0.022 (0.1342) | 0.068 (0.2099) | -0.042 (0.1252) | 0.028 (0.0643) | -0.014 (0.0870)
  Monocytes, 48 hours, 6,6,5,6,6,6,6,6,16: number analyzed (Participants) | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 16
  Monocytes, 48 hours, 6,6,5,6,6,6,6,6,16 | 0.048 (0.1052) | 0.043 (0.1198) | -0.104 (0.1146) | -0.050 (0.0885) | -0.002 (0.0854) | 0.083 (0.1533) | 0.083 (0.2224) | 0.037 (0.0441) | 0.002 (0.0795)
  Monocytes, 96 hours, n=6,6,6,6,6,6,6,6,15: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 15
  Monocytes, 96 hours, n=6,6,6,6,6,6,6,6,15 | 0.015 (0.1266) | 0.082 (0.1219) | -0.090 (0.1307) | -0.047 (0.0579) | -0.018 (0.1184) | 0.078 (0.1242) | 0.020 (0.1655) | 0.033 (0.0572) | 0.020 (0.0890)
  Monocytes,FU (Day 15), n= 6,6,6,6,6,6,6,6,16 | -0.003 (0.0771) | 0.048 (0.0826) | -0.022 (0.1309) | 0.020 (0.1619) | 0.045 (0.0896) | 0.115 (0.0789) | 0.008 (0.1439) | -0.003 (0.0855) | -0.002 (0.0878)
  Neutrophils, 24 hours, n=6,6,6,6,6,6,5,6,16: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 6 | 16
  Neutrophils, 24 hours, n=6,6,6,6,6,6,5,6,16 | 0.528 (0.5383) | 0.583 (0.6552) | -0.562 (0.7714) | 0.230 (0.8517) | 0.342 (0.4796) | -0.500 (2.0326) | 0.110 (0.2985) | 0.035 (0.6405) | 0.059 (0.7913)
  Neutrophils, 48 hours, n=6,6,5,6,6,6,6,6,16: number analyzed (Participants) | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 16
  Neutrophils, 48 hours, n=6,6,5,6,6,6,6,6,16 | 0.507 (0.8878) | -0.003 (0.5852) | -0.546 (0.6919) | -0.007 (0.9485) | 0.342 (0.9186) | -0.455 (1.6850) | 1.425 (2.7042) | 0.153 (0.5704) | -0.085 (0.7056)
  Neutrophils, 96 hours, n=6,6,6,6,6,6,6,6,15: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 15
  Neutrophils, 96 hours, n=6,6,6,6,6,6,6,6,15 | 0.587 (0.7991) | 0.628 (0.6082) | -0.575 (0.6277) | -0.027 (0.9432) | 0.513 (0.9082) | -0.218 (2.3225) | 0.440 (1.1395) | 0.218 (0.4922) | 0.055 (0.6401)
  Neutrophils, FU (Day 15), n= 6,6,6,6,6,6,6,6,16 | 0.398 (0.6349) | 0.345 (0.9399) | 0.077 (1.0609) | -0.037 (0.9710) | 0.302 (0.6797) | -0.643 (1.4316) | 0.120 (1.1397) | 0.475 (0.7676) | -0.107 (0.7009)
  Platelets, 24 hours, n=6,6,6,6,6,6,5,6,16: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 6 | 16
  Platelets, 24 hours, n=6,6,6,6,6,6,5,6,16 | -0.3 (11.40) | 9.7 (30.29) | -8.5 (16.11) | -17.5 (27.90) | -2.8 (14.48) | 7.2 (9.54) | -9.0 (37.33) | -1.7 (31.17) | -3.3 (34.99)
  Platelets, 48 hours, n=6,6,5,6,6,6,6,6,16: number analyzed (Participants) | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 16
  Platelets, 48 hours, n=6,6,5,6,6,6,6,6,16 | -1.5 (15.95) | -3.2 (17.33) | -11.0 (21.13) | -1.7 (13.08) | 0.7 (14.98) | 9.5 (11.64) | -14.7 (36.62) | -2.8 (18.97) | 0.8 (22.54)
  Platelets, 96 hours, n=6,6,6,6,6,6,6,6,15: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 15
  Platelets, 96 hours, n=6,6,6,6,6,6,6,6,15 | -8.2 (15.75) | 7.3 (14.65) | -6.8 (14.99) | 1.3 (17.29) | 2.3 (24.57) | 6.7 (15.02) | -13.2 (44.37) | 0.3 (24.34) | -1.7 (22.98)
  Platelets, FU (Day 15), n=6,6,6,6,6,6,6,6,16 | -10.4 (21.59) | 19.2 (14.66) | -16.7 (36.59) | 13.0 (15.85) | 6.5 (22.64) | 13.0 (29.48) | -13.0 (48.17) | -4.0 (18.64) | -1.6 (32.94)

3. Primary Outcome: Part 1: Change From Baseline in Hematology Parameters: Erythrocytes.
Description: Blood samples were collected to analyze the hematology parameters: erythrocytes. Day -2 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.Results are presented treatment wise.
Time Frame: Baseline (Day -2), 24 hours, 48 hours, 96 hours and Follow up (Day 15)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 10^12 cells/Liter
Arm/Group | Part 1: GSK3640254 1 mg | Part 1: GSK3640254 3 mg | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 30mg | Part 1: GSK3640254 100 mg | Part 1: GSK3640254 200 mg | Part 1: GSK3640254 400 mg | Part 1: GSK3640254 700 mg | Part 1: Single Dose Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16
10^12 cells/Liter
  24 hours, n=6,6,6,6,6,6,5,6,16: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 6 | 16
  24 hours, n=6,6,6,6,6,6,5,6,16 | 0.118 (0.2576) | 0.338 (0.1150) | -0.005 (0.1747) | 0.147 (0.2925) | 0.212 (0.2335) | 0.198 (0.0933) | 0.084 (0.1928) | 0.302 (0.1447) | 0.197 (0.2148)
  48 hours, n=6,6,5,6,6,6,6,6,16: number analyzed (Participants) | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 16
  48 hours, n=6,6,5,6,6,6,6,6,16 | 0.162 (0.2899) | 0.142 (0.1607) | -0.024 (0.2501) | 0.108 (0.3252) | 0.152 (0.1528) | 0.288 (0.1082) | 0.087 (0.2295) | 0.180 (0.2440) | 0.171 (0.2112)
  96 hours, n=6,6,6,6,6,6,6,6,15: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 15
  96 hours, n=6,6,6,6,6,6,6,6,15 | 0.155 (0.2290) | 0.202 (0.1683) | 0.083 (0.2499) | 0.178 (0.2320) | -0.035 (0.2672) | 0.112 (0.0674) | 0.062 (0.2528) | 0.237 (0.2530) | 0.189 (0.1834)
  Follow Up (Day 15), n=6,6,6,6,6,6,6,6,16 | 0.027 (0.1876) | 0.145 (0.2041) | -0.060 (0.3138) | 0.023 (0.3370) | -0.205 (0.1639) | 0.053 (0.1549) | -0.295 (0.2001) | 0.007 (0.2067) | 0.032 (0.2691)

4. Primary Outcome: Part 1: Change From Baseline in Hematology Parameters: Erythrocytes Mean Corpuscular Volume (Erythrocyte MCV).
Description: Blood samples were collected to analyze the hematology parameters: erythrocyte MCV. Day -2 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day -2), 24 hours, 48 hours, 96 hours and Follow up (Day 15)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Femtoliter
Arm/Group | Part 1: GSK3640254 1 mg | Part 1: GSK3640254 3 mg | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 30mg | Part 1: GSK3640254 100 mg | Part 1: GSK3640254 200 mg | Part 1: GSK3640254 400 mg | Part 1: GSK3640254 700 mg | Part 1: Single Dose Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16
Femtoliter
  24 hour, n=6,6,6,6,6,6,5,6,16: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 6 | 16
  24 hour, n=6,6,6,6,6,6,5,6,16 | -0.50 (1.390) | -0.03 (0.497) | 0.17 (0.689) | 0.70 (0.494) | -1.07 (0.575) | -0.28 (1.192) | -0.64 (0.754) | -0.25 (0.853) | 0.05 (0.797)
  48 hour, n=6,6,5,6,6,6,6,6,16: number analyzed (Participants) | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 16
  48 hour, n=6,6,5,6,6,6,6,6,16 | -0.42 (0.966) | 0.35 (1.231) | 0.06 (0.673) | 0.13 (0.659) | -0.57 (0.843) | 0.10 (1.135) | -1.18 (0.703) | -0.18 (0.725) | 0.24 (0.932)
  96 hour,n=6,6,6,6,6,6,6,6,15: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 15
  96 hour,n=6,6,6,6,6,6,6,6,15 | 1.75 (0.619) | 0.43 (0.950) | 0.02 (0.979) | -0.22 (1.030) | -0.85 (1.214) | 0.28 (1.177) | -0.15 (0.616) | -0.13 (0.388) | 0.20 (1.196)
  Follow up (Day 15), n=6,6,6,6,6,6,6,6,16 | 0.15 (1.263) | 1.83 (0.505) | 0.53 (0.850) | -0.20 (1.241) | -0.15 (1.253) | 0.42 (1.339) | -0.10 (1.567) | -0.28 (0.840) | 0.14 (1.153)

5. Primary Outcome: Part 1: Change From Baseline in Hematology Parameter: Erythrocytes Mean Corpuscular Hemoglobin (Erythrocyte MCH)
Description: Blood samples were collected to analyze the hematology parameter: Erythrocyte MCH. Day -2 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.Results are presented treatment wise.
Time Frame: Baseline (Day -2), 24 hours, 48 hours, 96 hours and Follow up (Day 15)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | Part 1: GSK3640254 1 mg | Part 1: GSK3640254 3 mg | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 30mg | Part 1: GSK3640254 100 mg | Part 1: GSK3640254 200 mg | Part 1: GSK3640254 400 mg | Part 1: GSK3640254 700 mg | Part 1: Single Dose Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16
Picograms
  24 hours, n=6,6,6,6,6,6,5,6,16: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 6 | 16
  24 hours, n=6,6,6,6,6,6,5,6,16 | 0.12 (0.337) | 0.18 (0.147) | 0.00 (0.438) | -0.15 (0.596) | 0.25 (0.485) | 0.15 (0.339) | 0.08 (0.963) | -0.07 (0.700) | 0.01 (0.635)
  48 hours, n=6,6,5,6,6,6,6,6,16: number analyzed (Participants) | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 16
  48 hours, n=6,6,5,6,6,6,6,6,16 | 0.15 (0.464) | 0.08 (0.271) | 0.14 (0.321) | 0.37 (0.779) | 0.73 (0.450) | -0.18 (0.397) | -0.03 (0.821) | 0.13 (0.446) | 0.18 (0.583)
  96 hours,n=6,6,6,6,6,6,6,6,15: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 15
  96 hours,n=6,6,6,6,6,6,6,6,15 | 0.47 (0.339) | 0.02 (0.194) | -0.33 (0.301) | 0.17 (1.111) | 0.63 (0.589) | -0.02 (0.319) | -0.13 (0.459) | -0.13 (0.497) | 0.17 (0.442)
  Follow up, Day 15,n=6,6,6,6,6,6,6,6,16 | -0.07 (0.266) | -0.27 (0.459) | 0.35 (0.660) | 0.03 (0.665) | 0.92 (0.741) | -0.40 (0.514) | -0.03 (0.207) | 0.02 (0.319) | 0.03 (0.639)

6. Primary Outcome: Part 1: Change From Baseline in Hematology Parameter: Hematocrit
Description: Blood samples were collected to analyze the hematology parameter: hematocrit. Day -2 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value. Results are presented treatment wise.
Time Frame: Baseline (Day -2), 24 hours, 48 hours, 96 hours and Follow up (Day 15)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage of red blood cells in blood
Arm/Group | Part 1: GSK3640254 1 mg | Part 1: GSK3640254 3 mg | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 30mg | Part 1: GSK3640254 100 mg | Part 1: GSK3640254 200 mg | Part 1: GSK3640254 400 mg | Part 1: GSK3640254 700 mg | Part 1: Single Dose Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16
Percentage of red blood cells in blood
  24 hours, n=6,6,6,6,6,6,5,6,16: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 6 | 16
  24 hours, n=6,6,6,6,6,6,5,6,16 | 0.0080 (0.02666) | 0.0288 (0.01150) | 0.0003 (0.01791) | 0.0163 (0.02526) | 0.0128 (0.02031) | 0.0155 (0.01058) | 0.0038 (0.01333) | 0.0250 (0.01416) | 0.0174 (0.0174)
  48 hours, n=6,6,5,6,6,6,6,6,16: number analyzed (Participants) | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 16
  48 hours, n=6,6,5,6,6,6,6,6,16 | 0.0123 (0.02767) | 0.0143 (0.01521) | -0.0018 (0.02255) | 0.0102 (0.02851) | 0.0103 (0.01256) | 0.0252 (0.00970) | 0.0013 (0.01739) | 0.0148 (0.02179) | 0.0163 (0.0163)
  96 hours,n=6,6,6,6,6,6,6,6,15: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 15
  96 hours,n=6,6,6,6,6,6,6,6,15 | 0.0223 (0.01896) | 0.0198 (0.01771) | 0.0078 (0.02337) | 0.0145 (0.02346) | -0.0072 (0.02753) | 0.0108 (0.00947) | 0.0045 (0.02345) | 0.0200 (0.02265) | 0.0177 (0.0177)
  Follow up (Day 15), n=6,6,6,6,6,6,6,6,16 | 0.0032 (0.02247) | 0.0222 (0.01879) | -0.0025 (0.02848) | 0.0012 (0.03201) | -0.0185 (0.01816) | 0.0070 (0.01534) | -0.0265 (0.01852) | -0.0007 (0.01945) | 0.0035 (0.02603)

7. Primary Outcome: Part 1: Change From Baseline in Hematology Parameter: Percentage of Reticulocytes
Description: Blood samples were collected to analyze the hematology parameter: percentage of reticulocytes. Day -2 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value. Results are presented treatment wise.
Time Frame: Baseline (Day -2), 24 hours, 48 hours, 96 hours and Follow up (Day 15)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | Part 1: GSK3640254 1 mg | Part 1: GSK3640254 3 mg | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 30mg | Part 1: GSK3640254 100 mg | Part 1: GSK3640254 200 mg | Part 1: GSK3640254 400 mg | Part 1: GSK3640254 700 mg | Part 1: Single Dose Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16
10^12 cells per liter
  24 hours, n=6,6,6,6,6,6,5,6,16: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 6 | 16
  24 hours, n=6,6,6,6,6,6,5,6,16 | 0.00050 (0.001390) | 0.00055 (0.001608) | 0.00118 (0.001955) | -0.00023 (0.002223) | 0.00022 (0.001694) | -0.00015 (0.001276) | 0.00156 (0.002490) | 0.00057 (0.000579) | 0.00071 (0.001808)
  48 hours, n=6,6,5,6,6,6,6,6,16: number analyzed (Participants) | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 16
  48 hours, n=6,6,5,6,6,6,6,6,16 | 0.00082 (0.001496) | 0.00123 (0.001334) | 0.00154 (0.001790) | -0.00017 (0.002028) | 0.00070 (0.001451) | 0.00075 (0.001838) | 0.00260 (0.002924) | 0.00117 (0.001859) | 0.00118 (0.002221)
  96 hours,n=6,6,6,6,6,6,6,6,15: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 15
  96 hours,n=6,6,6,6,6,6,6,6,15 | -0.00005 (0.002040) | 0.00160 (0.001615) | 0.00095 (0.002517) | 0.00023 (0.001965) | 0.00138 (0.001841) | 0.00060 (0.001663) | 0.00265 (0.002867) | 0.00175 (0.002019) | 0.00162 (0.002889)
  Follow up (Day 15), n=6,6,6,6,6,6,6,6,16 | -0.00018 (0.001273) | 0.00435 (0.001628) | -0.00077 (0.002293) | -0.00042 (0.002832) | 0.00092 (0.002495) | -0.00015 (0.001640) | -0.00002 (0.001841) | 0.00055 (0.002230) | 0.00061 (0.003329)

8. Primary Outcome: Part 1: Change From Baseline in Hematology Parameter: Hemoglobin (Hb)
Description: Blood samples were collected to analyze the hematology parameter: Hb. Day -2 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value. Results are presented treatment wise.
Time Frame: Baseline (Day -2), 24 hours, 48 hours, 96 hours and Follow up (Day 15)
Population: Safety Population. Only those participants with data available at the specified data points were analyzed (represented by n=X in the category titles).
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Part 1: GSK3640254 1 mg | Part 1: GSK3640254 3 mg | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 30mg | Part 1: GSK3640254 100 mg | Part 1: GSK3640254 200 mg | Part 1: GSK3640254 400 mg | Part 1: GSK3640254 700 mg | Part 1: Single Dose Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16
Grams per liter
  24 hours, n=6,6,6,6,6,6,5,6,16: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 6 | 16
  24 hours, n=6,6,6,6,6,6,5,6,16 | 4.2 (8.93) | 10.8 (3.43) | 0.0 (5.51) | 3.5 (7.34) | 7.7 (5.82) | 6.8 (1.72) | 3.0 (6.04) | 8.8 (7.91) | 5.9 (7.29)
  48 hours, n=6,6,5,6,6,6,6,6,16: number analyzed (Participants) | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 16
  48 hours, n=6,6,5,6,6,6,6,6,16 | 5.7 (10.65) | 4.7 (5.89) | 0.0 (6.60) | 5.2 (6.88) | 8.3 (3.20) | 7.7 (3.72) | 2.5 (6.35) | 6.2 (7.88) | 6.0 (7.85)
  96 hours, n=6,6,6,6,6,6,6,6,15: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 15
  96 hours, n=6,6,6,6,6,6,6,6,15 | 6.8 (6.27) | 6.0 (5.33) | 0.8 (6.49) | 6.3 (7.00) | 2.3 (7.97) | 3.2 (2.71) | 1.2 (9.13) | 6.5 (9.67) | 6.6 (5.51)
  Follow up (Day 15), n=6,6,6,6,6,6,6,6,16 | 0.5 (5.75) | 3.0 (7.24) | 0.0 (11.05) | 1.0 (7.97) | -1.5 (7.06) | -0.5 (3.39) | -9.2 (6.82) | 0.2 (6.37) | 1.0 (8.25)

9. Primary Outcome: Part 1: Change From Baseline in Clinical Chemistry Parameter: Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), Alkaline Phosphate (ALP)
Description: Blood samples were collected to analyze the chemistry parameter: ALT, AST, and ALP. Day -2 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value. Results are presented treatment wise.
Time Frame: Baseline (Day -2), 24 hours, 48 hours, 96 hours and Follow up (Day 15)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | Part 1: GSK3640254 1 mg | Part 1: GSK3640254 3 mg | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 30mg | Part 1: GSK3640254 100 mg | Part 1: GSK3640254 200 mg | Part 1: GSK3640254 400 mg | Part 1: GSK3640254 700 mg | Part 1: Single Dose Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16
International units per liter
  ALT, 24 hours, n=6,6,6,6,6,6,6,6,16 | -1.7 (4.55) | 0.3 (3.39) | 0.8 (3.60) | -3.8 (2.04) | -0.5 (4.93) | -3.8 (3.49) | 0.0 (5.44) | -0.3 (5.05) | -0.8 (4.68)
  ALT, 48 hours, n=6,6,6,6,6,6,6,5,16: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 16
  ALT, 48 hours, n=6,6,6,6,6,6,6,5,16 | -1.5 (5.75) | -0.2 (4.49) | 0.3 (4.37) | 1.2 (2.23) | 0.5 (4.04) | -2.7 (6.25) | -2.7 (4.89) | 5.0 (10.17) | -0.1 (4.94)
  ALT, 96 hours, n=6,6,6,6,6,6,6,6,15: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 15
  ALT, 96 hours, n=6,6,6,6,6,6,6,6,15 | -0.5 (5.01) | 4.0 (3.90) | 1.3 (4.68) | 2.2 (3.19) | 2.5 (5.47) | -3.5 (8.26) | 0.5 (4.85) | 3.8 (10.76) | 2.5 (8.08)
  ALT, FU (Day 15), n=6,6,6,6,6,6,6,6,16 | -0.3 (10.01) | 2.3 (4.32) | 2.3 (3.56) | 9.5 (14.46) | 5.2 (9.95) | 0.3 (14.35) | 1.0 (4.34) | 5.3 (6.06) | 5.1 (15.95)
  AST, 24 hours, n=6,6,6,6,6,6,6,6,16 | -5.7 (7.63) | -0.4 (3.13) | -2.5 (2.88) | -4.2 (1.94) | -3.5 (4.72) | -4.7 (6.74) | -0.7 (3.72) | -1.3 (2.94) | -3.0 (3.60)
  AST, 48 hours, n=6,6,6,6,6,6,6,5,16: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 16
  AST, 48 hours, n=6,6,6,6,6,6,6,5,16 | -4.3 (7.50) | -2.3 (3.83) | -3.0 (2.10) | -2.2 (1.72) | -0.7 (4.80) | -2.5 (3.33) | -2.0 (3.85) | 1.4 (5.86) | -2.6 (4.11)
  AST, 96 hours, n=6,6,6,6,6,6,6,6,15: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 15
  AST, 96 hours, n=6,6,6,6,6,6,6,6,15 | -4.2 (8.57) | -1.7 (3.20) | -4.2 (3.97) | -1.3 (2.73) | -3.3 (4.89) | -4.5 (4.85) | -1.8 (4.31) | -1.5 (4.89) | -1.4 (3.48)
  AST, FU (Day 15), n=6,6,6,6,6,6,6,6,16 | -1.5 (8.53) | 4.5 (9.57) | 1.0 (5.18) | -0.5 (2.88) | 4.5 (5.36) | -1.7 (2.80) | 2.2 (8.26) | 0.9 (5.87) | 0.9 (5.87)
  ALP, 24 hours, n=6,6,6,6,6,6,6,6,16 | 2.8 (4.54) | 6.0 (3.74) | 1.2 (8.28) | -1.0 (6.66) | -2.8 (6.15) | -1.2 (8.42) | -0.2 (4.67) | 0.7 (3.78) | -2.9 (4.10)
  ALP, 48 hours, n=6,6,6,6,6,6,6,5,16: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 16
  ALP, 48 hours, n=6,6,6,6,6,6,6,5,16 | 3.3 (4.93) | 1.7 (5.13) | 2.2 (6.24) | -0.8 (5.31) | -1.7 (6.65) | -1.5 (8.29) | -0.8 (5.31) | 0.6 (2.97) | -2.4 (4.84)
  ALP, 96 hours, n=6,6,6,6,6,6,6,6,15: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 15
  ALP, 96 hours, n=6,6,6,6,6,6,6,6,15 | 3.3 (4.18) | 5.2 (2.93) | 3.5 (10.09) | 0.0 (5.18) | 0.5 (4.85) | -4.8 (9.11) | 1.5 (6.19) | 1.2 (3.49) | -1.1 (4.16)
  ALP, FU (Day 15), n=6,6,6,6,6,6,6,6,16 | 0.3 (1.37) | 1.5 (3.27) | -0.5 (4.81) | 2.2 (6.62) | -1.2 (6.97) | -1.8 (6.01) | -0.8 (5.98) | -0.3 (1.97) | -0.4 (6.37)

10. Primary Outcome: Part 1: Change From Baseline in Clinical Chemistry Parameters : Bicarbonate, Calcium, Chloride, Magnesium, Phosphate, Potassium, Sodium, Urea
Description: Blood samples were collected to analyze the chemistry parameter: bicarbonate, calcium, chloride, magnesium, phosphate, potassium, sodium, urea. Day -2 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value. Results are presented treatment wise.
Time Frame: Baseline (Day -2), 24 hours, 48 hours, 96 hours and Follow up (Day 15)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Part 1: GSK3640254 1 mg | Part 1: GSK3640254 3 mg | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 30mg | Part 1: GSK3640254 100 mg | Part 1: GSK3640254 200 mg | Part 1: GSK3640254 400 mg | Part 1: GSK3640254 700 mg | Part 1: Single Dose Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16
Millimoles per liter
  Bicarbonate, 24 hours, n=6,6,6,6,6,6,6,6,16 | 0.7 (1.86) | 3.0 (3.03) | -3.2 (3.06) | 2.2 (2.04) | -0.2 (2.14) | 0.5 (1.76) | -2.2 (1.47) | 0.0 (1.67) | 0.8 (2.59)
  Bicarbonate, 48 hours, n=6,6,6,6,6,6,6,5,16: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 16
  Bicarbonate, 48 hours, n=6,6,6,6,6,6,6,5,16 | 0.3 (1.86) | 3.5 (2.66) | -1.3 (2.42) | 2.7 (1.86) | 2.2 (1.94) | 5.8 (3.71) | -0.5 (1.38) | -1.8 (1.64) | 2.1 (3.57)
  Bicarbonate, 96 hours, n=6,6,6,6,6,6,6,6,15: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 15
  Bicarbonate, 96 hours, n=6,6,6,6,6,6,6,6,15 | -1.2 (1.72) | 2.0 (3.41) | -2.0 (2.76) | 1.3 (2.50) | -1.2 (4.31) | 0.8 (1.94) | -2.2 (2.04) | -2.2 (2.32) | 1.1 (2.47)
  Bicarbonate,FU (Day 15), n=6,6,6,6,6,6,6,6,16 | 0.2 (1.47) | 1.5 (1.05) | -1.8 (2.64) | 1.7 (1.75) | 1.2 (1.94) | 1.2 (2.93) | -0.3 (2.88) | -0.8 (1.47) | 1.1 (1.65)
  Calcium, 24 hours, n=6,6,6,6,6,6,6,6,16 | -0.045 (0.0931) | 0.038 (0.0627) | -0.037 (0.0866) | -0.033 (0.0987) | -0.012 (0.0492) | 0.060 (0.0562) | 0.035 (0.0731) | 0.002 (0.0454) | 0.005 (0.0647)
  Calcium, 48 hours, n=6,6,6,6,6,6,6,5,16: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 16
  Calcium, 48 hours, n=6,6,6,6,6,6,6,5,16 | 0.047 (0.0997) | 0.042 (0.0581) | -0.032 (0.0731) | -0.008 (0.0808) | 0.008 (0.0736) | 0.145 (0.0568) | -0.017 (0.0476) | -0.018 (0.0349) | 0.031 (0.0762)
  Calcium, 96 hours, n=6,6,6,6,6,6,6,6,15: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 15
  Calcium, 96 hours, n=6,6,6,6,6,6,6,6,15 | -0.005 (0.0909) | 0.070 (0.0687) | -0.012 (0.0838) | 0.027 (0.0747) | -0.015 (0.0680) | 0.097 (0.0625) | 0.025 (0.0497) | -0.045 (0.0836) | 0.034 (0.0687)
  Calcium, FU (Day 15), n=6,6,6,6,6,6,6,6,16 | 0.003 (0.0686) | 0.060 (0.0620) | 0.008 (0.1194) | 0.003 (0.0709) | -0.047 (0.0528) | 0.043 (0.0753) | -0.017 (0.1134) | -0.027 (0.0455) | 0.033 (0.0694)
  Chloride, 24 hours, n=6,6,6,6,6,6,6,6,16 | 1.8 (1.47) | -2.2 (2.04) | 2.7 (2.07) | -0.5 (1.87) | 0.2 (3.06) | 0.5 (2.66) | -0.7 (2.16) | 0.3 (2.73) | 0.6 (2.00)
  Chloride, 48 hours, n=6,6,6,6,6,6,6,5,16: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 16
  Chloride, 48 hours, n=6,6,6,6,6,6,6,5,16 | 1.8 (1.47) | -0.8 (1.47) | 2.3 (1.63) | -2.0 (1.90) | -0.2 (2.32) | 0.7 (3.08) | -0.7 (2.73) | 0.6 (1.95) | 0.5 (1.75)
  Chloride, 96 hours, n=6,6,6,6,6,6,6,6,15: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 15
  Chloride, 96 hours, n=6,6,6,6,6,6,6,6,15 | 1.7 (1.21) | -1.2 (2.99) | 1.0 (2.00) | 0.0 (1.79) | -0.5 (2.88) | 0.3 (2.94) | 0.7 (2.16) | -1.3 (1.97) | 0.1 (2.76)
  Chloride, FU (Day 15), n=6,6,6,6,6,6,6,6,16 | 0.7 (1.37) | -0.3 (2.25) | 0.5 (1.64) | -0.3 (2.07) | 1.3 (3.39) | 0.8 (2.48) | 0.8 (2.48) | -0.7 (3.27) | -0.6 (1.75)
  Magnesium, 24 hours, n=6,6,6,6,6,6,6,6,16 | -0.018 (0.0483) | -0.017 (0.0350) | 0.023 (0.0393) | 0.023 (0.0398) | 0.003 (0.0393) | 0.033 (0.0398) | 0.003 (0.0339) | 0.012 (0.0560) | 0.014 (0.0495)
  Magnesium, 48 hours, n=6,6,6,6,6,6,6,5,16: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 16
  Magnesium, 48 hours, n=6,6,6,6,6,6,6,5,16 | 0.043 (0.0983) | 0.005 (0.0513) | 0.035 (0.0468) | 0.012 (0.0349) | 0.017 (0.0476) | 0.060 (0.0369) | 0.025 (0.0459) | 0.034 (0.0513) | 0.034 (0.0626)
  Magnesium, 96 hours, n=6,6,6,6,6,6,6,6,15: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 15
  Magnesium, 96 hours, n=6,6,6,6,6,6,6,6,15 | 0.010 (0.0525) | 0.022 (0.0488) | 0.037 (0.0535) | 0.015 (0.0568) | 0.002 (0.0264) | 0.048 (0.0204) | 0.033 (0.0308) | 0.007 (0.0476) | 0.042 (0.0507)
  Magnesium, FU (Day 15), n=6,6,6,6,6,6,6,6,16 | 0.008 (0.0643) | -0.035 (0.0367) | -0.020 (0.0583) | 0.010 (0.0502) | -0.017 (0.0361) | 0.017 (0.0367) | 0.013 (0.0550) | -0.015 (0.0468) | 0.002 (0.0489)
  Phosphate, 24 hours, n=6,6,6,6,6,6,6,6,16 | 0.088 (0.1074) | 0.117 (0.1777) | 0.098 (0.1843) | -0.080 (0.1370) | -0.003 (0.1279) | -0.010 (0.1803) | 0.032 (0.1647) | -0.018 (0.0968) | 0.020 (0.1363)
  Phosphate, 48 hours, n=6,6,6,6,6,6,6,5,16: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 16
  Phosphate, 48 hours, n=6,6,6,6,6,6,6,5,16 | 0.148 (0.0679) | -0.022 (0.1713) | 0.107 (0.1540) | -0.063 (0.1528) | -0.043 (0.1499) | -0.058 (0.1816) | 0.025 (0.1801) | -0.076 (0.0963) | 0.022 (0.1561)
  Phosphate, 96 hours, n=6,6,6,6,6,6,6,6,15: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 15
  Phosphate, 96 hours, n=6,6,6,6,6,6,6,6,15 | 0.077 (0.1084) | 0.122 (0.1854) | 0.098 (0.1485) | -0.055 (0.1934) | -0.028 (0.0995) | -0.027 (0.1645) | 0.092 (0.1240) | 0.042 (0.1144) | 0.029 (0.1391)
  Phosphate, FU (Day 15), n=6,6,6,6,6,6,6,6,16 | 0.107 (0.1224) | -0.018 (0.1230) | 0.1230 (0.1378) | -0.090 (0.1485) | 0.042 (0.1865) | -0.055 (0.1407) | 0.063 (0.1138) | 0.002 (0.1341) | -0.022 (0.1285)
  Potassium, 24 hours, n=6,6,6,6,6,6,6,6,16 | 0.03 (0.647) | 0.42 (0.313) | 0.33 (0.327) | 0.20 (0.290) | 0.20 (0.276) | 0.22 (0.313) | 0.10 (0.245) | -0.05 (0.423) | 0.25 (0.316)
  Potassium, 48 hours, n=6,6,6,6,6,6,6,5,16: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 16
  Potassium, 48 hours, n=6,6,6,6,6,6,6,5,16 | 0.28 (0.417) | 0.30 (0.310) | 0.25 (0.217) | 0.07 (0.258) | 0.20 (0.253) | 0.30 (0.228) | 0.07 (0.163) | 0.06 (0.251) | 0.16 (0.278)
  Potassium, 96 hours, n=6,6,6,6,6,6,6,6,15: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 15
  Potassium, 96 hours, n=6,6,6,6,6,6,6,6,15 | 0.00 (0.525) | 0.30 (0.335) | 0.38 (0.306) | 0.12 (0.232) | 0.20 (0.352) | 0.20 (0.316) | 0.08 (0.232) | -0.12 (0.204) | 0.30 (0.314)
  Potassium, FU (Day 15), n=6,6,6,6,6,6,6,6,16 | 0.12 (0.436) | 0.43 (0.413) | -0.05 (0.207) | -0.03 (0.356) | 0.07 (0.250) | 0.18 (0.183) | 0.05 (0.339) | -0.27 (0.314) | 0.10 (0.379)
  Sodium, 24 hours, n=6,6,6,6,6,6,6,6,16 | 0.0 (1.26) | 0.0 (1.90) | 0.3 (2.16) | -0.7 (1.63) | -1.5 (0.55) | -0.3 (2.42) | -1.3 (1.21) | 0.5 (2.26) | 0.3 (1.95)
  Sodium, 48 hours, n=6,6,6,6,6,6,6,5,16: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 16
  Sodium, 48 hours, n=6,6,6,6,6,6,6,5,16 | 1.0 (1.10) | -0.2 (2.14) | 1.0 (1.67) | -0.7 (1.37) | -1.8 (1.60) | 1.2 (2.23) | -1.3 (2.25) | 0.8 (1.92) | 0.8 (1.80)
  Sodium, 96 hours, n=6,6,6,6,6,6,6,6,15: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 15
  Sodium, 96 hours, n=6,6,6,6,6,6,6,6,15 | 0.8 (1.47) | 0.5 (1.64) | 0.7 (1.21) | 1.3 (3.01) | -1.7 (1.86) | 0.0 (0.20) | 0.8 (1.83) | 1.3 (1.03) | 0.5 (2.42)
  Sodium, FU (Day 15), n=6,6,6,6,6,6,6,6,16 | 0.8 (2.14) | 0.3 (2.07) | -0.2 (1.47) | -0.2 (1.47) | 0.8 (1.72) | 0.7 (2.07) | 0.5 (2.17) | 0.0 (2.19) | 0.4 (1.82)
  Urea, 24 hours, n=6,6,6,6,6,6,6,6,16 | 0.033320 (0.3443425) | 0.283220 (1.0396160) | 0.299880 (0.6630596) | -0.649740 (1.0517198) | -0.166600 (0.8450414) | -0.599760 (0.7717016) | 0.133280 (0.3880028) | -0.849660 (1.3570283) | -0.187425 (0.9102217)
  Urea, 48 hours, n=6,6,6,6,6,6,6,5,16: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 16
  Urea, 48 hours, n=6,6,6,6,6,6,6,5,16 | -0.316540 (0.8081731) | 0.416500 (0.8769556) | 0.116620 (0.7701895) | -0.683060 (1.0103710) | -0.233240 (0.9601712) | -0.316540 (0.6366649) | 0.083300 (0.7108180) | -1.099560 (0.8242913) | -0.187425 (1.0590572)
  Urea, 96 hours, n=6,6,6,6,6,6,6,6,15: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 15
  Urea, 96 hours, n=6,6,6,6,6,6,6,6,15 | -0.116620 (0.7274909) | 0.233240 (0.9476011) | 0.316540 (1.0510863) | -0.733040 (1.1736967) | -0.433160 (0.5986483) | 0.049980 (0.5955804) | 0.166600 (0.9241120) | -0.916300 (1.5178348) | 0.046648 (1.2598057)
  Urea,FU (Day 15), n=6,6,6,6,6,6,6,6,16 | -0.483140 (0.9491815) | 0.466480 (0.9929136) | 0.466480 (0.3828177) | -0.499800 (0.5930586) | -0.233240 (2.0187631) | -0.649740 (0.7173480) | -0.033320 (1.0907403) | -1.332800 (1.4230410) | -0.099960 (0.6590288)

11. Primary Outcome: Part 1: Change From Baseline in Cholesterol, Glucose, High Density Lipoprotein (HDL) Cholesterol, Low Density Cholesterol (LDL) Cholesterol, Triglycerides
Description: Blood samples were collected to analyze the chemistry parameter: cholesterol, glucose, HDL cholesterol, LDL cholesterol, triglycerides. Day -2 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value. Results are presented treatment wise.
Time Frame: Baseline (Day -2) and Day 1 (96 hours) and Follow up (Day 15)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Part 1: GSK3640254 1 mg | Part 1: GSK3640254 3 mg | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 30mg | Part 1: GSK3640254 100 mg | Part 1: GSK3640254 200 mg | Part 1: GSK3640254 400 mg | Part 1: GSK3640254 700 mg | Part 1: Single Dose Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16
Millimoles per liter
  Cholesterol,Day1,96 hours,n=5,6,6,6,5,6,6,6,14: number analyzed (Participants) | 5 | 6 | 6 | 6 | 5 | 6 | 6 | 6 | 14
  Cholesterol,Day1,96 hours,n=5,6,6,6,5,6,6,6,14 | 0.40 (0.324) | 0.32 (0.271) | -0.05 (0.628) | 0.02 (0.422) | -0.06 (0.699) | 0.13 (0.516) | 0.45 (0.373) | 0.43 (0.641) | 0.30 (0.445)
  Cholesterol, FU (Day 15), n=6,6,6,6,6,6,6,6,16 | 0.25 (0.404) | 0.23 (0.327) | 0.07 (0.579) | 0.23 (0.493) | -0.16 (0.590) | -0.40 (0.562) | 0.08 (0.445) | 0.22 (0.496) | 0.16 (0.566)
  HDL cholesterol,Day1,96 hours,n=6,6,6,6,5,6,6,6,15: number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 6 | 6 | 6 | 15
  HDL cholesterol,Day1,96 hours,n=6,6,6,6,5,6,6,6,15 | -0.02 (0.041) | -0.05 (0.105) | -0.15 (0.152) | -0.12 (0.147) | -0.22 (0.084) | -0.12 (0.098) | -0.02 (0.133) | -0.13 (0.103) | -0.08 (0.174)
  HDL cholesterol, FU (Day 15), n=6,6,6,6,5,6,6,6,16: number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 6 | 6 | 6 | 16
  HDL cholesterol, FU (Day 15), n=6,6,6,6,5,6,6,6,16 | 0.07 (0.137) | -0.05 (0.122) | -0.02 (0.160) | 0.00 (0.179) | -0.18 (0.148) | -0.05 (0.105) | -0.02 (0.264) | -0.03 (0.103) | 0.00 (0.219)
  LDL cholesterol,Day1, 96hours,n=5,6,6,6,5,6,6,6,14: number analyzed (Participants) | 5 | 6 | 6 | 6 | 5 | 6 | 6 | 6 | 14
  LDL cholesterol,Day1, 96hours,n=5,6,6,6,5,6,6,6,14 | 0.30 (0.122) | 0.10 (0.562) | -0.12 (0.519) | -0.13 (0.408) | -0.04 (0.428) | -0.03 (0.361) | 0.43 (0.441) | 0.25 (0.281) | 0.16 (0.386)
  LDL cholesterol, FU(Day 15), n=6,6,6,6,5,6,6,6,16: number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 6 | 6 | 6 | 16
  LDL cholesterol, FU(Day 15), n=6,6,6,6,5,6,6,6,16 | 0.30 (0.210) | 0.15 (0.295) | 0.22 (0.564) | 0.07 (0.314) | -0.14 (0.472) | -0.35 (0.451) | 0.37 (0.308) | 0.07 (0.327) | 0.13 (0.491)
  Triglycerides,Day1,96 hours,n=5,6,6,6,5,6,6,6,14: number analyzed (Participants) | 5 | 6 | 6 | 6 | 5 | 6 | 6 | 6 | 14
  Triglycerides,Day1,96 hours,n=5,6,6,6,5,6,6,6,14 | 0.28 (0.531) | 0.60 (1.079) | 0.45 (0.468) | 0.62 (1.026) | 0.52 (0.931) | 0.60 (0.883) | 0.03 (0.468) | 0.70 (0.834) | 0.49 (0.360)
  Triglycerides, FU (Day 15),n=6,6,6,6,5,6,6,6,16: number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 6 | 6 | 6 | 16
  Triglycerides, FU (Day 15),n=6,6,6,6,5,6,6,6,16 | -0.20 (0.297) | 0.32 (0.838) | -0.30 (0.303) | 0.40 (0.940) | 0.40 (0.831) | 0.02 (0.279) | -0.55 (0.501) | 0.40 (0.410) | 0.05 (0.588)

12. Primary Outcome: Part 1: Change From Baseline in Chemistry Parameter: Glucose
Description: Blood samples were collected to analyze the chemistry parameter: glucose . Day -2 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value. Results are presented treatment wise.
Time Frame: Baseline (Day -2) and Day 1 (96 hours) and Follow up (Day 15)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Part 1: GSK3640254 1 mg | Part 1: GSK3640254 3 mg | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 30mg | Part 1: GSK3640254 100 mg | Part 1: GSK3640254 200 mg | Part 1: GSK3640254 400 mg | Part 1: GSK3640254 700 mg | Part 1: Single Dose Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16
Millimoles per liter
  Day 1 (96 hours), n=5,6,6,6,6,6,6,6,14: number analyzed (Participants) | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 14
  Day 1 (96 hours), n=5,6,6,6,6,6,6,6,14 | -0.16 (0.288) | -0.30 (0.110) | -0.25 (0.414) | -0.28 (0.527) | -0.17 (0.446) | -0.08 (0.349) | -0.07 (0.432) | -0.33 (0.175) | -0.21 (0.279)
  FU (Day 15), n=6,6,6,6,6,6,6,6,16 | -0.03 (0.513) | -0.05 (0.345) | -0.12 (0.605) | -0.22 (0.471) | 0.07 (0.582) | -0.27 (0.367) | -0.27 (0.745) | 0.00 (0.374) | -0.04 (0.379)

13. Primary Outcome: Part 1: Change From Baseline in Clinical Chemistry Parameter: Bilirubin, Creatinine, Direct Bilirubin
Description: Blood samples were collected to analyze the chemistry parameter: bilirubin, creatinine, direct bilirubin . Day -2 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value. Results are presented treatment wise.
Time Frame: Baseline (Day -2), 24 hours, 48 hours, 96 hours and Follow up (Day 15)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Part 1: GSK3640254 1 mg | Part 1: GSK3640254 3 mg | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 30mg | Part 1: GSK3640254 100 mg | Part 1: GSK3640254 200 mg | Part 1: GSK3640254 400 mg | Part 1: GSK3640254 700 mg | Part 1: Single Dose Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16
Grams per liter
  Bilirubin, 24 hours, n=6,6,6,6,6,6,6,6,16 | -2.5 (2.88) | -0.2 (3.37) | -5.3 (3.33) | -1.5 (5.32) | 0.2 (3.19) | -1.7 (2.94) | -2.5 (1.97) | -0.3 (1.37) | -1.2 (3.19)
  Bilirubin, 48 hours, n=6,6,6,6,6,6,6,5,16: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 16
  Bilirubin, 48 hours, n=6,6,6,6,6,6,6,5,16 | -2.2 (3.19) | -0.8 (4.26) | -4.7 (3.20) | -0.7 (4.13) | 0.3 (2.50) | 0.3 (1.51) | -0.5 (2.35) | -1.6 (2.07) | -0.6 (2.97)
  Bilirubin, 96 hours, n=6,6,6,6,6,6,6,6,15: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 15
  Bilirubin, 96 hours, n=6,6,6,6,6,6,6,6,15 | -3.2 (2.32) | -2.5 (4.04) | -3.8 (3.60) | -1.3 (4.80) | -1.7 (3.14) | -0.2 (2.23) | -2.2 (2.79) | -1.05 (1.05) | -0.6 (2.61)
  Bilirubin, FU (Day 15),n=6,6,6,6,6,6,6,6,16 | -0.8 (3.43) | 3.3 (4.13) | -0.8 (2.56) | 2.5 (2.88) | 1.0 (5.10) | -1.0 (3.10) | 2.2 (4.92) | 2.0 (2.97) | 1.2 (4.20)
  Creatinine, 24 hours, n=6,6,6,6,6,6,6,6,16 | -7.0 (7.13) | 3.2 (5.85) | -0.5 (3.62) | 0.2 (5.49) | -1.2 (1.83) | 6.8 (4.62) | -0.7 (6.12) | -1.5 (9.03) | 0.6 (6.83)
  Creatinine, 48 hours, n=6,6,6,6,6,6,6,5,16: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 16
  Creatinine, 48 hours, n=6,6,6,6,6,6,6,5,16 | -6.7 (7.15) | 7.2 (4.96) | -1.2 (2.14) | -3.8 (5.34) | 0.8 (4.92) | 6.5 (6.25) | -1.7 (7.39) | -2.8 (8.76) | 0.8 (6.69)
  Creatinine, 96 hours, n=6,6,6,6,6,6,6,6,15: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 15
  Creatinine, 96 hours, n=6,6,6,6,6,6,6,6,15 | -2.5 (7.34) | 8.7 (4.89) | 3.2 (4.71) | 0.0 (5.33) | 0.0 (8.72) | 7.2 (4.36) | -5.3 (6.44) | -0.7 (5.47) | 4.6 (7.56)
  Creatinine, FU (Day 15), n=6,6,6,6,6,6,6,6,16 | -2.5 (6.38) | 9.3 (7.76) | -1.3 (5.09) | -1.7 (7.20) | 2.5 (4.97) | 3.0 (3.95) | -0.8 (7.05) | -11.2 (9.02) | 1.9 (6.69)
  Direct bilirubin, 24 hours, n=6,6,6,6,6,6,6,6,16 | -1.0 (1.26) | -0.5 (1.29) | -1.2 (1.30) | 0.2 (1.48) | -0.2 (1.10) | -1.0 (0.71) | -1.0 (0.63) | -0.3 (0.82) | -0.3 (1.23)
  Direct bilirubin, 48 hours, n=6,6,6,6,6,6,6,5,16: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 16
  Direct bilirubin, 48 hours, n=6,6,6,6,6,6,6,5,16 | -1.0 (1.55) | -0.8 (1.26) | -1.2 (0.75) | -0.3 (1.03) | 0.0 (0.71) | -0.2 (0.45) | -0.5 (0.55) | -0.8 (0.96) | -0.5 (1.10)
  Direct bilirubin, 96 hours, n=6,6,6,6,6,6,6,6,15: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 15
  Direct bilirubin, 96 hours, n=6,6,6,6,6,6,6,6,15 | -0.8 (1.48) | -1.0 (1.15) | -0.6 (1.14) | -0.3 (1.37) | -0.3 (0.50) | -0.2 (0.84) | -0.8 (0.45) | -0.8 (0.50) | -0.3 (0.90)
  Direct bilirubin, FU (Day 15),n=6,6,6,6,6,6,6,6,16 | -0.7 (1.21) | 1.0 (1.22) | 0.2 (0.75) | 1.0 (0.89) | 0.8 (0.96) | 0.0 (1.41) | 0.5 (1.52) | 0.7 (1.37) | 0.4 (1.36)

14. Primary Outcome: Part 1: Change From Baseline in Clinical Chemistry Parameter: Protein
Description: Blood samples were collected to analyze the chemistry parameter: Protein. Day -2 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day -2), 24 hours, 48 hours, 96 hours and Follow up (Day 15)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Part 1: GSK3640254 1 mg | Part 1: GSK3640254 3 mg | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 30mg | Part 1: GSK3640254 100 mg | Part 1: GSK3640254 200 mg | Part 1: GSK3640254 400 mg | Part 1: GSK3640254 700 mg | Part 1: Single Dose Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16
Grams per liter
  24 hours, n=6,6,6,6,6,6,6,6,16 | -0.3 (3.39) | 2.5 (0.84) | -5.2 (3.76) | -1.0 (3.16) | -1.2 (1.72) | 0.7 (1.21) | 0.3 (2.73) | 2.3 (2.25) | -0.8 (2.37)
  48 hours, n=6,6,6,6,6,6,6,5,16: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 16
  48 hours, n=6,6,6,6,6,6,6,5,16 | 0.7 (5.16) | 0.0 (1.26) | -4.0 (4.05) | -2.3 (2.42) | 0.3 (1.51) | 2.2 (1.33) | -0.3 (3.88) | 1.8 (2.28) | 0.2 (3.31)
  96 hours, n=6,6,6,6,6,6,6,6,15: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 15
  96 hours, n=6,6,6,6,6,6,6,6,15 | 1.2 (3.60) | 1.5 (3.39) | -2.0 (4.73) | 1.0 (4.10) | -1.7 (5.20) | 0.8 (1.94) | -0.3 (2.94) | 0.8 (3.60) | 1.3 (3.75)
  FU (Day 15),n=6,6,6,6,6,6,6,6,16 | -0.5 (3.62) | 0.7 (2.25) | -1.3 (6.31) | 0.2 (3.66) | -2.7 (3.20) | 1.7 (2.42) | -1.7 (3.98) | 1.7 (1.86) | 1.5 (3.85)

15. Primary Outcome: Part 1: Number of Participants With Abnormal Urinalysis
Description: Urine samples were collected at given time points to analyze the abnormal findings for potential of hydrogen (pH), glucose, protein, blood, ketones, bilirubin, urobilinogen, nitrite, leukocyte esterase by dipstick.
Time Frame: Up to Day 15
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK3640254 1 mg | Part 1: GSK3640254 3 mg | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 30mg | Part 1: GSK3640254 100 mg | Part 1: GSK3640254 200 mg | Part 1: GSK3640254 400 mg | Part 1: GSK3640254 700 mg | Part 1: Single Dose Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

16. Primary Outcome: Part 1: Change From Baseline in Vital Signs: Diastolic Blood Pressure (DBP) and Systolic Blood Pressure (SBP)
Description: SBP and DBP were measured in semi-supine position after 5 minutes rest for the participants at indicated time points. Day -1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value. Results are presented treatment wise.
Time Frame: Baseline (Day -1), 1,2,4.5,6,12,24,48,72,96 hours post dose and Follow up (Day 15)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Part 1: GSK3640254 1 mg | Part 1: GSK3640254 3 mg | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 30mg | Part 1: GSK3640254 100 mg | Part 1: GSK3640254 200 mg | Part 1: GSK3640254 400 mg | Part 1: GSK3640254 700 mg | Part 1: Single Dose Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16
Millimeters of mercury (mmHg)
  SBP, 1 hour n=6,6,6,6,6,6,6,6,16 | 2.5 (11.67) | 3.2 (4.45) | 6.3 (6.22) | 4.7 (6.77) | 6.2 (7.63) | 2.2 (11.07) | 5.8 (10.57) | 3.5 (4.93) | 8.1 (7.25)
  SBP, 2 hours n=6,6,6,6,6,6,6,6,16 | -0.7 (7.84) | 2.2 (4.17) | 8.8 (3.06) | 10.7 (6.62) | 0.5 (7.50) | 5.5 (8.46) | 5.7 (14.02) | 6.2 (6.11) | 4.4 (8.05)
  SBP, 4.5 hours, n=6,6,6,6,6,6,6,6,16 | 1.8 (7.22) | 5.3 (5.20) | 8.8 (5.60) | 5.3 (6.12) | 6.7 (7.42) | 10.8 (9.81) | 8.7 (11.04) | 4.0 (6.84) | 7.4 (11.04)
  SBP, 6 hours n=6,6,6,6,6,6,6,6,16 | 4.7 (5.75) | 4.7 (6.41) | 3.7 (4.63) | 9.5 (7.06) | 2.8 (7.73) | 4.0 (10.47) | 5.8 (12.81) | 6.5 (6.09) | 8.3 (10.97)
  SBP, 12 hours n=6,6,6,6,6,6,6,6,16 | 3.8 (6.24) | 8.7 (6.77) | 10.2 (5.04) | 8.2 (6.62) | 2.5 (8.29) | 3.3 (7.23) | 2.5 (17.62) | 6.3 (3.39) | 7.6 (7.90)
  SBP, 24 hours n=6,6,6,6,6,6,6,6,16 | -1.5 (5.54) | 3.2 (2.79) | 9.0 (6.32) | 3.3 (7.58) | -0.3 (4.46) | 2.7 (5.72) | 5.8 (8.30) | 0.8 (7.57) | 5.1 (10.68)
  SBP, 48 hours n=6,6,6,6,6,6,6,6,16 | -4.3 (6.59) | 1.3 (5.35) | 2.5 (8.22) | 0.3 (9.79) | 2.0 (11.45) | -0.5 (7.50) | 2.5 (6.98) | 2.2 (9.24) | 1.0 (8.68)
  SBP,72 hours n=6,6,6,6,6,6,6,6,16 | -2.0 (5.66) | 2.0 (7.24) | -0.8 (5.49) | 2.2 (8.52) | -3.0 (6.57) | 1.0 (6.00) | 2.5 (11.93) | 3.0 (12.02) | 2.4 (6.13)
  SBP, 96 hours n=6,6,6,6,6,6,6,6,15: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 15
  SBP, 96 hours n=6,6,6,6,6,6,6,6,15 | 1.8 (5.42) | 1.3 (5.35) | 6.0 (11.40) | 5.3 (12.71) | 3.0 (5.80) | 6.3 (7.53) | 2.5 (14.34) | 0.7 (6.19) | 4.5 (9.02)
  SBP, FU(Day 15), n=6,6,6,6,6,6,6,6,16 | 6.7 (9.18) | 1.0 (7.69) | 11.5 (7.92) | 6.8 (7.22) | 4.5 (10.21) | 4.5 (6.02) | 11.5 (3.33) | 7.8 (4.22) | 7.3 (10.20)
  DBP, 1 hour n=6,6,6,6,6,6,6,6,16 | -3.2 (8.84) | -3.7 (2.07) | 0.8 (6.18) | -1.2 (5.53) | -0.3 (4.32) | -2.0 (4.56) | 1.3 (9.87) | 0.5 (2.88) | 0.3 (8.62)
  DBP, 2 hours, n=6,6,6,6,6,6,6,6,16 | -7.5 (8.96) | -1.3 (3.27) | 1.0 (4.24) | -1.3 (6.83) | -2.7 (3.08) | -3.3 (3.93) | 1.0 (10.45) | 0.5 (2.35) | 0.5 (8.42)
  DBP, 4.5 hours, n=6,6,6,6,6,6,6,6,16 | -4.8 (6.91) | 2.3 (6.44) | 6.7 (6.77) | 1.7 (6.83) | 2.2 (3.06) | 1.5 (4.55) | 2.2 (6.31) | 6.3 (8.16) | 6.8 (10.10)
  DBP, 6 hours, n=6,6,6,6,6,6,6,6,16 | -3.5 (4.42) | -3.7 (4.93) | 0.2 (5.71) | 2.0 (3.74) | -2.2 (5.15) | -2.0 (6.48) | 1.8 (9.15) | 3.2 (7.78) | 2.4 (9.76)
  DBP, 12 hours, n=6,6,6,6,6,6,6,6,16 | 0.8 (8.23) | 0.3 (2.58) | 4.2 (3.76) | 4.3 (9.09) | 1.0 (5.10) | 1.0 (6.10) | 1.5 (12.61) | 5.3 (3.83) | 4.8 (7.64)
  DBP, 24 hours, n=6,6,6,6,6,6,6,6,16 | -0.3 (3.01) | -0.5 (3.78) | 4.7 (5.35) | 2.8 (7.44) | 0.0 (4.00) | 0.8 (5.56) | 6.2 (8.04) | 3.3 (4.63) | 3.7 (9.16)
  DBP, 48 hours, n=6,6,6,6,6,6,6,6,16 | -3.0 (6.29) | -1.7 (6.56) | 3.0 (5.29) | -2.5 (7.56) | 3.7 (5.65) | -1.3 (5.43) | 1.7 (8.71) | 1.0 (4.73) | 4.3 (8.90)
  DBP,72 hours, n=6,6,6,6,6,6,6,6,16 | -3.2 (6.08) | 0.0 (6.00) | 1.7 (7.17) | 1.0 (6.84) | -0.5 (5.09) | 1.7 (2.73) | 2.3 (8.71) | 4.7 (6.56) | 4.3 (8.02)
  DBP, 96 hours, n=6,6,6,6,6,6,6,6,15: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 15
  DBP, 96 hours, n=6,6,6,6,6,6,6,6,15 | -2.1 (6.59) | 1.0 (3.10) | 5.0 (6.69) | 2.5 (8.02) | 2.7 (3.78) | 2.3 (6.06) | 1.5 (12.63) | -0.2 (5.42) | 4.0 (7.39)
  DBP, FU(Day 15), n=6,6,6,6,6,6,6,6,16 | 0.7 (12.56) | -4.5 (5.50) | 6.8 (4.88) | 1.7 (7.37) | 2.5 (6.19) | 3.7 (5.20) | 7.3 (3.83) | 7.3 (5.35) | 7.1 (9.92)

17. Primary Outcome: Part 1: Change From Baseline in Vital Signs: Pulse Rate
Description: Pulse rate was measured in semi-supine position after 5 minutes rest for the participants at indicated time points. Day -1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value. Results are presented treatment wise.
Time Frame: Baseline (Day -1), 1,2,4.5,6,12,24,48,72,96 hours post dose and Follow up (Day 15)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Part 1: GSK3640254 1 mg | Part 1: GSK3640254 3 mg | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 30mg | Part 1: GSK3640254 100 mg | Part 1: GSK3640254 200 mg | Part 1: GSK3640254 400 mg | Part 1: GSK3640254 700 mg | Part 1: Single Dose Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16
Beats per minute
  1 hour n=6,6,6,6,6,6,6,6,16 | 13.3 (6.71) | 5.2 (2.48) | 14.5 (4.04) | 13.7 (5.05) | 11.3 (4.80) | 7.5 (3.67) | 9.0 (3.85) | 7.0 (2.97) | 9.6 (6.97)
  2 hours, n=6,6,6,6,6,6,6,6,16 | 7.3 (4.89) | 3.2 (4.96) | 6.8 (4.75) | 10.7 (9.09) | 12.8 (6.05) | 6.0 (3.22) | 7.0 (5.80) | 3.7 (9.65) | 8.2 (3.99)
  4.5 hours, n=6,6,6,6,6,6,6,6,16 | 6.5 (6.72) | 2.0 (7.56) | 3.7 (1.97) | 5.8 (4.40) | 8.2 (11.97) | 5.5 (3.94) | 4.2 (8.08) | 6.2 (6.85) | 6.4 (5.94)
  6 hours,n=6,6,6,6,6,6,6,6,16 | 16.8 (7.41) | 7.7 (5.85) | 9.7 (3.98) | 11.3 (6.02) | 11.2 (6.65) | 7.7 (3.88) | 8.3 (4.72) | 8.0 (3.16) | 10.4 (6.59)
  12 hours, n=6,6,6,6,6,6,6,6,16 | 10.2 (4.40) | 5.7 (7.55) | 11.8 (6.85) | 9.0 (5.83) | 11.0 (4.90) | 6.5 (8.96) | 8.0 (11.26) | 6.0 (7.51) | 7.3 (5.61)
  24 hours, n=6,6,6,6,6,6,6,6,16 | 5.2 (4.58) | 3.3 (4.37) | 2.3 (6.56) | 4.5 (9.48) | 6.7 (10.15) | 2.5 (5.68) | 5.8 (10.38) | 1.0 (4.86) | 0.2 (3.89)
  48 hours, n=6,6,6,6,6,6,6,6,16 | 0.8 (5.67) | 3.5 (7.31) | 3.2 (4.58) | 4.5 (6.89) | 4.8 (6.46) | -2.3 (6.83) | 10.8 (15.89) | 1.5 (6.35) | 1.5 (3.88)
  72 hours, n=6,6,6,6,6,6,6,6,16 | 2.0 (8.58) | 3.8 (5.00) | 2.8 (4.31) | 6.8 (4.49) | 2.0 (3.29) | -0.3 (6.19) | 4.5 (6.28) | -0.2 (7.14) | 1.4 (5.40)
  96 hours, n=6,6,6,6,6,6,6,6,15: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 15
  96 hours, n=6,6,6,6,6,6,6,6,15 | 12.5 (12.93) | 4.8 (4.83) | 4.8 (5.15) | 9.2 (6.88) | 5.7 (4.37) | 4.0 (2.45) | 2.8 (4.54) | 8.0 (4.47) | 2.5 (4.29)
  FU (Day 15), n=6,6,6,6,6,6,6,6,16 | 6.2 (4.71) | 3.3 (8.07) | 3.2 (6.52) | 6.3 (10.07) | 3.5 (3.99) | -0.7 (11.93) | 4.8 (6.97) | 6.3 (8.24) | 1.3 (5.74)

18. Primary Outcome: Part 1: Change From Baseline in Vital Signs: Temperature
Description: Temperature was measured in semi-supine position after 5 minutes rest for the participants at indicated time points. Day -1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value. Results are presented treatment wise.
Time Frame: Baseline (Day -1), 1,2,4.5,6,12,24,48,72,96 hours post dose and Follow up (Day 15)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | Part 1: GSK3640254 1 mg | Part 1: GSK3640254 3 mg | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 30mg | Part 1: GSK3640254 100 mg | Part 1: GSK3640254 200 mg | Part 1: GSK3640254 400 mg | Part 1: GSK3640254 700 mg | Part 1: Single Dose Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16
Degree Celsius
  1 hour, n=6,6,6,6,6,6,6,6,16 | 0.33 (0.186) | 0.15 (0.378) | 0.03 (0.333) | 0.18 (0.376) | 0.10 (0.303) | 0.00 (0.245) | 0.28 (0.256) | 0.22 (0.407) | 0.19 (0.267)
  2 hours, n=6,6,6,6,6,6,6,6,16 | 0.20 (0.237) | 0.00 (0.322) | 0.15 (0.378) | 0.28 (0.256) | 0.02 (0.256) | 0.27 (0.250) | 0.17 (0.388) | 0.52 (0.279) | 0.23 (0.322)
  4.5 hours, n=6,6,6,6,6,6,6,6,16 | 0.35 (0.308) | 0.23 (0.356) | 0.03 (0.350) | 0.07 (0.280) | 0.12 (0.360) | 0.45 (0.321) | 0.33 (0.308) | 0.42 (0.426) | 0.22 (0.299)
  6 hours, n=6,6,6,6,6,6,6,6,16 | 0.45 (0.274) | 0.27 (0.234) | 0.15 (0.339) | 0.42 (0.223) | 0.20 (0.210) | 0.45 (0.394) | 0.38 (0.264) | 0.75 (0.217) | 0.29 (0.390)
  12 hours, n=6,6,6,6,6,6,6,6,16 | 0.30 (0.219) | 0.20 (0.261) | 0.17 (0.350) | 0.20 (0.283) | 0.27 (0.493) | 0.18 (0.426) | 0.07 (0.175) | 0.53 (0.398) | 0.12 (0.259)
  24 hours, n=6,6,6,6,6,6,6,6,16 | -0.13 (0.266) | 0.10 (0.210) | 0.07 (0.175) | 0.05 (0.105) | 0.05 (0.596) | 0.10 (0.310) | 0.17 (0.103) | 0.23 (0.427) | 0.03 (0.244)
  48 hours, n=6,6,6,6,6,6,6,6,16 | -0.03 (0.234) | 0.10 (0.460) | -0.18 (0.214) | 0.07 (0.356) | -0.17 (0.250) | -0.03 (0.463) | 0.42 (0.694) | 0.27 (0.489) | 0.04 (0.301)
  72 hours, n=6,6,6,6,6,6,6,6,16 | 0.10 (0.110) | 0.23 (0.427) | 0.00 (0.316) | 0.18 (0.306) | -0.12 (0.488) | 0.17 (0.446) | 0.25 (0.217) | 0.15 (0.362) | 0.03 (0.317)
  96 hours, n=6,6,6,6,6,6,6,6,15: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 15
  96 hours, n=6,6,6,6,6,6,6,6,15 | 0.02 (0.232) | 0.10 (0.255) | 0.12 (0.160) | -0.18 (0.214) | -0.17 (0.628) | 0.22 (0.402) | 0.17 (0.216) | 0.08 (0.240) | -0.07 (0.313)
  FU (Day 15), n=6,6,6,6,6,6,6,6,16 | 0.05 (0.327) | -0.03 (0.344) | 0.12 (0.331) | 0.00 (0.518) | 0.20 (0.506) | 0.13 (0.344) | 0.18 (0.293) | 0.47 (0.398) | 0.11 (0.344)

19. Primary Outcome: Part 1: Change From Baseline in Vital Sign: Respiratory Rate
Description: Respiratory rate was measured in semi-supine position after 5 minutes rest for the participants at indicated time points. Day -1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value. Results are presented treatment wise.
Time Frame: Baseline (Day -1), 1,2,4.5,6,12,24,48,72,96 hours post dose and Follow up (Day 15)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Part 1: GSK3640254 1 mg | Part 1: GSK3640254 3 mg | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 30mg | Part 1: GSK3640254 100 mg | Part 1: GSK3640254 200 mg | Part 1: GSK3640254 400 mg | Part 1: GSK3640254 700 mg | Part 1: Single Dose Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16
Breaths per minute
  1 hour, n=6,6,6,6,6,6,6,6,16 | 1.5 (1.52) | 0.8 (2.14) | -0.3 (1.97) | 1.0 (0.89) | -1.0 (2.37) | 0.3 (1.51) | 0.5 (1.38) | 0.8 (2.04) | 0.1 (2.69)
  2 hours, n=6,6,6,6,6,6,6,6,16 | 1.7 (1.51) | 1.3 (3.27) | 1.0 (2.19) | 0.7 (1.37) | 0.5 (1.38) | 0.8 (2.14) | -0.5 (3.08) | 1.3 (2.25) | 0.3 (2.02)
  4.5 hours, n=6,6,6,6,6,6,6,6,16 | 1.8 (1.72) | 0.8 (3.31) | 1.7 (3.20) | 0.8 (1.33) | 0.3 (1.21) | 0.7 (1.63) | 1.0 (1.41) | 0.7 (2.16) | 1.9 (2.31)
  6 hours, n=6,6,6,6,6,6,6,6,16 | 0.7 (1.97) | 0.3 (2.34) | -1.7 (1.86) | 2.3 (2.80) | -0.2 (2.04) | 0.7 (2.73) | 0.5 (1.97) | 1.3 (1.75) | 1.0 (3.35)
  12 hours, n=6,6,6,6,6,6,6,6,16 | 2.2 (2.14) | 2.8 (4.26) | 2.2 (4.36) | 2.7 (2.34) | -1.7 (2.88) | -0.2 (1.33) | 1.3 (2.34) | 1.0 (2.53) | 2.2 (2.59)
  24 hours, n=6,6,6,6,6,6,6,6,16 | 0.7 (1.51) | -0.3 (1.03) | 0.7 (2.80) | 0.3 (2.80) | -2.0 (1.67) | 1.0 (2.61) | -0.2 (0.98) | 1.5 (2.07) | 0.9 (2.66)
  48 hours, n=6,6,6,6,6,6,6,6,16 | 0.7 (1.97) | -0.2 (2.32) | 0.5 (3.08) | 1.2 (2.04) | 0.0 (1.26) | 1.7 (1.21) | 1.7 (1.37) | 0.3 (2.25) | -0.3 (3.15)
  72 hours, n=6,6,6,6,6,6,6,6,16 | 0.2 (1.47) | 0.0 (2.19) | 0.3 (2.58) | 0.7 (3.50) | -0.5 (2.35) | -0.3 (1.97) | -1.5 (2.35) | 0.5 (4.14) | -0.3 (2.73)
  96 hours, n=6,6,6,6,6,6,6,6,15: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 15
  96 hours, n=6,6,6,6,6,6,6,6,15 | 1.3 (1.97) | 0.5 (2.07) | 0.0 (2.00) | -1.0 (2.37) | 0.2 (4.02) | 0.0 (1.26) | -1.0 (2.68) | 0.3 (2.58) | 0.3 (2.37)
  FU (Day 15), n=6,6,6,6,6,6,6,6,15: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 15
  FU (Day 15), n=6,6,6,6,6,6,6,6,15 | 0.2 (2.71) | -0.8 (2.48) | 0.5 (3.27) | 0.0 (2.90) | 0.5 (2.43) | -1.2 (2.64) | -0.5 (1.87) | 1.2 (2.86) | 0.3 (2.74)

20. Primary Outcome: Part 1: Number of Participants With Abnormal Electrocardiogram (ECG) Findings
Description: 12-lead ECGs were measured in a semi-supine position using an automated ECG machine after approximately 5 minutes of rest for the participant. Abnormal findings were categorized as clinically significant (CS) and not clinically significant (NCS).
Time Frame: Baseline (Day 1 predose), 1,2,4,6,12,24,48,72,96 hours post dose and Follow up (Day 15)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK3640254 1 mg | Part 1: GSK3640254 3 mg | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 30mg | Part 1: GSK3640254 100 mg | Part 1: GSK3640254 200 mg | Part 1: GSK3640254 400 mg | Part 1: GSK3640254 700 mg | Part 1: Single Dose Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16
Participants
  CS, Day 1,1 hour n=6,6,6,6,6,6,6,6,16 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CS, Day 1,2 hours, n=6,6,6,6,6,6,6,6,16 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CS, Day 1, 4 hours, n=6,6,6,6,6,6,6,6,16 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CS, Day 1, 6 hours, n=6,6,6,6,6,6,6,6,16 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CS, Day 1, 12 hours, n=6,6,6,6,6,6,6,6,16 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CS, Day 1, 24 hours, n=6,6,6,6,6,6,6,6,16 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CS,Day 1, 48 hours, n=6,6,6,6,6,6,6,6,16 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CS, Day 1, 72 hours, n=6,6,6,6,6,6,6,6,16 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CS, Day 1, 96 hour n=6,6,6,6,6,6,6,6,15: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 15
  CS, Day 1, 96 hour n=6,6,6,6,6,6,6,6,15 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CS, FU (Day 15), n=6,6,6,6,6,6,6,6,16 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  NCS, Day 1,1 hour n=6,6,6,6,6,6,6,6,16 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  NCS, Day 1,2 hours, n=6,6,6,6,6,6,6,6,16 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  NCS, Day 1, 4 hours, n=6,6,6,6,6,6,6,6,16 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  NCS, Day 1, 6 hours, n=6,6,6,6,6,6,6,6,16 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  NCS,Day 1, 12 hours, n=6,6,6,6,6,6,6,6,16 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  NCS, Day 1, 24 hours, n=6,6,6,6,6,6,6,6,16 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  NCS,Day 1, 48 hours n=6,6,6,6,6,6,6,6,16 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
  NCS, Day 1, 72 hours, n=6,6,6,6,6,6,6,6,16 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  NCS, Day 1, 96 hour n=6,6,6,6,6,6,6,6,15: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 15
  NCS, Day 1, 96 hour n=6,6,6,6,6,6,6,6,15 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  NCS, FU (Day 15), n=6,6,6,6,6,6,6,6,16 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1

21. Primary Outcome: Part 2: Number of Participants AEs and SAEs
Description: An AE is any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect or any other situation according to medical or scientific judgment were categorized as SAE. Results are presented treatment wise.
Time Frame: Up to Day 28
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Groups:
- Part 2: GSK3640254 50 mg: Participants received repeated dose of GSK3640254 50 mg once daily up to 14 days
- Part 2: GSK3640254 100 mg: Participants received repeated dose of GSK3640254 100 mg once daily up to 14 days
- Part 2: GSK3640254 200 mg + Expansion: Participants received repeated dose of GSK3640254 200 mg once daily up to 14 days
- Part 2: GSK3640254 320 mg: Participants received repeated dose of GSK3640254 320 mg once daily up to 14 days
Arm/Group | Part 2: GSK3640254 50 mg | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 200 mg + Expansion | Part 2: GSK3640254 320 mg | Part 2: Repeated Dose Placebo
Number analyzed (Participants) | 6 | 6 | 25 | 7 | 14
Participants
  AE | 4 | 5 | 19 | 6 | 10
  SAE | 0 | 0 | 0 | 0 | 0

22. Primary Outcome: Part 2: Change From Baseline in Abnormal Hematology Findings: Basophils, Eosinophils, Leukocytes, Lymphocytes, Monocytes, Neutrophils, Platelets.
Description: Blood samples were collected at indicated time points to analyze the hematology parameters: basophils, eosinophils, leukocytes, lymphocytes, monocytes, neutrophils and platelets. Day -2 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value. Results are presented treatment wise.
Time Frame: Baseline (Day -2), Pre dose on Days 2,4,6,8,10,12,14 Day 14 : 48 and 96 hours post dose, Follow up (Day 28)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: 10^9 cells/Liter
Arm/Group | Part 2: GSK3640254 50 mg | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 200 mg + Expansion | Part 2: GSK3640254 320 mg | Part 2: Repeated Dose Placebo
Number analyzed (Participants) | 6 | 6 | 25 | 7 | 14
10^9 cells/Liter
  Basophils, Day 2, predose, n=6,6,25,7,14 | 0.003 (0.0103) | 0.000 (0.0110) | -0.004 (0.0111) | 0.001 (0.0069) | -0.004 (0.0108)
  Basophils, Day 4, predose, n=6,6,25,7,14 | -0.002 (0.0117) | 0.005 (0.0217) | -0.001 (0.0108) | 0.001 (0.0107) | -0.002 (0.0119)
  Basophils, Day 6, predose, n=6,6,25,7,14 | 0.002 (0.0075) | 0.003 (0.0151) | 0.001 (0.0124) | 0.009 (0.0135) | -0.002 (0.0105)
  Basophils, Day 8 predose, n=6,6,25,7,14 | 0.005 (0.0138) | 0.012 (0.0214) | 0.004 (0.0147) | 0.014 (0.0098) | -0.002 (0.0105)
  Basophils, Day 10, predose, n=6,6,25,7,14 | 0.005 (0.0055) | 0.013 (0.0163) | 0.010 (0.0108) | 0.011 (0.0121) | 0.001 (0.0123)
  Basophils, Day 12, predose, n=6,6,25,7,14 | 0.002 (0.0075) | 0.017 (0.0163) | 0.008 (0.0121) | 0.010 (0.0082) | -0.001 (0.0100)
  Basophils, Day 14, predose, n=6,6,25,6,14: number analyzed (Participants) | 6 | 6 | 25 | 6 | 14
  Basophils, Day 14, predose, n=6,6,25,6,14 | 0.003 (0.0052) | 0.002 (0.0214) | 0.007 (0.0140) | 0.017 (0.0082) | -0.003 (0.0114)
  Basophils, Day 14, 48 hours, n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  Basophils, Day 14, 48 hours, n=6,6,24,6,14 | 0.002 (0.0075) | 0.010 (0.0190) | 0.007 (0.0137) | 0.005 (0.0138) | -0.001 (0.0103)
  Basophils, Day 14, 96 hours, n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  Basophils, Day 14, 96 hours, n=6,6,24,6,14 | 0.002 (0.0075) | 0.010 (0.0228) | 0.004 (0.0110) | 0.007 (0.0121) | -0.004 (0.0165)
  Basophils, FU(Day 28), n=6,6,25,7,14 | -0.007 (0.0103) | 0.003 (0.0137) | -0.003 (0.0124) | -0.001 (0.0069) | -0.006 (0.0150)
  Eosinophils, Day 2, predose, n=6,6,25,7,14 | 0.015 (0.0176) | 0.032 (0.0147) | 0.006 (0.0728) | 0.050 (0.0663) | -0.001 (0.0438)
  Eosinophils, Day 4, predose, n=6,6,25,7,14 | 0.015 (0.0536) | 0.013 (0.0455) | 0.012 (0.0867) | 0.043 (0.0605) | -0.006 (0.0520)
  Eosinophils, Day 6, predose, n=6,6,25,7,14 | 0.043 (0.0665) | 0.007 (0.0528) | 0.000 (0.0876) | 0.034 (0.0832) | 0.000 (0.0411)
  Eosinophils, Day 8 predose, n=6,6,25,7,14 | 0.027 (0.0516) | 0.030 (0.0529) | -0.005 (0.0838) | 0.024 (0.0683) | -0.007 (0.0395)
  Eosinophils, Day 10, predose, n=6,6,25,7,14 | 0.028 (0.0426) | 0.053 (0.0539) | 0.025 (0.1057) | 0.026 (0.0824) | -0.012 (0.0437)
  Eosinophils, Day 12, predose, n=6,6,25,7,14 | 0.008 (0.0768) | 0.067 (0.0472) | 0.021 (0.1075) | 0.033 (0.0862) | -0.012 (0.0519)
  Eosinophils, Day 14, predose, n=6,6,25,6,14: number analyzed (Participants) | 6 | 6 | 25 | 6 | 14
  Eosinophils, Day 14, predose, n=6,6,25,6,14 | 0.017 (0.0602) | 0.013 (0.0468) | 0.019 (0.1192) | 0.048 (0.0794) | 0.011 (0.0589)
  Eosinophils, Day 14, 48 hours, n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  Eosinophils, Day 14, 48 hours, n=6,6,24,6,14 | 0.003 (0.0468) | 0.047 (0.0513) | 0.000 (0.1193) | 0.048 (0.0893) | 0.009 (0.0770)
  Eosinophils, Day 14, 96 hours, n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  Eosinophils, Day 14, 96 hours, n=6,6,24,6,14 | 0.045 (0.0647) | 0.043 (0.0437) | 0.004 (0.1167) | 0.050 (0.0851) | 0.001 (0.0584)
  Eosinophils, FU (Day 28), n=6,6,25,7,14 | -0.055 (0.0373) | 0.017 (0.0659) | -0.003 (0.1617) | 0.023 (0.0804) | -0.041 (0.0618)
  Leukocytes, Day 2, predose, n=6,6,25,7,14 | 0.203 (0.8721) | 0.275 (0.4329) | 0.355 (1.6576) | -0.081 (0.4831) | -0.202 (1.2439)
  Leukocytes, Day 4, predose, n=6,6,25,7,14 | 0.170 (0.8864) | 0.123 (0.5792) | -0.096 (0.9361) | 0.063 (0.9600) | -0.250 (1.3609)
  Leukocytes, Day 6, predose, n=6,6,25,7,14 | 0.158 (1.1274) | 0.052 (0.4839) | 0.100 (1.3054) | -0.347 (0.6065) | -0.026 (1.3748)
  Leukocytes, Day 8 predose, n=6,6,25,7,14 | 0.043 (0.8500) | 0.178 (0.6011) | -0.011 (0.9496) | -0.481 (1.2000) | -0.144 (1.3225)
  Leukocytes, Day 10, predose, n=6,6,25,7,14 | 0.117 (0.8565) | 0.515 (0.4821) | 0.296 (0.8216) | -0.584 (1.1299) | 0.064 (1.5507)
  Leukocytes, Day 12, predose, n=6,6,25,7,14 | 0.538 (1.0626) | 0.810 (0.4692) | 0.165 (0.8511) | -0.567 (1.2112) | -0.052 (1.4813)
  Leukocytes, Day 14, predose, n=6,6,25,6,14: number analyzed (Participants) | 6 | 6 | 25 | 6 | 14
  Leukocytes, Day 14, predose, n=6,6,25,6,14 | 0.200 (0.8402) | -0.053 (0.4230) | 0.180 (1.0249) | -0.433 (0.9609) | 0.046 (1.3461)
  Leukocytes, Day 14, 48 hours, n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  Leukocytes, Day 14, 48 hours, n=6,6,24,6,14 | 0.028 (0.7348) | 0.187 (0.4774) | 0.097 (1.0672) | -0.597 (1.2776) | 0.104 (1.2821)
  Leukocytes, Day 14, 96 hours, n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  Leukocytes, Day 14, 96 hours, n=6,6,24,6,14 | 0.438 (1.0624) | 0.300 (0.4367) | 0.336 (1.1083) | -0.248 (1.6414) | 0.347 (1.3089)
  Leukocytes, FU (Day 28), n=6,6,25,7,14 | -1.148 (0.7008) | 0.263 (1.6261) | -0.209 (0.8990) | -0.709 (1.2790) | -0.049 (1.1939)
  Lymphocytes, Day 2, predose, n=6,6,25,7,14 | 0.003 (0.4892) | 0.092 (0.4111) | 0.013 (0.3249) | 0.163 (0.3174) | -0.026 (0.4478)
  Lymphocytes, Day 4, predose, n=6,6,25,7,14 | -0.008 (0.6814) | -0.067 (0.5230) | 0.000 (0.3242) | 0.194 (0.4500) | -0.003 (0.4739)
  Lymphocytes, Day 6, predose, n=6,6,25,7,14 | -0.035 (0.7416) | -0.017 (0.5384) | 0.147 (0.3174) | 0.210 (0.5157) | 0.112 (0.3739)
  Lymphocytes, Day 8 predose, n=6,6,25,7,14 | -0.035 (0.6427) | 0.100 (0.5655) | 0.140 (0.2862) | 0.229 (0.4557) | 0.013 (0.4660)
  Lymphocytes, Day 10, predose, n=6,6,25,7,14 | 0.053 (0.7320) | 0.185 (0.5404) | 0.232 (0.3580) | 0.190 (0.5199) | 0.085 (0.4055)
  Lymphocytes, Day 12, predose, n=6,6,25,7,14 | 0.177 (0.7096) | 0.332 (0.3874) | 0.180 (0.4106) | 0.231 (0.5225) | 0.054 (0.5013)
  Lymphocytes, Day 14, predose, n=6,6,25,6,14: number analyzed (Participants) | 6 | 6 | 25 | 6 | 14
  Lymphocytes, Day 14, predose, n=6,6,25,6,14 | -0.078 (0.5286) | -0.055 (0.4773) | 0.186 (0.2944) | 0.125 (0.4923) | 0.061 (0.4643)
  Lymphocytes, Day 14, 48 hours, n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  Lymphocytes, Day 14, 48 hours, n=6,6,24,6,14 | -0.022 (0.5561) | 0.135 (0.3746) | 0.180 (0.3403) | 0.072 (0.4776) | 0.044 (0.4554)
  Lymphocytes, Day 14, 96 hours, n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  Lymphocytes, Day 14, 96 hours, n=6,6,24,6,14 | 0.060 (0.5114) | 0.255 (0.4602) | 0.247 (0.3308) | 0.193 (0.7185) | 0.059 (0.4478)
  Lymphocytes, FU (Day 28), n=6,6,25,7,14 | -0.512 (0.5189) | -0.280 (0.5637) | -0.144 (0.4368) | -0.237 (0.3583) | -0.184 (0.2858)
  Monocytes, Day 2, predose, n=6,6,25,7,14 | 0.003 (0.1046) | -0.038 (0.0791) | 0.011 (0.1690) | -0.026 (0.0948) | -0.042 (0.0982)
  Monocytes, Day 4, predose, n=6,6,25,7,14 | -0.023 (0.0804) | -0.037 (0.0905) | -0.001 (0.1085) | -0.023 (0.1052) | -0.029 (0.1018)
  Monocytes, Day 6, predose, n=6,6,25,7,14 | -0.030 (0.1489) | -0.075 (0.0817) | -0.019 (0.1169) | -0.067 (0.0808) | -0.021 (0.1045)
  Monocytes, Day 8 predose, n=6,6,25,7,14 | 0.012 (0.1068) | -0.057 (0.1063) | -0.018 (0.1006) | -0.001 (0.1192) | -0.005 (0.1005)
  Monocytes, Day 10, predose, n=6,6,25,7,14 | 0.003 (0.1204) | 0.020 (0.1115) | 0.016 (0.0881) | -0.021 (0.1122) | -0.001 (0.1356)
  Monocytes, Day 12, predose, n=6,6,25,7,14 | 0.023 (0.0942) | 0.022 (0.1269) | -0.002 (0.0926) | -0.011 (0.1530) | -0.009 (0.1244)
  Monocytes, Day 14, predose, n=6,6,25,6,14: number analyzed (Participants) | 6 | 6 | 25 | 6 | 14
  Monocytes, Day 14, predose, n=6,6,25,6,14 | 0.037 (0.1084) | -0.008 (0.0773) | -0.023 (0.1044) | -0.027 (0.1226) | 0.003 (0.1007)
  Monocytes, Day 14, 48 hours, n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  Monocytes, Day 14, 48 hours, n=6,6,24,6,14 | -0.005 (0.1093) | -0.040 (0.0947) | -0.019 (0.1158) | -0.050 (0.1352) | 0.004 (0.0756)
  Monocytes, Day 14, 96 hours, n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  Monocytes, Day 14, 96 hours, n=6,6,24,6,14 | 0.035 (0.0961) | -0.030 (0.1077) | 0.006 (0.1323) | -0.002 (0.1450) | 0.038 (0.1207)
  Monocytes, FU (Day 28), n=6,6,25,7,14 | -0.083 (0.1037) | -0.030 (0.1188) | -0.036 (0.0937) | 0.013 (0.1883) | -0.051 (0.0778)
  Neutrophils, Day 2, predose, n=6,6,25,7,14 | 0.178 (0.5500) | 0.190 (0.5981) | 0.328 (1.5779) | -0.273 (0.6049) | -0.128 (1.0189)
  Neutrophils, Day 4, predose, n=6,6,25,7,14 | 0.188 (0.3853) | 0.207 (0.3747) | -0.107 (0.8863) | -0.153 (1.0017) | -0.209 (1.0416)
  Neutrophils, Day 6, predose, n=6,6,25,7,14 | 0.177 (0.4173) | 0.135 (0.3031) | -0.030 (1.1214) | -0.533 (0.6285) | -0.114 (1.1418)
  Neutrophils, Day 8 predose, n=6,6,25,7,14 | 0.038 (0.2525) | 0.097 (0.3894) | -0.132 (0.8619) | -0.746 (1.2632) | -0.141 (1.0976)
  Neutrophils, Day 10, predose, n=6,6,25,7,14 | 0.028 (0.1317) | 0.240 (0.3099) | 0.012 (0.8357) | -0.791 (1.1634) | -0.008 (1.3122)
  Neutrophils, Day 12, predose, n=6,6,25,7,14 | 0.328 (0.3414) | 0.373 (0.3690) | -0.042 (0.7593) | -0.831 (1.1224) | -0.083 (1.1305)
  Neutrophils, Day 14, predose, n=6,6,25,6,14: number analyzed (Participants) | 6 | 6 | 25 | 6 | 14
  Neutrophils, Day 14, predose, n=6,6,25,6,14 | 0.222 (0.4540) | -0.007 (0.4620) | -0.011 (0.9244) | -0.598 (0.9450) | -0.026 (1.1249)
  Neutrophils, Day 14, 48 hours, n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  Neutrophils, Day 14, 48 hours, n=6,6,24,6,14 | 0.048 (0.3746) | 0.035 (0.7028) | -0.072 (0.9007) | -0.673 (1.2453) | 0.049 (1.1598)
  Neutrophils, Day 14, 96 hours, n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  Neutrophils, Day 14, 96 hours, n=6,6,24,6,14 | 0.292 (0.5710) | 0.017 (0.5775) | 0.075 (0.9796) | -0.497 (1.0625) | 0.255 (1.1764)
  Neutrophils, FU (Day 28), n=6,6,25,7,14 | -0.490 (0.3072) | 0.555 (1.9413) | -0.024 (0.7404) | -0.509 (1.3465) | 0.235 (1.3115)
  Platelets, Day 2, predose, n=6,5,25,7,14: number analyzed (Participants) | 6 | 5 | 25 | 7 | 14
  Platelets, Day 2, predose, n=6,5,25,7,14 | -0.7 (18.78) | 9.8 (6.94) | 5.4 (13.46) | 17.9 (18.89) | 1.3 (20.45)
  Platelets, Day 4, predose, n=6,5,25,7,14: number analyzed (Participants) | 6 | 5 | 25 | 7 | 14
  Platelets, Day 4, predose, n=6,5,25,7,14 | 2.5 (12.76) | -11.2 (8.23) | 2.5 (16.28) | 17.6 (31.86) | -3.6 (21.81)
  Platelets, Day 6, predose, n=6,6,25,7,14 | 11.2 (20.61) | 10.3 (14.73) | 3.4 (18.67) | 17.1 (13.28) | 3.3 (25.28)
  Platelets, Day 8 predose, n=6,5,25,7,14: number analyzed (Participants) | 6 | 5 | 25 | 7 | 14
  Platelets, Day 8 predose, n=6,5,25,7,14 | 0.8 (8.82) | 4.4 (13.87) | 8.6 (19.14) | 16.7 (21.66) | 0.4 (31.14)
  Platelets, Day 10, predose, n=6,6,25,7,14 | 3.7 (16.38) | 14.7 (11.34) | 8.0 (30.98) | 14.3 (12.38) | 4.8 (31.48)
  Platelets, Day 12, predose, n=6,6,25,7,14 | 4.5 (27.40) | 9.8 (19.02) | 3.6 (34.68) | 6.1 (15.00) | 2.9 (28.62)
  Platelets, Day 14, predose, n=6,6,25,6,14: number analyzed (Participants) | 6 | 6 | 25 | 6 | 14
  Platelets, Day 14, predose, n=6,6,25,6,14 | 5.3 (23.52) | -6.2 (19.30) | 8.3 (25.49) | 7.8 (19.74) | -2.9 (31.90)
  Platelets, Day 14, 48 hours, n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  Platelets, Day 14, 48 hours, n=6,6,24,6,14 | -3.0 (13.73) | -2.8 (13.70) | 1.3 (21.79) | -2.2 (17.99) | -1.1 (34.32)
  Platelets, Day 14, 96 hours, n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  Platelets, Day 14, 96 hours, n=6,6,24,6,14 | -4.3 (9.93) | -3.3 (20.74) | 1.0 (23.54) | -17.3 (33.99) | -5.4 (25.19)
  Platelets, FU (Day 28), n=6,6,25,7,14 | -8.7 (10.75) | -11.8 (20.02) | -3.9 (21.61) | -4.0 (28.3) | -5.3 (39.09)

23. Primary Outcome: Part 2: Change From Baseline in Hematology Parameter: Erythrocytes
Description: Blood samples were collected at indicated time points to analyze the hematology parameters: Erythrocytes. Day -2 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day -2), Pre dose on Days 2,4,6,8,10,12,14 Day 14: 48 and 96 hours post dose, Follow up (Day 28)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: 10^12 cells/Liter
Arm/Group | Part 2: GSK3640254 50 mg | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 200 mg + Expansion | Part 2: GSK3640254 320 mg | Part 2: Repeated Dose Placebo
Number analyzed (Participants) | 6 | 6 | 25 | 7 | 14
10^12 cells/Liter
  Day 2, predose, n=6,6,25,7,14 | 0.135 (0.2601) | 0.200 (0.1411) | 0.128 (0.2539) | 0.440 (0.1458) | 0.131 (0.2100)
  Day 4, predose, n=6,6,25,7,14 | 0.193 (0.2322) | 0.112 (0.1057) | 0.086 (0.2099) | 0.544 (0.1318) | 0.091 (0.1589)
  Day 6, predose, n=6,6,25,7,14 | 0.197 (0.3267) | 0.230 (0.0994) | 0.088 (0.2160) | 0.323 (0.1614) | 0.146 (0.1480)
  Day 8 predose, n=6,6,25,7,14 | 0.035 (0.3056) | 0.272 (0.1685) | 0.088 (0.2352) | 0.327 (0.1940) | 0.115 (0.1816)
  Day 10, predose, n=6,6,25,7,14 | 0.082 (0.3415) | 0.293 (0.2238) | 0.179 (0.1861) | 0.306 (0.1334) | 0.206 (0.1637)
  Day 12, predose, n=6,6,25,7,14 | 0.078 (0.2423) | 0.387 (0.1643) | 0.139 (0.2004) | 0.296 (0.1049) | 0.179 (0.1372)
  Day 14, predose, n=6,6,25,6,14: number analyzed (Participants) | 6 | 6 | 25 | 6 | 14
  Day 14, predose, n=6,6,25,6,14 | 0.017 (0.2243) | 0.037 (0.1394) | 0.031 (0.2429) | 0.385 (0.2288) | 0.005 (0.1931)
  Day 14, 48 hours, n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  Day 14, 48 hours, n=6,6,24,6,14 | -0.002 (0.2416) | 0.177 (0.2253) | 0.109 (0.2116) | 0.323 (0.2219) | 0.182 (0.2198)
  Day 14, 96 hours, n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  Day 14, 96 hours, n=6,6,24,6,14 | 0.042 (0.1597) | 0.215 (0.2095) | 0.068 (0.2039) | 0.327 (0.1159) | 0.156 (0.1938)
  FU (Day 28),n=6,6,25,7,14 | -0.187 (0.1632) | -0.123 (0.1835) | -0.093 (0.2015) | 0.050 (0.2484) | -0.081 (0.2517)

24. Primary Outcome: Part 2: Change From Baseline in Hematology Parameter: Erythrocytes MCV
Description: Blood samples were collected at indicated time points to analyze the hematology parameters: Erythrocyte MCV. Day -2 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day -2), pre dose on Days 2,4,6,8,10,12,14 Day 14: 48 and 96 hours post dose, Follow up (Day 28)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Femtoliter
Arm/Group | Part 2: GSK3640254 50 mg | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 200 mg + Expansion | Part 2: GSK3640254 320 mg | Part 2: Repeated Dose Placebo
Number analyzed (Participants) | 6 | 6 | 25 | 7 | 14
Femtoliter
  Day 2, predose, n=6,6,25,7,14 | -0.20 (0.559) | -0.63 (0.989) | -0.27 (1.223) | -1.13 (1.280) | -0.16 (1.126)
  Day 4, predose, n=6,6,25,7,14 | -0.50 (0.777) | -1.05 (1.009) | -0.18 (1.321) | -0.19 (1.227) | 0.17 (0.675)
  Day 6, predose, n=6,6,25,7,14 | -0.25 (0.683) | 0.10 (1.368) | -0.02 (1.422) | -1.30 (1.390) | 0.62 (1.188)
  Day 8 predose, n=6,6,25,7,14 | 0.03 (0.308) | -0.60 (1.226) | -0.53 (1.390) | -0.67 (1.566) | 0.79 (1.299)
  Day 10, predose, n=6,6,25,7,14 | -0.02 (0.534) | -0.73 (1.025) | -0.70 (1.635) | -0.90 (0.933) | 0.21 (1.278)
  Day 12, predose, n=6,6,25,7,14 | -0.33 (0.838) | -0.55 (1.017) | -0.34 (0.908) | -0.99 (0.747) | 0.16 (1.161)
  Day 14, predose, n=6,6,25,6,14: number analyzed (Participants) | 6 | 6 | 25 | 6 | 14
  Day 14, predose, n=6,6,25,6,14 | -0.73 (0.864) | 0.72 (0.995) | -0.86 (1.693) | -1.92 (1.059) | 0.26 (1.585)
  Day 14, 48 hours, n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  Day 14, 48 hours, n=6,6,24,6,14 | 0.52 (0.560) | -0.40 (1.322) | -0.67 (1.209) | -1.30 (0.629) | 0.01 (1.210)
  Day 14, 96 hours, n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  Day 14, 96 hours, n=6,6,24,6,14 | -0.55 (0.409) | -0.25 (1.122) | -0.53 (1.361) | -0.50 (0.738) | 0.14 (1.329)
  FU (Day 28), n=6,6,25,7,14 | 0.00 (0.678) | 0.63 (0.459) | -0.65 (1.447) | -1.19 (0.832) | 0.61 (1.215)

25. Primary Outcome: Part 2: Change From Baseline in Hematology Parameter: Erythrocytes Mean Corpuscular Hemoglobin (Erythrocyte MCH)
Description: Blood samples were collected at indicated time points to analyze the hematology parameter: Erythrocyte MCH. Day -1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day -2), pre dose on Days 2,4,6,8,10,12,14 Day 14: 48 and 96 hours post dose, Follow up (Day 28)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | Part 2: GSK3640254 50 mg | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 200 mg + Expansion | Part 2: GSK3640254 320 mg | Part 2: Repeated Dose Placebo
Number analyzed (Participants) | 6 | 6 | 25 | 7 | 14
Picograms
  Day 2, predose, n=6,6,25,7,14 | -0.10 (0.443) | -0.35 (0.217) | -0.08 (0.578) | -0.46 (0.670) | -0.14 (0.759)
  Day 4, predose, n=6,6,25,7,14 | -0.32 (0.306) | -0.03 (0.367) | 0.06 (0.607) | -0.40 (0.408) | 0.09 (0.684)
  Day 6, predose, n=6,6,25,7,14 | -0.43 (0.413) | -0.78 (0.172) | 0.06 (0.788) | -0.30 (0.606) | -0.06 (0.677)
  Day 8 predose, n=6,6,25,7,14 | -0.23 (0.602) | -0.55 (0.226) | 0.08 (0.785) | -0.43 (0.577) | 0.21 (0.673)
  Day 10, predose, n=6,6,25,7,14 | -0.22 (0.571) | -0.67 (0.339) | -0.08 (0.573) | -0.26 (0.544) | 0.01 (0.617)
  Day 12, predose, n=6,6,25,7,14 | 0.00 (0.522) | -0.68 (0.248) | 0.00 (0.450) | -0.10 (0.742) | -0.06 (0.557)
  Day 14, predose, n=6,6,25,6,14: number analyzed (Participants) | 6 | 6 | 25 | 6 | 14
  Day 14, predose, n=6,6,25,6,14 | 0.00 (0.310) | -0.72 (0.264) | -0.02 (0.724) | -0.57 (0.728) | -0.04 (0.637)
  Day 14, 48 hours, n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  Day 14, 48 hours, n=6,6,24,6,14 | 0.08 (0.504) | -0.68 (0.293) | -0.12 (0.598) | -0.17 (0.698) | -0.15 (0.557)
  Day 14, 96 hours, n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  Day 14, 96 hours, n=6,6,24,6,14 | -0.25 (0.647) | -0.87 (0.216) | -0.20 (0.520) | -0.65 (0.740) | 0.00 (0.477)
  FU, (Day 28), n=6,6,25,7,14 | 0.03 (0.427) | -0.60 (0.237) | -0.04 (0.644) | -0.36 (0.412) | 0.01 (0.637)

26. Primary Outcome: Part 2: Change From Baseline in Hematology Parameter: Hematocrit
Description: Blood samples were collected at indicated time points to analyze the hematology parameter: hematocrit. Day -2 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value. Results are presented treatment wise.
Time Frame: Baseline (Day -2), pre dose on Days 2,4,6,8,10,12,14 Day 14: 48 and 96 hours post dose, Follow up (Day 28)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Percentage of red blood cells in blood
Arm/Group | Part 2: GSK3640254 50 mg | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 200 mg + Expansion | Part 2: GSK3640254 320 mg | Part 2: Repeated Dose Placebo
Number analyzed (Participants) | 6 | 6 | 25 | 7 | 14
Percentage of red blood cells in blood
  Day 2, predose, n=6,6,25,7,14 | 0.0102 (0.02300) | 0.0140 (0.01425) | 0.0096 (0.01995) | 0.0314 (0.01122) | 0.0108 (0.01712)
  Day 4, predose, n=6,6,25,7,14 | 0.0133 (0.02270) | 0.0043 (0.01154) | 0.0066 (0.01855) | 0.0453 (0.01067) | 0.0085 (0.01459)
  Day 6, predose, n=6,6,25,7,14 | 0.0148 (0.03205) | 0.0202 (0.01304) | 0.0075 (0.01857) | 0.0206 (0.01397) | 0.0155 (0.01108)
  Day 8 predose, n=6,6,25,7,14 | 0.0025 (0.02788) | 0.0203 (0.01250) | 0.0049 (0.01827) | 0.0241 (0.01378) | 0.0137 (0.01431)
  Day 10, predose, n=6,6,25,7,14 | 0.0063 (0.03144) | 0.0217 (0.01697) | 0.0119 (0.02108) | 0.0216 (0.00872) | 0.0191 (0.01466)
  Day 12, predose, n=6,6,25,7,14 | 0.0047 (0.02439) | 0.0302 (0.01396) | 0.0102 (0.01872) | 0.0203 (0.00739) | 0.0159 (0.01201)
  Day 14, predose, n=6,6,25,6,14: number analyzed (Participants) | 6 | 6 | 25 | 6 | 14
  Day 14, predose, n=6,6,25,6,14 | -0.0027 (0.02276) | 0.0070 (0.01053) | -0.0014 (0.02132) | 0.0227 (0.01825) | 0.0019 (0.01499)
  Day 14, 96 hours, n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  Day 14, 96 hours, n=6,6,24,6,14 | 0.0003 (0.01419) | 0.0170 (0.01665) | 0.0032 (0.01808) | 0.0255 (0.01086) | 0.0145 (0.01594)
  Day 14, 48 hours, n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  Day 14, 48 hours, n=6,6,24,6,14 | 0.0018 (0.01969) | 0.0133 (0.01375) | 0.0060 (0.01664) | 0.0212 (0.01734) | 0.0157 (0.01601)
  FU (Day 28), n=6,6,25,7,14 | -0.0158 (0.01587) | -0.0070 (0.01628) | -0.0110 (0.01675) | -0.0013 (0.01739) | -0.0046 (0.02040)

27. Primary Outcome: Part 2: Change From Baseline in Hematology Parameter: Percentage of Reticulocytes
Description: as for outcome 7
Time Frame: Baseline (Day -2), pre dose on Days 2,4,6,8,10,12,14 Day 14: 48 and 96 hours post dose, Follow up (Day 28)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | Part 2: GSK3640254 50 mg | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 200 mg + Expansion | Part 2: GSK3640254 320 mg | Part 2: Repeated Dose Placebo
Number analyzed (Participants) | 6 | 6 | 25 | 7 | 14
10^12 cells per liter
  Day 2, predose, n=6,6,25,7,14 | 0.00093 (0.001204) | -0.00103 (0.001214) | 0.00088 (0.001818) | -0.00037 (0.001190) | 0.00117 (0.001333)
  Day 4, predose, n=6,6,25,7,14 | 0.00215 (0.001099) | -0.00032 (0.001440) | 0.00131 (0.002263) | 0.00124 (0.001996) | 0.00157 (0.001778)
  Day 6, predose, n=6,6,25,7,14 | 0.00232 (0.000999) | 0.00138 (0.001118) | 0.00125 (0.002761) | 0.00106 (0.002192) | 0.00208 (0.001785)
  Day 8 predose, n=6,6,25,7,14 | 0.00173 (0.001143) | 0.00213 (0.000894) | 0.00154 (0.002999) | 0.00031 (0.001780) | 0.00243 (0.002265)
  Day 10, predose, n=6,6,25,7,14 | 0.00203 (0.000804) | 0.00255 (0.001450) | 0.00153 (0.002881) | -0.00023 (0.001186) | 0.00154 (0.002233)
  Day 12, predose, n=6,6,25,7,14 | 0.00220 (0.001075) | 0.00313 (0.001468) | 0.00205 (0.002889) | 0.00007 (0.001643) | 0.00161 (0.002094)
  Day 14, predose, n=6,6,25,6,14: number analyzed (Participants) | 6 | 6 | 25 | 6 | 14
  Day 14, predose, n=6,6,25,6,14 | 0.00287 (0.001810) | 0.00318 (0.000842) | 0.00212 (0.002924) | -0.00015 (0.001621) | 0.00171 (0.002176)
  Day 14, 48 hours, n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  Day 14, 48 hours, n=6,6,24,6,14 | 0.00270 (0.001788) | 0.00295 (0.001524) | 0.00205 (0.003168) | 0.00063 (0.001429) | 0.00184 (0.003189)
  Day 14, 96 hours, n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  Day 14, 96 hours, n=6,6,24,6,14 | 0.00222 (0.001766) | 0.00163 (0.001780) | 0.00195 (0.003251) | 0.00013 (0.001680) | 0.00111 (0.002838)
  FU, (Day 28), n=6,6,25,7,14 | 0.00177 (0.001581) | 0.00212 (0.002369) | 0.00095 (0.003073) | -0.00084 (0.003085) | 0.00104 (0.002853)

28. Primary Outcome: Part 2: Change From Baseline in Hematology Parameter: Hb
Description: Blood samples were collected at indicated time points to analyze the hematology parameter: Hb. Day -2 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day -2), pre dose on Days 2,4,6,8,10,12,14 Day 14: 48 and 96 hours post dose, Follow up (Day 28)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Part 2: GSK3640254 50 mg | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 200 mg + Expansion | Part 2: GSK3640254 320 mg | Part 2: Repeated Dose Placebo
Number analyzed (Participants) | 6 | 6 | 25 | 7 | 14
Grams per liter
  Day 2, predose, n=6,6,25,7,14 | 3.3 (6.28) | 4.3 (4.13) | 3.4 (7.18) | 10.6 (3.31) | 3.4 (5.73)
  Day 4, predose, n=6,6,25,7,14 | 3.8 (5.49) | 3.2 (2.48) | 2.8 (6.28) | 13.9 (3.02) | 3.1 (4.71)
  Day 6, predose, n=6,6,25,7,14 | 3.5 (8.57) | 2.8 (3.19) | 3.0 (5.91) | 7.7 (3.77) | 3.9 (3.87)
  Day 8 predose, n=6,6,25,7,14 | -0.3 (6.95) | 5.3 (5.89) | 3.1 (5.93) | 7.3 (4.31) | 4.2 (5.91)
  Day 10, predose, n=6,6,25,7,14 | 1.2 (8.45) | 5.5 (6.22) | 4.9 (6.56) | 7.7 (3.50) | 6.3 (5.80)
  Day 12, predose, n=6,6,25,7,14 | 2.3 (6.62) | 8.0 (5.83) | 4.1 (5.70) | 8.1 (3.08) | 4.9 (4.10)
  Day 14, predose, n=6,6,25,6,14: number analyzed (Participants) | 6 | 6 | 25 | 6 | 14
  Day 14, predose, n=6,6,25,6,14 | 0.3 (5.20) | -2.5 (4.23) | 0.9 (7.16) | 8.3 (3.33) | 0.2 (6.15)
  Day 14, 48 hours, n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  Day 14, 48 hours, n=6,6,24,6,14 | 0.2 (4.92) | 1.8 (7.39) | 2.8 (6.37) | 8.8 (4.58) | 4.5 (6.42)
  Day 14, 96 hours, n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  Day 14, 96 hours, n=6,6,24,6,14 | -0.2 (3.13) | 2.2 (5.98) | 1.1 (6.52) | 6.5 (2.88) | 4.7 (5.09)
  FU (Day 28), n=6,6,25,7,14 | -5.3 (4.18) | -6.5 (5.82) | -2.9 (5.51) | -0.3 (7.54) | -2.6 (7.42)

29. Primary Outcome: Part 2: Change From Baseline in Chemistry Parameter: ALT, AST,ALP
Description: Blood samples were collected to analyze the chemistry parameter: ALT, AST,ALP. Day -2was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value. Results are presented treatment wise.
Time Frame: Baseline (Day -2), pre dose on Days 2,4,6,8,10,12,14 Day14: 48 and 96 hours post dose, Follow up (Day 28)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | Part 2: GSK3640254 50 mg | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 200 mg + Expansion | Part 2: GSK3640254 320 mg | Part 2: Repeated Dose Placebo
Number analyzed (Participants) | 6 | 6 | 25 | 7 | 14
International units per liter
  ALT, Day 2, predose, n=6,6,25,7,14 | -1.2 (5.08) | 1.0 (4.56) | 0.5 (3.43) | 1.7 (2.63) | -0.4 (3.71)
  ALT, Day 4, predose, n=6,6,25,7,14 | 0.0 (5.44) | -1.3 (6.35) | 1.4 (4.66) | 3.4 (5.32) | 0.3 (4.01)
  ALT, Day 6, predose, n=6,6,25,7,14 | 3.2 (6.55) | -0.2 (7.86) | 0.9 (4.95) | 0.3 (4.07) | 0.9 (7.45)
  ALT, Day 8 predose, n=6,6,25,7,14 | 3.0 (7.62) | -6.4 (9.66) | 1.8 (6.22) | 1.7 (4.68) | -0.4 (7.51)
  ALT, Day 10, predose, n=6,6,25,7,14 | 2.2 (8.04) | 0.8 (11.75) | 3.5 (6.85) | 0.7 (4.89) | 0.4 (11.55)
  ALT, Day 12, predose, n=6,6,25,7,14 | 4.8 (10.85) | 1.8 (13.76) | 1.8 (6.08) | 0.1 (4.49) | -0.4 (14.70)
  ALT, Day 14, predose, n=5,5,25,6,14: number analyzed (Participants) | 5 | 5 | 25 | 6 | 14
  ALT, Day 14, predose, n=5,5,25,6,14 | 1.4 (9.26) | -2.6 (12.97) | 2.6 (6.37) | -1.0 (4.10) | -1.2 (13.45)
  ALT, Day 14, 48 hours, n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  ALT, Day 14, 48 hours, n=6,6,24,6,14 | 5.8 (15.54) | 1.7 (13.69) | 3.7 (6.19) | -0.3 (3.50) | 1.0 (13.94)
  ALT, Day 14, 96 hours, n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  ALT, Day 14, 96 hours, n=6,6,24,6,14 | 6.0 (10.35) | -0.3 (13.34) | 3.9 (6.98) | 1.8 (6.85) | 1.1 (15.54)
  ALT, FU (Day 28), n=6,6,25,7,14 | 2.5 (5.09) | 7.0 (20.39) | 4.6 (9.22) | -1.3 (3.30) | 0.3 (8.41)
  ALP, Day 2, predose, n=6,6,25,7,14 | -0.7 (1.37) | -3.7 (4.97) | -0.9 (4.66) | -0.1 (3.67) | -2.3 (5.74)
  ALP, Day 4, predose, n=6,6,25,7,14 | 3.7 (3.67) | -7.2 (5.23) | 0.3 (5.01) | 1.6 (6.75) | -2.1 (4.31)
  ALP, Day 6, predose, n=6,6,25,7,14 | 3.3 (7.28) | -5.2 (4.62) | 0.3 (5.41) | 0.9 (5.52) | -0.6 (4.88)
  ALP, Day 8 predose, n=6,5,25,7,14: number analyzed (Participants) | 6 | 5 | 25 | 7 | 14
  ALP, Day 8 predose, n=6,5,25,7,14 | 1.0 (4.52) | -4.4 (4.51) | -0.1 (5.33) | -0.4 (7.41) | -1.4 (5.96)
  ALP, Day 10, predose, n=6,6,25,7,14 | 0.8 (4.92) | -6.2 (3.19) | -0.3 (5.53) | -1.0 (8.85) | -1.2 (5.94)
  ALP, Day 12, predose, n=6,6,25,7,14 | -1.2 (3.92) | -5.7 (3.39) | 0.2 (5.80) | -0.1 (11.44) | -1.4 (6.12)
  ALP, Day 14, predose, n=5,5,25,6,14: number analyzed (Participants) | 5 | 5 | 25 | 6 | 14
  ALP, Day 14, predose, n=5,5,25,6,14 | -3.6 (7.13) | -8.8 (6.10) | -2.2 (4.87) | 0.8 (3.19) | -4.2 (6.17)
  ALP, Day 14, 48 hours, n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  ALP, Day 14, 48 hours, n=6,6,24,6,14 | -1.3 (4.93) | -6.0 (4.73) | -1.6 (5.06) | 1.2 (5.53) | -1.5 (6.02)
  ALP, Day 14, 96 hours, n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  ALP, Day 14, 96 hours, n=6,6,24,6,14 | 2.7 (5.13) | -6.8 (6.01) | -1.8 (5.67) | 1.2 (3.31) | -1.3 (6.09)
  ALP, FU (Day 28), n=6,6,25,7,14 | 1.5 (5.75) | -6.2 (5.91) | -2.4 (5.41) | -2.4 (8.36) | -1.9 (7.29)
  AST, Day 2, predose, n=5,6,24,7,14: number analyzed (Participants) | 5 | 6 | 24 | 7 | 14
  AST, Day 2, predose, n=5,6,24,7,14 | -1.4 (3.58) | -1.2 (2.79) | -1.5 (3.51) | -1.3 (4.89) | -2.5 (3.01)
  AST, Day 4, predose, n=5,6,25,7,14: number analyzed (Participants) | 5 | 6 | 25 | 7 | 14
  AST, Day 4, predose, n=5,6,25,7,14 | 0.6 (2.88) | -3.0 (3.10) | -1.4 (4.22) | -2.4 (4.24) | -1.5 (4.29)
  AST, Day 6, predose, n=5,6,25,7,14: number analyzed (Participants) | 5 | 6 | 25 | 7 | 14
  AST, Day 6, predose, n=5,6,25,7,14 | 0.0 (4.18) | -1.3 (3.88) | -1.7 (3.79) | -3.6 (2.94) | -1.9 (5.40)
  AST, Day 8 predose, n=5,5,25,7,14: number analyzed (Participants) | 5 | 5 | 25 | 7 | 14
  AST, Day 8 predose, n=5,5,25,7,14 | 0.6 (4.34) | -6.4 (4.04) | -0.8 (4.64) | -3.1 (4.06) | -1.1 (6.28)
  AST, Day 10, predose, n=5,6,25,7,14: number analyzed (Participants) | 5 | 6 | 25 | 7 | 14
  AST, Day 10, predose, n=5,6,25,7,14 | 0.0 (3.24) | -2.8 (3.60) | -1.6 (4.24) | -3.6 (3.15) | -1.5 (7.62)
  AST, Day 12, predose, n=5,6,25,7,14: number analyzed (Participants) | 5 | 6 | 25 | 7 | 14
  AST, Day 12, predose, n=5,6,25,7,14 | 0.2 (4.32) | -3.3 (5.09) | -2.0 (4.63) | -4.1 (4.38) | -1.6 (7.53)
  AST, Day 14, predose, n=4,5,23,5,12: number analyzed (Participants) | 4 | 5 | 23 | 5 | 12
  AST, Day 14, predose, n=4,5,23,5,12 | 2.8 (3.30) | -5.6 (6.02) | -2.0 (3.42) | -1.6 (5.68) | -2.8 (7.38)
  AST, Day 14, 48 hours, n=5,6,24,6,14: number analyzed (Participants) | 5 | 6 | 24 | 6 | 14
  AST, Day 14, 48 hours, n=5,6,24,6,14 | 0.8 (4.44) | -3.0 (4.69) | -1.8 (3.95) | -3.5 (2.88) | -2.4 (7.67)
  AST, Day 14, 96 hours, n=5,6,24,6,14: number analyzed (Participants) | 5 | 6 | 24 | 6 | 14
  AST, Day 14, 96 hours, n=5,6,24,6,14 | 2.4 (4.22) | -2.8 (4.45) | -2.0 (3.93) | -2.2 (6.43) | -1.2 (9.22)
  AST, FU (Day 28), n=6,6,25,7,14 | 2.0 (6.67) | 2.5 (5.89) | 2.8 (5.75) | 0.6 (6.55) | 0.7 (4.70)

30. Primary Outcome: Part 1: Change From Baseline in Bicarbonate, Calcium, Chloride, Cholesterol, Magnesium, Phosphate, Potassium, Sodium, Urea
Description: Blood samples were collected to analyze the chemistry parameter: bicarbonate, calcium, chloride, magnesium, phosphate, potassium, sodium, urea. Day -2 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day -2), pre dose on Days 2,4,6,8,10,12,14 Day 14: 48 and 96 hours post dose, Follow up (Day 28)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Part 2: GSK3640254 50 mg | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 200 mg + Expansion | Part 2: GSK3640254 320 mg | Part 2: Repeated Dose Placebo
Number analyzed (Participants) | 6 | 6 | 25 | 7 | 14
Millimoles per liter
  Bicarbonate, Day 2, predose, n=6,6,25,7,14 | 0.7 (2.80) | -1.3 (2.07) | 0.2 (2.31) | 1.1 (1.57) | 0.4 (1.95)
  Bicarbonate, Day 4, predose, n=6,6,25,7,14 | 1.8 (1.72) | -3.3 (1.97) | 1.0 (2.23) | 3.1 (3.08) | 2.1 (2.09)
  Bicarbonate, Day 6, predose, n=6,6,25,7,14 | 0.2 (2.40) | -4.5 (1.22) | 1.0 (2.17) | 0.4 (1.81) | 1.8 (1.72)
  Bicarbonate, Day 8 predose, n=6,6,25,7,14 | -0.7 (1.86) | -1.5 (1.87) | 1.0 (1.63) | 1.3 (1.70) | 1.6 (1.91)
  Bicarbonate, Day 10, predose, n=6,6,25,7,14 | -0.5 (2.81) | -0.2 (1.72) | 2.4 (3.29) | 2.0 (1.63) | 2.4 (2.24)
  Bicarbonate, Day 12, predose, n=6,6,25,7,14 | -1.8 (1.60) | -0.5 (1.64) | 1.3 (2.17) | 3.4 (2.82) | 1.6 (1.65)
  Bicarbonate, Day 14, predose, n=6,6,25,6,12: number analyzed (Participants) | 6 | 6 | 25 | 6 | 12
  Bicarbonate, Day 14, predose, n=6,6,25,6,12 | -1.2 (0.98) | -1.2 (1.72) | 0.1 (1.93) | 1.5 (1.05) | 1.0 (1.62)
  Bicarbonate, Day 14, 48 hours, n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  Bicarbonate, Day 14, 48 hours, n=6,6,24,6,14 | 0.2 (1.47) | 0.8 (0.98) | 2.2 (2.30) | 2.5 (3.56) | 3.0 (2.11)
  Bicarbonate, Day 14, 96 hours, n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  Bicarbonate, Day 14, 96 hours, n=6,6,24,6,14 | -1.2 (1.72) | 1.0 (1.67) | 1.7 (1.55) | 4.3 (2.16) | 2.3 (2.05)
  Bicarbonate, FU (Day 28), n=6,6,25,7,14 | 0.3 (2.94) | -1.0 (0.63) | 0.3 (2.50) | 2.3 (2.56) | 0.8 (1.72)
  Calcium, Day 2, predose, n=6,6,25,7,14 | -0.005 (0.0497) | 0.012 (0.0354) | 0.003 (0.0701) | 0.104 (0.0627) | 0.003 (0.0722)
  Calcium, Day 4, predose, n=6,6,25,7,14 | 0.022 (0.0791) | 0.010 (0.0385) | 0.013 (0.0580) | 0.117 (0.0574) | 0.030 (0.0479)
  Calcium, Day 6, predose, n=6,6,25,7,14 | 0.028 (0.1063) | 0.003 (0.0505) | -0.020 (0.0607) | 0.083 (0.0512) | 0.011 (0.0578)
  Calcium, Day 8 predose, n=6,6,25,7,14 | 0.005 (0.0528) | 0.003 (0.0378) | 0.006 (0.0575) | 0.074 (0.0387) | 0.028 (0.0641)
  Calcium, Day 10, predose, n=6,6,25,7,14 | 0.000 (0.0890) | 0.017 (0.0408) | 0.014 (0.0699) | 0.079 (0.0763) | 0.024 (0.0628)
  Calcium, Day 12, predose, n=6,6,25,7,14 | -0.063 (0.0619) | -0.010 (0.0551) | 0.024 (0.0667) | 0.066 (0.0608) | 0.025 (0.0617)
  Calcium, Day 14, predose, n=6,6,25,6,12: number analyzed (Participants) | 6 | 6 | 25 | 6 | 12
  Calcium, Day 14, predose, n=6,6,25,6,12 | -0.063 (0.0779) | -0.034 (0.0404) | -0.015 (0.0843) | 0.028 (0.0512) | 0.008 (0.0715)
  Calcium, Day 14, 48 hours, n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  Calcium, Day 14, 48 hours, n=6,6,24,6,14 | -0.017 (0.0592) | 0.012 (0.0462) | 0.035 (0.0566) | 0.072 (0.0806) | 0.033 (0.0770)
  Calcium, Day 14, 96 hours, n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  Calcium, Day 14, 96 hours, n=6,6,24,6,14 | 0.005 (0.0459) | 0.027 (0.0472) | 0.037 (0.0526) | 0.078 (0.1042) | 0.046 (0.0580)
  Calcium, FU(Day 28), n=6,6,25,7,14 | -0.042 (0.0471) | 0.003 (0.0550) | -0.018 (0.0572) | 0.039 (0.0891) | 0.019 (0.0827)
  Chloride, Day 2, predose, n=6,6,25,7,14 | 0.7 (1.03) | 2.0 (2.10) | 0.4 (1.45) | -0.1 (1.57) | 1.1 (1.98)
  Chloride, Day 4, predose, n=6,6,25,7,14 | 0.7 (1.63) | 2.3 (1.63) | 0.1 (1.72) | 0.0 (2.45) | 0.9 (1.90)
  Chloride, Day 6, predose, n=6,6,25,7,14 | -0.2 (1.17) | 0.7 (1.21) | 0.2 (2.01) | 0.4 (1.40) | 0.4 (2.10)
  Chloride, Day 8 predose, n=6,6,25,7,14 | 0.5 (1.38) | 1.8 (1.33) | -0.2 (1.67) | 1.3 (1.70) | 0.6 (2.14)
  Chloride, Day 10, predose, n=6,6,25,7,14 | 2.0 (1.41) | 1.7 (1.03) | 0.0 (1.99) | 0.7 (2.43) | 0.7 (1.77)
  Chloride, Day 12, predose, n=6,6,25,7,14 | 0.3 (1.75) | 2.0 (1.26) | 0.8 (1.80) | 0.7 (2.29) | 1.3 (2.23)
  Chloride, Day 14, predose, n=6,6,25,6,12: number analyzed (Participants) | 6 | 6 | 25 | 6 | 12
  Chloride, Day 14, predose, n=6,6,25,6,12 | 1.8 (2.14) | 2.2 (1.17) | 0.9 (2.12) | 0.2 (1.47) | 1.0 (2.11)
  Chloride, Day 14, 48 hours, n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  Chloride, Day 14, 48 hours, n=6,6,24,6,14 | 3.2 (1.72) | 1.0 (1.41) | 1.0 (1.76) | 1.0 (2.53) | 1.1 (2.37)
  Chloride, Day 14, 96 hours, n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  Chloride, Day 14, 96 hours, n=6,6,24,6,14 | 1.0 (0.00) | 2.8 (1.33) | 0.6 (1.71) | -0.5 (1.87) | 0.5 (2.21)
  Chloride, FU(Day 28), n=6,6,25,7,14 | 1.3 (1.21) | 0.5 (1.38) | 0.4 (1.55) | 0.3 (2.43) | 0.8 (1.89)
  Magnesium, Day 2, predose, n=6,6,25,7,14 | 0.055 (0.0596) | -0.012 (0.0436) | -0.004 (0.0486) | 0.016 (0.0624) | -0.006 (0.0422)
  Magnesium, Day 4, predose, n=6,6,25,7,14 | 0.063 (0.0472) | -0.027 (0.0520) | 0.005 (0.0415) | 0.027 (0.0577) | 0.007 (0.0347)
  Magnesium, Day 6, predose, n=6,6,25,7,14 | 0.053 (0.0388) | -0.027 (0.0589) | 0.019 (0.0476) | 0.017 (0.0399) | 0.008 (0.0556)
  Magnesium, Day 8 predose, n=6,6,25,7,14 | 0.075 (0.0532) | 0.000 (0.0420) | 0.002 (0.0426) | 0.019 (0.0438) | 0.004 (0.0420)
  Magnesium, Day 10, predose, n=6,6,25,7,14 | 0.047 (0.0543) | -0.003 (0.0361) | 0.018 (0.0472) | 0.017 (0.0390) | 0.000 (0.0566)
  Magnesium, Day 12, predose, n=6,6,25,7,14 | 0.038 (0.0585) | 0.013 (0.0505) | 0.014 (0.0401) | 0.007 (0.0446) | 0.004 (0.0390)
  Magnesium, Day 14, predose, n=5,6,25,6,14: number analyzed (Participants) | 5 | 6 | 25 | 6 | 14
  Magnesium, Day 14, predose, n=5,6,25,6,14 | 0.030 (0.0495) | -0.013 (0.0653) | 0.019 (0.0473) | -0.002 (0.0343) | -0.001 (0.0551)
  Magnesium, Day 14, 48 hours, n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  Magnesium, Day 14, 48 hours, n=6,6,24,6,14 | 0.040 (0.0555) | -0.022 (0.0445) | 0.011 (0.0355) | 0.020 (0.0603) | -0.001 (0.0363)
  Magnesium, Day 14, 96 hours, n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  Magnesium, Day 14, 96 hours, n=6,6,24,6,14 | 0.025 (0.0485) | -0.007 (0.0423) | 0.011 (0.0360) | 0.022 (0.0331) | -0.002 (0.0662)
  Magnesium, FU (Day 28), n=6,6,25,7,14 | 0.037 (0.0509) | -0.027 (0.0589) | 0.001 (0.0387) | -0.003 (0.0415) | -0.009 (0.0469)
  Phosphate, Day 2, predose, n=6,6,25,7,14 | 0.068 (0.1636) | 0.062 (0.0760) | -0.024 (0.1248) | 0.086 (0.1585) | 0.035 (0.2069)
  Phosphate, Day 4, predose, n=6,6,25,7,14 | 0.057 (0.1091) | 0.017 (0.1237) | -0.003 (0.1382) | 0.057 (0.1045) | 0.036 (0.1835)
  Phosphate, Day 6, predose, n=6,6,25,7,14 | 0.100 (0.1324) | 0.038 (0.1080) | -0.014 (0.1375) | 0.164 (0.1018) | 0.060 (0.2119)
  Phosphate, Day 8 predose, n=6,6,25,7,14 | 0.150 (0.1145) | 0.075 (0.1140) | 0.021 (0.1285) | 0.121 (0.1644) | 0.074 (0.2112)
  Phosphate, Day 10, predose, n=6,6,25,7,14 | 0.150 (0.1848) | 0.118 (0.0937) | 0.061 (0.1372) | 0.140 (0.1344) | 0.129 (0.1626)
  Phosphate, Day 12, predose, n=6,6,25,7,14 | 0.155 (0.1428) | 0.090 (0.0827) | 0.085 (0.1704) | 0.193 (0.1329) | 0.139 (0.2000)
  Phosphate, Day 14, predose, n=5,6,25,6,14: number analyzed (Participants) | 5 | 6 | 25 | 6 | 14
  Phosphate, Day 14, predose, n=5,6,25,6,14 | 0.212 (0.1587) | 0.087 (0.1388) | 0.043 (0.1363) | 0.170 (0.1030) | 0.101 (0.2161)
  Phosphate, Day 14, 48 hours, n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  Phosphate, Day 14, 48 hours, n=6,6,24,6,14 | 0.208 (0.1382) | 0.063 (0.1516) | 0.093 (0.1517) | 0.052 (0.1446) | 0.082 (0.1873)
  Phosphate, Day 14, 96 hours, n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  Phosphate, Day 14, 96 hours, n=6,6,24,6,14 | 0.178 (0.1869) | 0.140 (0.1255) | 0.089 (0.1510) | 0.085 (0.1536) | 0.119 (0.2051)
  Phosphate, FU (Day 28), n=6,6,25,7,14 | -0.013 (0.1363) | -0.020 (0.1418) | -0.047 (0.1837) | 0.010 (0.1795) | 0.010 (0.1741)
  Potassium, Day 2, predose, n=6,6,25,7,14 | 0.10 (0.390) | -0.10 (0.190) | 0.12 (0.340) | 0.41 (0.662) | 0.14 (0.203)
  Potassium, Day 4, predose, n=6,6,25,7,14 | 0.28 (0.279) | -0.07 (0.216) | 0.17 (0.369) | 0.20 (0.383) | 0.19 (0.141)
  Potassium, Day 6, predose, n=6,6,25,7,14 | 0.30 (0.529) | 0.12 (0.264) | 0.11 (0.396) | 0.21 (0.285) | 0.06 (0.234)
  Potassium, Day 8 predose, n=6,5,25,7,14: number analyzed (Participants) | 6 | 5 | 25 | 7 | 14
  Potassium, Day 8 predose, n=6,5,25,7,14 | 0.23 (0.216) | -0.06 (0.152) | 0.04 (0.364) | 0.20 (0.374) | 0.17 (0.307)
  Potassium, Day 10, predose, n=6,6,25,7,14 | 0.32 (0.519) | -0.08 (0.194) | 0.06 (0.406) | 0.21 (0.358) | 0.09 (0.138)
  Potassium, Day 12, predose, n=6,6,25,7,14 | 0.38 (0.431) | -0.13 (0.280) | 0.08 (0.384) | 0.17 (0.399) | 0.22 (0.176)
  Potassium, Day 14, predose, n=5,5,24,6,13: number analyzed (Participants) | 5 | 5 | 24 | 6 | 13
  Potassium, Day 14, predose, n=5,5,24,6,13 | -0.12 (0.277) | -0.20 (0.300) | -0.06 (0.388) | -0.05 (0.327) | 0.19 (0.348)
  Potassium, Day 14, 48 hours, n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  Potassium, Day 14, 48 hours, n=6,6,24,6,14 | 0.27 (0.509) | -0.18 (0.204) | 0.07 (0.338) | -0.08 (0.331) | 0.04 (0.214)
  Potassium, Day 14, 96 hours, n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  Potassium, Day 14, 96 hours, n=6,6,24,6,14 | 0.07 (0.333) | -0.13 (0.137) | 0.00 (0.393) | 0.08 (0.172) | 0.13 (0.261)
  Potassium, FU (Day 28), n=6,6,25,7,14 | 0.05 (0.383) | -0.08 (0.160) | -0.06 (0.347) | -0.13 (0.335) | 0.21 (0.530)
  Sodium, Day 2, predose, n=6,6,25,7,14 | 0.2 (1.47) | 1.2 (1.47) | -0.5 (1.48) | -1.1 (1.86) | 0.1 (2.11)
  Sodium, Day 4, predose, n=6,6,25,7,14 | 1.5 (1.87) | 1.5 (1.38) | -0.3 (1.17) | 0.9 (1.77) | 0.8 (1.93)
  Sodium, Day 6, predose, n=6,6,25,7,14 | -0.3 (1.21) | 1.2 (1.17) | -0.7 (1.14) | -0.1 (1.07) | 0.5 (1.70)
  Sodium, Day 8 predose, n=6,6,25,7,14 | 0.5 (1.38) | 1.8 (0.75) | -1.0 (1.15) | 0.4 (1.40) | 0.7 (2.16)
  Sodium, Day 10, predose, n=6,6,25,7,14 | 1.5 (1.22) | 2.8 (0.98) | 0.3 (2.10) | 1.0 (1.63) | 0.9 (2.07)
  Sodium, Day 12, predose, n=6,6,25,7,14 | 1.2 (0.98) | 1.7 (1.03) | 0.2 (1.53) | 0.9 (1.57) | 1.2 (1.89)
  Sodium, Day 14, predose, n=6,6,25,6,14: number analyzed (Participants) | 6 | 6 | 25 | 6 | 14
  Sodium, Day 14, predose, n=6,6,25,6,14 | 0.5 (1.52) | 2.2 (1.17) | -1.1 (1.83) | -0.5 (0.55) | 0.1 (2.34)
  Sodium, Day 14, 48 hours, n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  Sodium, Day 14, 48 hours, n=6,6,24,6,14 | 3.3 (1.75) | 1.0 (0.89) | 0.4 (1.35) | 0.5 (0.84) | 1.3 (2.27)
  Sodium, Day 14, 96 hours, n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  Sodium, Day 14, 96 hours, n=6,6,24,6,14 | 1.5 (1.52) | 2.3 (0.82) | 0.6 (1.59) | 0.3 (1.03) | 1.1 (2.59)
  Sodium, FU(Day 28), n=6,6,25,7,14 | 1.8 (2.48) | 0.8 (1.72) | -0.1 (1.58) | 0.0 (1.73) | 0.9 (2.32)
  Urea, Day 2, predose, n=6,6,25,7,14 | -0.583100 (1.7190989) | -0.383180 (0.8994549) | -0.279888 (1.3039577) | 0.242760 (0.8615469) | -0.221340 (1.0565530)
  Urea, Day 4, predose, n=6,6,25,7,14 | -0.982940 (2.0645229) | -0.616420 (0.8994549) | -0.415834 (1.2169831) | -0.157080 (0.7761282) | -0.535500 (1.2302718)
  Urea, Day 6, predose, n=6,6,25,7,14 | -0.533120 (1.6805969) | -0.566440 (1.0685283) | -0.439824 (1.3090563) | -0.414120 (0.8948673) | -0.606900 (1.0361954)
  Urea, Day 8 predose, n=6,6,25,7,14 | -0.716380 (1.4324888) | -0.982940 (1.2427511) | -0.287885 (1.1923207) | -0.257040 (0.7543661) | -0.249900 (1.2544880)
  Urea, Day 10, predose, n=6,6,25,7,14 | -0.866320 (1.6805969) | -0.066640 (0.8843306) | -0.491803 (1.1108310) | -0.842520 (0.7064873) | -0.207060 (1.4392234)
  Urea, Day 12, predose, n=6,6,25,7,14 | -1.032920 (1.7088970) | -0.466480 (1.1821793) | -0.139944 (1.1809813) | -1.013880 (0.9698843) | -0.399840 (1.2423284)
  Urea, Day 14, predose, n=6,6,25,6,14: number analyzed (Participants) | 6 | 6 | 25 | 6 | 14
  Urea, Day 14, predose, n=6,6,25,6,14 | -1.049580 (1.9204291) | -1.166200 (1.6051804) | -0.399840 (1.2290067) | -0.882980 (0.9192335) | -0.271320 (1.2493792)
  Urea, Day 14, 48 hours, n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  Urea, Day 14, 48 hours, n=6,6,24,6,14 | -0.916300 (1.5165176) | -0.533120 (1.2237107) | -0.703885 (1.1463627) | -0.949620 (1.1991034) | -0.521220 (1.4681527)
  Urea, Day 14, 96 hours, n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  Urea, Day 14, 96 hours, n=6,6,24,6,14 | -0.949620 (1.5674926) | -0.483140 (0.9278887) | -0.749700 (1.1904312) | -0.499800 (0.8387115) | -0.556920 (1.1341178)
  Urea, FU (Day 28), n=6,6,25,7,14 | -0.882980 (1.2603155) | -1.166200 (0.9580876) | -0.411835 (1.0341231) | -0.571200 (0.6208106) | -0.778260 (0.9818953)

31. Primary Outcome: Part 2: Change From Baseline in Cholesterol, HDL Cholesterol, LDL Cholesterol, Triglycerides
Description: Blood samples were collected at indicated time points to analyze the chemistry parameter: cholesterol, HDL cholesterol, LDL cholesterol, triglycerides. Day -2 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value. Results are presented treatment wise.
Time Frame: Baseline (Day -2), Day 8 (pre dose), Day 14 (48 hours) post dose and Follow up (Day 28)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Part 2: GSK3640254 50 mg | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 200 mg + Expansion | Part 2: GSK3640254 320 mg | Part 2: Repeated Dose Placebo
Number analyzed (Participants) | 6 | 6 | 25 | 7 | 14
Millimoles per liter
  Cholesterol, Day 8, (predose) n=5,6,25,7,13: number analyzed (Participants) | 5 | 6 | 25 | 7 | 13
  Cholesterol, Day 8, (predose) n=5,6,25,7,13 | 0.08 (0.192) | 0.07 (0.631) | 0.16 (0.466) | 0.36 (0.369) | 0.38 (0.440)
  Cholesterol, Day 14 (48 hours), n= 6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  Cholesterol, Day 14 (48 hours), n= 6,6,24,6,14 | -0.05 (0.373) | 0.23 (0.589) | 0.23 (0.531) | 0.40 (0.696) | 0.38 (0.647)
  Cholesterol, FU (Day 28), n= 6,6,25,7,14 | -0.28 (0.147) | 0.15 (0.619) | -0.04 (0.461) | -0.29 (0.955) | -0.04 (0.434)
  HDL Cholesterol, Day 8, (predose) n=5,6,25,7,14: number analyzed (Participants) | 5 | 6 | 25 | 7 | 14
  HDL Cholesterol, Day 8, (predose) n=5,6,25,7,14 | -0.03 (0.121) | 0.00 (0.167) | -0.14 (0.235) | -0.13 (0.150) | -0.14 (0.203)
  HDL Cholesterol, Day 14 (48 hours), n= 6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  HDL Cholesterol, Day 14 (48 hours), n= 6,6,24,6,14 | -0.08 (0.075) | -0.10 (0.179) | -0.18 (0.129) | -0.08 (0.194) | -0.20 (0.260)
  HDL Cholesterol, FU (Day 28), n= 6,6,25,7,14 | 0.02 (0.041) | 0.00 (0.179) | -0.12 (0.277) | 0.01 (0.372) | -0.14 (0.195)
  LDL Cholesterol, Day 8, (predose) n=5,6,25,7,13: number analyzed (Participants) | 5 | 6 | 25 | 7 | 13
  LDL Cholesterol, Day 8, (predose) n=5,6,25,7,13 | 0.08 (0.217) | 0.03 (0.463) | 0.27 (0.407) | 0.49 (0.453) | 0.42 (0.420)
  LDL Cholesterol, Day 14 (48 hours), n= 6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  LDL Cholesterol, Day 14 (48 hours), n= 6,6,24,6,14 | -0.03 (0.234) | 0.27 (0.388) | 0.33 (0.442) | 0.33 (0.615) | 0.47 (0.517)
  LDL Cholesterol, FU (Day 28),n= 6,6,25,7,14 | -0.23 (0.216) | 0.12 (0.556) | 0.12 (0.456) | -0.33 (0.565) | 0.06 (0.455)
  Triglycerides, Day 8, (predose) n=5,6,25,7,13: number analyzed (Participants) | 5 | 6 | 25 | 7 | 13
  Triglycerides, Day 8, (predose) n=5,6,25,7,13 | 0.12 (0.492) | 0.07 (0.137) | 0.08 (0.314) | -0.04 (0.424) | 0.22 (0.215)
  Triglycerides, Day 14 (48 hours), n= 6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  Triglycerides, Day 14 (48 hours), n= 6,6,24,6,14 | 0.20 (0.502) | 0.15 (0.266) | 0.18 (0.400) | 0.28 (0.479) | 0.26 (0.285)
  Triglycerides, FU (Day 28), n= 6,6,25,7,14 | -0.12 (0.471) | 0.07 (0.356) | -0.06 (0.349) | 0.06 (0.538) | 0.14 (0.665)

32. Primary Outcome: Part 2: Change From Baseline in Chemistry Parameter: Glucose
Description: Blood samples were collected at indicated time points to analyze the chemistry parameter: glucose . Day -2 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value. Results are presented treatment wise.
Time Frame: Baseline (Day -2), Day 8 (predose), Day 14 (48 hours) post dose and Follow up (Day 28)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Part 2: GSK3640254 50 mg | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 200 mg + Expansion | Part 2: GSK3640254 320 mg | Part 2: Repeated Dose Placebo
Number analyzed (Participants) | 6 | 6 | 25 | 7 | 14
Millimoles per liter
  Day 8, (predose) n=5,6,25,7,13: number analyzed (Participants) | 5 | 6 | 25 | 7 | 13
  Day 8, (predose) n=5,6,25,7,13 | 0.02 (0.550) | 0.20 (0.237) | -0.10 (0.278) | -0.09 (0.398) | -0.12 (0.394)
  Day 14 (48 hours), n= 6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  Day 14 (48 hours), n= 6,6,24,6,14 | 0.15 (0.532) | 0.03 (0.350) | -0.23 (0.275) | 0.00 (0.329) | -0.21 (0.405)
  FU (Day 28), n= 6,6,25,7,14 | 0.05 (0.824) | 0.15 (0.389) | -0.12 (0.375) | 0.20 (0.507) | -0.02 (0.458)

33. Primary Outcome: Part 2: Change From Baseline in Chemistry Parameter: Bilirubin, Creatinine, Direct Bilirubin
Description: as for outcome 13
Time Frame: Baseline (Day -2), pre dose on Days 2,4,6,8,10,12,14 Day 14: 48 and 96 hours post dose, Follow up (Day 28)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Part 2: GSK3640254 50 mg | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 200 mg + Expansion | Part 2: GSK3640254 320 mg | Part 2: Repeated Dose Placebo
Number analyzed (Participants) | 6 | 6 | 25 | 7 | 14
Micromoles per liter
  Bilirubin, Day 2, predose, n=6,6,25,7,14 | -1.3 (1.97) | -0.8 (2.14) | -0.7 (4.03) | -2.6 (2.94) | -0.9 (4.01)
  Bilirubin, Day 4, predose, n=6,6,25,7,14 | -1.5 (2.59) | 0.2 (0.98) | -0.7 (3.53) | 0.3 (1.50) | 0.3 (3.50)
  Bilirubin, Day 6, predose, n=6,6,25,7,14 | -0.8 (1.72) | -2.2 (1.72) | -1.0 (3.67) | -1.1 (3.63) | -0.7 (3.58)
  Bilirubin, Day 8 predose, n=6,6,25,7,14 | -1.7 (2.07) | -0.5 (1.38) | -0.9 (3.73) | -1.3 (3.64) | -0.1 (3.65)
  Bilirubin, Day 10, predose, n=6,6,25,7,14 | -1.8 (2.64) | -0.2 (2.04) | 0.0 (3.52) | -0.6 (4.20) | -0.1 (3.41)
  Bilirubin, Day 12, predose, n=6,6,25,7,14 | -1.8 (1.83) | 0.2 (2.48) | -1.3 (3.31) | -1.4 (3.69) | -1.1 (3.17)
  Bilirubin, Day 14, predose, n=6,6,25,6,14: number analyzed (Participants) | 6 | 6 | 25 | 6 | 14
  Bilirubin, Day 14, predose, n=6,6,25,6,14 | -0.3 (1.37) | -0.3 (1.86) | -1.0 (3.65) | -1.8 (3.54) | -0.4 (3.75)
  Bilirubin, Day 14, 48 hours, n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  Bilirubin, Day 14, 48 hours, n=6,6,24,6,14 | -1.7 (2.07) | 1.2 (2.64) | 0.1 (3.71) | -0.8 (3.60) | 0.0 (3.35)
  Bilirubin, Day 14, 96 hours, n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  Bilirubin, Day 14, 96 hours, n=6,6,24,6,14 | -1.2 (1.17) | 1.0 (1.79) | -0.4 (4.71) | -1.0 (3.74) | 0.2 (4.02)
  Bilirubin, FU (Day 28), n=6,6,25,7,14 | 1.2 (2.04) | 1.8 (2.40) | 2.3 (7.28) | 0.6 (4.35) | -0.1 (3.90)
  Creatinine, Day 2, predose, n=6,6,25,7,14 | 0.7 (2.50) | 8.2 (3.87) | -3.0 (5.30) | 6.1 (8.30) | 0.4 (3.23)
  Creatinine, Day 4, predose, n=6,6,25,7,14 | 4.7 (4.72) | 1.8 (3.43) | 1.9 (6.05) | 3.1 (3.24) | 1.4 (8.90)
  Creatinine, Day 6, predose, n=6,6,25,7,14 | 3.3 (5.72) | 3.3 (4.41) | -2.2 (6.13) | 5.6 (7.23) | 0.5 (7.47)
  Creatinine, Day 8 predose, n=6,6,25,7,14 | 2.7 (7.74) | 13.8 (4.67) | 2.6 (6.31) | 6.9 (6.52) | 3.6 (9.71)
  Creatinine, Day 10, predose, n=6,6,25,7,14 | 5.8 (8.66) | 7.5 (5.39) | 0.8 (6.16) | 6.4 (3.46) | 4.7 (5.80)
  Creatinine, Day 12, predose, n=6,6,25,7,14 | 4.5 (7.29) | 6.8 (5.74) | 2.0 (8.62) | 3.0 (3.96) | 3.6 (7.44)
  Creatinine, Day 14, predose, n=6,6,25,6,14: number analyzed (Participants) | 6 | 6 | 25 | 6 | 14
  Creatinine, Day 14, predose, n=6,6,25,6,14 | -2.3 (3.83) | 1.7 (3.83) | 1.2 (6.31) | 4.3 (5.05) | 3.6 (8.31)
  Creatinine, Day 14, 48 hours, n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  Creatinine, Day 14, 48 hours, n=6,6,24,6,14 | 4.2 (6.88) | 7.8 (5.46) | 1.5 (7.08) | 8.5 (6.83) | 4.0 (7.92)
  Creatinine, Day 14, 96 hours, n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  Creatinine, Day 14, 96 hours, n=6,6,24,6,14 | 6.0 (5.10) | 15.3 (6.53) | 5.5 (8.81) | 10.2 (5.56) | 8.8 (6.22)
  Creatinine, FU (Day 28), n=6,6,25,7,14 | -0.7 (8.91) | 4.5 (4.89) | -0.3 (7.66) | 3.6 (3.55) | 1.7 (5.17)
  Direct Bilirubin, Day 2, predose, n=6,6,25,7,14 | -0.6 (0.55) | 0.0 (1.00) | -0.4 (1.18) | -1.5 (1.73) | -0.5 (1.31)
  Direct Bilirubin, Day 4, predose, n=6,6,25,7,14 | -0.8 (0.45) | -0.3 (0.82) | -0.4 (1.03) | -0.2 (0.41) | 0.0 (0.95)
  Direct Bilirubin, Day 6, predose, n=6,6,25,7,14 | -0.4 (0.55) | -1.0 (0.82) | -0.4 (1.20) | -0.5 (1.22) | -0.3 (1.36)
  Direct Bilirubin, Day 8 predose, n=6,6,25,7,14 | -0.4 (0.89) | 0.2 (1.10) | -0.3 (1.19) | -0.3 (1.03) | -0.3 (1.37)
  Direct Bilirubin, Day 10, predose, n=6,6,25,7,14 | -0.4 (0.89) | 0.0 (1.26) | 0.0 (1.13) | -0.6 (1.52) | -0.3 (1.14)
  Direct Bilirubin, Day 12, predose, n=6,6,25,7,14 | -0.4 (0.55) | -0.4 (1.14) | -0.5 (0.99) | -0.6 (1.52) | -0.4 (1.24)
  Direct Bilirubin, Day 14, predose, n=6,6,25,6,14: number analyzed (Participants) | 6 | 6 | 25 | 6 | 14
  Direct Bilirubin, Day 14, predose, n=6,6,25,6,14 | 0.0 (0.82) | 0.0 (0.82) | -0.4 (1.26) | -2.5 (0.71) | -0.4 (1.43)
  Direct Bilirubin, Day 14, 48 hours, n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  Direct Bilirubin, Day 14, 48 hours, n=6,6,24,6,14 | -0.8 (0.45) | -0.2 (0.98) | -0.2 (1.14) | -0.2 (1.30) | -0.3 (1.30)
  Direct Bilirubin, Day 14, 96 hours, n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  Direct Bilirubin, Day 14, 96 hours, n=6,6,24,6,14 | -0.4 (0.55) | -0.2 (0.84) | -0.2 (1.40) | -0.6 (0.89) | -0.3 (1.48)
  Direct bilirubin, FU (Day 28), n=6,6,25,7,14 | 0.8 (0.84) | 0.3 (1.21) | 0.7 (2.17) | 0.4 (1.52) | 0.2 (1.54)

34. Primary Outcome: Part 2: Change From Baseline in Chemistry Parameter: Protein
Description: Blood samples were collected to analyze the chemistry parameter: Protein. Day -2 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value. Results are presented treatment wise.
Time Frame: Baseline (Day -2), pre dose on Days 2,4,6,8,10,12,14 Day 14: 48 and 96 hours post dose, Follow up (Day 28)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Part 2: GSK3640254 50 mg | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 200 mg + Expansion | Part 2: GSK3640254 320 mg | Part 2: Repeated Dose Placebo
Number analyzed (Participants) | 6 | 6 | 25 | 7 | 14
Grams per liter
  Day 2, predose, n=6,6,25,7,14 | -0.5 (2.35) | -1.0 (2.19) | 0.2 (3.34) | 1.7 (2.14) | -0.9 (3.32)
  Day 4, predose, n=6,6,25,7,14 | 1.5 (3.02) | 0.0 (2.37) | -0.3 (2.78) | 5.9 (3.53) | -0.6 (2.82)
  Day 6, predose, n=6,6,25,7,14 | 0.7 (5.61) | -1.3 (1.75) | -0.1 (2.53) | 2.1 (2.48) | 0.0 (2.86)
  Day 8 predose, n=6,6,25,7,14 | -1.0 (3.03) | -0.8 (2.48) | -0.5 (2.69) | 1.4 (2.15) | 0.1 (2.56)
  Day 10, predose, n=6,6,25,7,14 | -0.5 (4.04) | 0.7 (1.97) | -0.6 (3.12) | 1.7 (1.98) | 0.0 (4.08)
  Day 12, predose, n=6,6,25,7,14 | -2.7 (3.08) | -1.0 (2.45) | -0.3 (2.72) | 2.9 (2.12) | -0.3 (3.36)
  Day 14, predose, n=6,6,25,6,14: number analyzed (Participants) | 6 | 6 | 25 | 6 | 14
  Day 14, predose, n=6,6,25,6,14 | -2.5 (4.32) | -3.5 (1.87) | -2.0 (4.14) | 0.2 (1.94) | -1.8 (3.85)
  Day 14, 48 hours, n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  Day 14, 48 hours, n=6,6,24,6,14 | -2.2 (3.31) | -1.7 (2.50) | -1.8 (3.57) | 2.0 (2.00) | -0.2 (3.79)
  Day 14, 96 hours, n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  Day 14, 96 hours, n=6,6,24,6,14 | 0.0 (2.53) | -0.8 (2.64) | -1.1 (3.90) | 2.7 (2.42) | 0.6 (3.90)
  FU (Day 28), n=6,6,25,7,14 | -1.0 (2.28) | -1.2 (1.94) | -0.5 (3.43) | 0.4 (3.26) | 0.4 (4.05)

35. Primary Outcome: Part 2: Number of Participants With Abnormal Urinalysis
Description: Urine samples were collected analyze the abnormal findings for potential of hydrogen (pH), glucose, protein, blood, ketones, bilirubin, urobilinogen, nitrite, leukocyte esterase by dipstick.
Time Frame: Up to Day 28
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: GSK3640254 50 mg | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 200 mg + Expansion | Part 2: GSK3640254 320 mg | Part 2: Repeated Dose Placebo
Number analyzed (Participants) | 6 | 6 | 25 | 7 | 14
Participants | 0 | 0 | 0 | 0 | 0

36. Primary Outcome: Part 2: Change From Baseline in Vital Signs: SBP and DBP
Description: as for outcome 16
Time Frame: Baseline (Day -1), pre dose on Days 1,2,4,6,8,10,12,and 14 (pre dose and 72 hours) and Follow up (Day 28)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Part 2: GSK3640254 50 mg | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 200 mg + Expansion | Part 2: GSK3640254 320 mg | Part 2: Repeated Dose Placebo
Number analyzed (Participants) | 6 | 6 | 25 | 7 | 14
Millimeters of mercury (mmHg)
  SBP, Day 1, predose, n=6,6,25,7,14 | 0.5 (4.76) | 1.2 (9.87) | -0.5 (4.68) | 2.9 (5.76) | -1.1 (8.48)
  SBP, Day 2, predose, n=6,6,25,7,14 | 0.5 (2.88) | 1.0 (10.30) | 0.6 (6.47) | 2.6 (3.40) | -2.6 (7.84)
  SBP, Day 4, predose, n=6,6,25,7,14 | -0.3 (5.79) | -0.5 (9.20) | -2.2 (6.33) | 3.0 (5.42) | -3.3 (12.67)
  SBP, Day 6, predose, n=6,6,25,7,14 | -2.7 (5.09) | 1.2 (9.87) | 0.0 (5.72) | 3.0 (7.48) | -1.2 (12.94)
  SBP, Day 8, predose, n=6,6,25,7,14 | -2.5 (3.73) | 3.3 (9.85) | -1.4 (6.19) | 4.3 (5.65) | -1.4 (11.80)
  SBP, Day 10, predose, n=6,6,25,7,14 | -2.8 (3.06) | 0.8 (9.37) | -1.9 (6.66) | 3.7 (4.11) | -5.2 (12.77)
  SBP, Day 12, predose, n=6,6,25,7,14 | -2.8 (2.64) | 0.8 (10.15) | -2.0 (5.70) | 3.3 (5.71) | -4.6 (11.88)
  SBP, Day 14, predose, n=6,6,25,7,14 | -0.8 (3.97) | 0.3 (14.00) | -1.3 (7.31) | 3.8 (5.56) | -4.1 (12.33)
  SBP, Day 14, 72 hours, n=6,6,25,7,14 | 1.3 (3.33) | 0.2 (10.98) | -2.3 (6.21) | 0.2 (6.85) | -2.0 (11.07)
  SBP, follow up, n=6,6,25,7,14 | -3.0 (8.56) | 1.3 (1.75) | 0.8 (6.43) | 4.1 (7.60) | 1.2 (7.03)
  DBP, Day 1, predose, n=6,6,25,7,14 | -2.7 (5.65) | -0.4 (2.76) | -0.9 (5.78) | 2.3 (5.41) | -0.8 (5.73)
  DBP, Day 2, predose, n=6,6,25,7,14 | -1.0 (3.03) | -0.3 (5.20) | 0.9 (6.93) | 2.2 (4.28) | 0.8 (4.76)
  DBP, Day 4, predose, n=6,6,25,7,14 | -2.7 (5.85) | -0.3 (5.68) | -1.6 (7.18) | 3.1 (3.80) | -1.3 (4.94)
  DBP, Day 6, predose, n=6,6,25,7,14 | -4.7 (7.17) | 2.0 (2.19) | 0.2 (5.21) | 1.9 (4.06) | -1.6 (4.62)
  DBP, Day 8, predose, n=6,6,25,7,14 | -2.5 (7.89) | 0.5 (3.73) | -1.3 (6.52) | 0.1 (4.63) | 0.3 (4.70)
  DBP, Day 10, predose, n=6,6,25,7,14 | -3.2 (6.27) | 0.8 (4.71) | -1.2 (5.79) | 3.3 (4.96) | -2.1 (7.13)
  DBP, Day 12, n=6,6,25,7,14 | 0.7 (1.86) | 0.5 (4.85) | -1.9 (6.16) | 0.9 (5.01) | -2.3 (7.45)
  DBP, Day 14, predose, n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  DBP, Day 14, predose, n=6,6,24,6,14 | 0.2 (3.13) | -0.8 (2.56) | -1.0 (6.93) | 0.8 (3.76) | -1.9 (7.07)
  DBP, Day 14, 72 hours n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  DBP, Day 14, 72 hours n=6,6,24,6,14 | -0.3 (2.88) | -1.7 (2.42) | -2.0 (6.03) | -1.2 (4.67) | -1.6 (4.50)
  DBP, FU (Day 28), n=6,6,25,7,14 | -3.0 (8.56) | 1.3 (1.75) | 0.8 (6.43) | 7 (4.1) | 1.2 (7.03)

37. Primary Outcome: Part 2: Change From Baseline in Vital Sign: Pulse Rate
Description: Pulse rate was measured in semi-supine position after 5 minutes rest for the participants at indicated time points. Day -1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day -1), pre dose on Days 1,2,4,6,8,10,12, and 14 (pre dose and 72 hours) and Follow up (Day 28)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Part 2: GSK3640254 50 mg | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 200 mg + Expansion | Part 2: GSK3640254 320 mg | Part 2: Repeated Dose Placebo
Number analyzed (Participants) | 6 | 6 | 25 | 7 | 14
Beats per minute
  Day 1, predose, n=6,6,25,7,14 | -0.3 (4.27) | 0.6 (1.86) | 1.6 (4.98) | -3.4 (3.31) | 5.3 (5.61)
  Day 2, predose, n=6,6,25,7,14 | 0.3 (4.18) | 0.5 (4.93) | 2.5 (7.22) | 2.1 (5.79) | 3.1 (5.66)
  Day 4, predose, n=6,6,25,7,14 | 1.5 (3.27) | 1.5 (5.96) | 0.2 (6.17) | 2.7 (7.63) | 4.1 (6.34)
  Day 6, predose, n=6,6,25,7,14 | 3.8 (3.60) | 2.5 (5.47) | 0.8 (6.55) | 3.4 (4.43) | 3.2 (7.16)
  Day 8, predose, n=6,6,25,7,14 | -0.5 (3.94) | 1.3 (4.89) | 1.4 (8.02) | 2.7 (6.70) | 2.1 (5.34)
  Day 10, predose, n=6,6,25,7,14 | 0.5 (3.94) | 3.3 (5.79) | 1.0 (7.21) | 0.4 (5.62) | 1.8 (6.93)
  Day 12, predose, n=6,6,25,7,14 | 3.5 (4.51) | 2.5 (7.87) | -0.1 (8.02) | 3.1 (10.64) | 2.5 (8.12)
  Day 14, predose, n=6,6,25,6,14: number analyzed (Participants) | 6 | 6 | 25 | 6 | 14
  Day 14, predose, n=6,6,25,6,14 | 3.5 (3.62) | -0.2 (5.12) | -0.2 (7.40) | 1.5 (3.83) | 0.3 (4.61)
  Day 14, 72 hours, n=6,6,25,6,14: number analyzed (Participants) | 6 | 6 | 25 | 6 | 14
  Day 14, 72 hours, n=6,6,25,6,14 | 7.0 (7.62) | 1.8 (4.40) | 2.9 (6.91) | 4.2 (4.31) | 5.0 (6.82)
  FU (Day 28), n=6,6,25,7,14 | 6.3 (6.62) | -1.3 (10.63) | 0.8 (9.36) | 9.6 (7.96) | 6.3 (7.33)

38. Primary Outcome: Part 2: Change From Baseline in Vital Sign: Temperature
Description: as for outcome 18
Time Frame: Baseline (Day -1), pre dose on Days 1,2,4,6,8,10,12, and 14 (pre dose and 72 hours) and Follow up (Day 28)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | Part 2: GSK3640254 50 mg | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 200 mg + Expansion | Part 2: GSK3640254 320 mg | Part 2: Repeated Dose Placebo
Number analyzed (Participants) | 6 | 6 | 25 | 7 | 14
Degree Celsius
  Day 1, predose, n=6,6,25,7,14 | 0.38 (0.313) | 0.08 (0.222) | 0.11 (0.414) | 0.11 (0.308) | 0.09 (0.276)
  Day 2, predose, n=6,6,25,7,14 | 0.25 (0.281) | 0.18 (0.331) | -0.04 (0.507) | -0.11 (0.279) | 0.14 (0.367)
  Day 4, predose, n=6,6,25,7,14 | 0.44 (0.512) | 0.28 (0.271) | 0.04 (0.425) | 0.11 (0.204) | 0.14 (0.374)
  Day 6, predose, n=6,6,25,7,14 | 0.33 (0.489) | 0.25 (0.226) | -0.04 (0.342) | -0.11 (0.491) | 0.14 (0.405)
  Day 8, predose, n=6,6,25,7,14 | 0.05 (0.373) | 0.20 (0.322) | 0.05 (0.255) | -0.09 (0.372) | -0.02 (0.379)
  Day 10, predose, n=6,6,25,7,14 | 0.30 (0.498) | 0.10 (0.593) | -0.01 (0.355) | -0.10 (0.289) | 0.09 (0.455)
  Day 12, predose, n=6,6,25,7,14 | 0.23 (0.489) | 0.23 (0.314) | -0.02 (0.415) | 0.03 (0.320) | 0.06 (0.393)
  Day 14, predose, n=6,6,25,6,14: number analyzed (Participants) | 6 | 6 | 25 | 6 | 14
  Day 14, predose, n=6,6,25,6,14 | 0.30 (0.290) | 0.13 (0.258) | 0.05 (0.309) | 0.05 (0.266) | -0.02 (0.395)
  Day 14, 72 hours, n=6,6,25,6,14: number analyzed (Participants) | 6 | 6 | 25 | 6 | 14
  Day 14, 72 hours, n=6,6,25,6,14 | 0.30 (0.310) | 0.15 (0.302) | 0.06 (0.330) | 0.22 (0.256) | 0.06 (0.363)
  FU (Day 28), n=6,6,25,7,14 | 0.42 (0.264) | 0.37 (0.441) | 0.04 (0.586) | 0.23 (0.364) | 0.21 (0.317)

39. Primary Outcome: Part 2: Change From Baseline in Vital Sign: Respiratory Rate
Description: as for outcome 19
Time Frame: Baseline (Day -1), pre dose on Days 1,2,4,6,8,10,12 and 14 (pre dose and 72 hours) and Follow up (Day 28)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Part 2: GSK3640254 50 mg | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 200 mg + Expansion | Part 2: GSK3640254 320 mg | Part 2: Repeated Dose Placebo
Number analyzed (Participants) | 6 | 6 | 25 | 7 | 14
Breaths per minute
  Day 1, predose, n=6,6,25,7,14 | -1.0 (2.37) | 2.2 (3.49) | 0.2 (2.15) | 0.1 (2.27) | 0.8 (2.22)
  Day 2, predose, n=6,6,25,7,14 | -0.5 (2.88) | 2.3 (1.21) | 0.4 (2.00) | 1.6 (1.72) | 0.5 (1.95)
  Day 4, predose, n=6,6,25,7,14 | -0.5 (2.17) | 2.2 (1.94) | -0.2 (1.50) | 0.6 (2.44) | 0.2 (1.53)
  Day 6, predose, n=6,6,25,7,14 | 0.7 (2.25) | 0.2 (1.47) | 0.1 (1.73) | 0.0 (1.91) | -0.4 (1.65)
  Day 8, predose, n=6,6,25,7,14 | -1.2 (3.06) | 1.7 (1.03) | 0.0 (2.37) | 0.6 (1.90) | 0.5 (1.91)
  Day 10, predose, n=6,6,25,7,14 | -0.3 (3.20) | 1.5 (2.35) | 0.9 (1.69) | 0.6 (0.98) | 0.5 (1.74)
  Day 12, predose, n=6,6,25,7,14 | -0.7 (2.25) | 2.3 (2.80) | 0.4 (1.96) | -0.1 (1.35) | 0.4 (2.62)
  Day 14, predose, n=6,6,25,6,14: number analyzed (Participants) | 6 | 6 | 25 | 6 | 14
  Day 14, predose, n=6,6,25,6,14 | -0.8 (2.14) | 2.7 (1.51) | 0.6 (1.98) | -0.2 (2.23) | 0.4 (2.24)
  Day 14, 72 hours, n=6,6,25,6,14: number analyzed (Participants) | 6 | 6 | 25 | 6 | 14
  Day 14, 72 hours, n=6,6,25,6,14 | -1.0 (1.41) | 2.7 (1.63) | 0.5 (1.56) | -0.5 (1.97) | -0.4 (1.98)
  FU (Day 28), n=6,6,25,7,14 | -0.5 (2.95) | 0.8 (1.72) | 1.1 (2.38) | 0.1 (0.69) | 0.6 (2.10)

40. Primary Outcome: Part 2: Number of Participants With Abnormal ECG Findings
Description: 12-lead ECG were obtained at given time points. Abnormal findings were categorized as clinically significant (CS) and not clinically significant (NCS).Results are presented treatment wise.
Time Frame: Day 1 (0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4.5, 5, 5.5, 6, 8, 12, 24 hours); Pre-dose on Days 3, 4, 6, 8, 10, 12; Day 14: Pre-dose, 1, 2, 4.5, 5, 6, 12, 24, 48, 72 and 96 hours post-dose and follow up (Day 28)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: GSK3640254 50 mg | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 200 mg + Expansion | Part 2: GSK3640254 320 mg | Part 2: Repeated Dose Placebo
Number analyzed (Participants) | 6 | 6 | 25 | 7 | 14
Participants
  CS, Day 1, 0.5 hours, n=4,0,0,0,2: number analyzed (Participants) | 4 | 0 | 0 | 0 | 2
  CS, Day 1, 0.5 hours, n=4,0,0,0,2 | 0 |  |  |  | 0
  CS, Day 1,1 hour, n=6,6,25,7,14 | 0 | 0 | 0 | 0 | 0
  CS, Day 1, 1.5 hours, n=4,0,0,0,1: number analyzed (Participants) | 4 | 0 | 0 | 0 | 1
  CS, Day 1, 1.5 hours, n=4,0,0,0,1 | 0 |  |  |  | 0
  CS,Day 1, 2hours, n=6,6,25,7,14 | 0 | 0 | 0 | 0 | 0
  CS,Day 1, 2.5 hours, n=4,0,0,0,1: number analyzed (Participants) | 4 | 0 | 0 | 0 | 1
  CS,Day 1, 2.5 hours, n=4,0,0,0,1 | 0 |  |  |  | 0
  CS, Day 1, 3 hours n=4,0,0,0,1: number analyzed (Participants) | 4 | 0 | 0 | 0 | 1
  CS, Day 1, 3 hours n=4,0,0,0,1 | 0 |  |  |  | 0
  CS,Day 1, 3.5 hours, n=4,0,0,0,1: number analyzed (Participants) | 4 | 0 | 0 | 0 | 1
  CS,Day 1, 3.5 hours, n=4,0,0,0,1 | 0 |  |  |  | 0
  CS, Day 1, 4.5 hours, n=6,6,25,7,14 | 0 | 0 | 0 | 0 | 0
  CS, Day 1, 5hours, n=4,0,0,0,1: number analyzed (Participants) | 4 | 0 | 0 | 0 | 1
  CS, Day 1, 5hours, n=4,0,0,0,1 | 0 |  |  |  | 0
  CS, Day 1,5.5 hours, n=4,0,0,0,1: number analyzed (Participants) | 4 | 0 | 0 | 0 | 1
  CS, Day 1,5.5 hours, n=4,0,0,0,1 | 0 |  |  |  | 0
  CS,Day 1, 6hours, n=6,6,25,7,14 | 0 | 0 | 0 | 0 | 0
  CS,Day 1, 8 hours, n=4,0,0,0,1: number analyzed (Participants) | 4 | 0 | 0 | 0 | 1
  CS,Day 1, 8 hours, n=4,0,0,0,1 | 0 |  |  |  | 0
  CS, Day 1, 12 hours, n=6,6,25,7,14 | 0 | 0 | 0 | 0 | 0
  CS, Day 1, 24 hours, n=6,6,25,7,14 | 0 | 0 | 0 | 0 | 0
  CS,Day 3, Predose, n=6,6,25,7,14 | 0 | 0 | 0 | 0 | 0
  CS,Day 4, Predose, n=6,6,25,7,14 | 0 | 0 | 0 | 0 | 0
  CS,Day 6, Predose, n=6,6,25,7,14 | 0 | 0 | 0 | 0 | 0
  CS,Day 8, Predose, n=6,6,25,7,14 | 0 | 0 | 0 | 0 | 0
  CS,Day 10, Predose, n=6,6,25,7,14 | 0 | 0 | 0 | 0 | 0
  CS,Day 12, Predose, n=6,6,25,7,14 | 0 | 0 | 0 | 0 | 0
  CS,Day 14, Predose, n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  CS,Day 14, Predose, n=6,6,24,6,14 | 0 | 0 | 0 | 0 | 0
  CS, Day 14, 1hour, n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  CS, Day 14, 1hour, n=6,6,24,6,14 | 0 | 0 | 0 | 0 | 0
  CS,Day 14, 2 hours, n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  CS,Day 14, 2 hours, n=6,6,24,6,14 | 0 | 0 | 0 | 0 | 0
  CS,Day 14, 4.5hours, n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  CS,Day 14, 4.5hours, n=6,6,24,6,14 | 0 | 0 | 0 | 0 | 0
  CS,Day 14, 5hours, n=0,0,0,0,1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1
  CS,Day 14, 5hours, n=0,0,0,0,1 |  |  |  |  | 0
  CS,Day 14, 6 hours, n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  CS,Day 14, 6 hours, n=6,6,24,6,14 | 0 | 0 | 0 | 0 | 0
  CS,Day 14, 12 hours, n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  CS,Day 14, 12 hours, n=6,6,24,6,14 | 0 | 0 | 0 | 0 | 0
  CS,Day 14, 24 hours, n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  CS,Day 14, 24 hours, n=6,6,24,6,14 | 0 | 0 | 0 | 0 | 0
  CS,Day 14, 48 hours, n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  CS,Day 14, 48 hours, n=6,6,24,6,14 | 0 | 0 | 0 | 0 | 0
  CS,Day 14, 72 hours, n=6,6,24, 6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  CS,Day 14, 72 hours, n=6,6,24, 6,14 | 0 | 0 | 0 | 0 | 0
  CS,Day 14, 96 hours, n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  CS,Day 14, 96 hours, n=6,6,24,6,14 | 0 | 0 | 0 | 0 | 0
  CS, FU (Day 28), n=6,6,25,7,14 | 0 | 0 | 0 | 0 | 0
  NCS, Day 1,0.5 hours, n=4,0,0,0,2: number analyzed (Participants) | 4 | 0 | 0 | 0 | 2
  NCS, Day 1,0.5 hours, n=4,0,0,0,2 | 1 |  |  |  | 0
  NCS, Day 1,1 hour, n=6,6,25,7,14 | 0 | 0 | 0 | 0 | 1
  NCS, Day 1, 1.5 hours, n=4,0,0,0,1: number analyzed (Participants) | 4 | 0 | 0 | 0 | 1
  NCS, Day 1, 1.5 hours, n=4,0,0,0,1 | 1 |  |  |  | 0
  NCS,Day 1, 2hours, n=6,6,25,7,14 | 0 | 0 | 2 | 0 | 0
  NCS,Day 1, 2.5 hours, n=4,0,0,0,1: number analyzed (Participants) | 4 | 0 | 0 | 0 | 1
  NCS,Day 1, 2.5 hours, n=4,0,0,0,1 | 0 |  |  |  | 0
  NCS Day 1, 3 hours n=4,0,0,0,1: number analyzed (Participants) | 4 | 0 | 0 | 0 | 1
  NCS Day 1, 3 hours n=4,0,0,0,1 | 0 | 0 | 0 | 0 | 0
  NCS,Day 1, 3.5 hours, n=4,0,0,0,1: number analyzed (Participants) | 4 | 0 | 0 | 0 | 1
  NCS,Day 1, 3.5 hours, n=4,0,0,0,1 | 0 |  |  |  | 0
  NCS, Day 1, 4.5 hours, n=6,6,25,7,14 | 0 | 0 | 1 | 1 | 0
  NCS, Day 1, 5hours n=4,0,0,0,1: number analyzed (Participants) | 4 | 0 | 0 | 0 | 1
  NCS, Day 1, 5hours n=4,0,0,0,1 | 0 |  |  |  | 0
  NCS, Day 1,5.5 hours, n=4,0,0,0,1: number analyzed (Participants) | 4 | 0 | 0 | 0 | 1
  NCS, Day 1,5.5 hours, n=4,0,0,0,1 | 0 | 0 | 0 | 0 | 0
  NCS,Day 1, 6hours, n=6,6,25,7,14 | 0 | 0 | 2 | 0 | 0
  NCS,Day 1, 8 hours, n=4,0,0,0,1: number analyzed (Participants) | 4 | 0 | 0 | 0 | 1
  NCS,Day 1, 8 hours, n=4,0,0,0,1 | 0 |  |  |  | 0
  NCS, Day 1, 12 hours, n=6,6,25,7,14 | 0 | 0 | 0 | 0 | 0
  NCS,Day 3, Predose, n=6,6,25,7,14 | 0 | 1 | 1 | 0 | 0
  NCS,Day 4, Predose, n=6,6,25,7,14 | 0 | 0 | 1 | 1 | 0
  NCS,Day 6, Predose, n=6,6,25,7,14 | 0 | 0 | 2 | 0 | 1
  NCS,Day 8, Predose, n=6,6,25,7,14 | 1 | 0 | 1 | 0 | 0
  NCS,Day 10, Predose, n=6,6,25,7,14 | 0 | 0 | 0 | 0 | 1
  NCS,Day 12, Predose, n=6,6,25,7,14 | 0 | 0 | 1 | 0 | 1
  NCS,Day 14, Predose, n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  NCS,Day 14, Predose, n=6,6,24,6,14 | 1 | 0 | 1 | 0 | 0
  NCS, Day 14, 1hour, n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  NCS, Day 14, 1hour, n=6,6,24,6,14 | 1 | 0 | 0 | 0 | 1
  NCS,Day 14, 2 hours, n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  NCS,Day 14, 2 hours, n=6,6,24,6,14 | 1 | 0 | 0 | 0 | 1
  NCS,Day 14, 4.5 hours, n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  NCS,Day 14, 4.5 hours, n=6,6,24,6,14 | 0 | 0 | 0 | 0 | 0
  NCS,Day 14, 5hours, n=0,0,0,0,1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1
  NCS,Day 14, 5hours, n=0,0,0,0,1 |  |  |  |  | 0
  NCS, Day 14, 6 hours, n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  NCS, Day 14, 6 hours, n=6,6,24,6,14 | 0 | 0 | 1 | 0 | 1
  NCS,Day 14, 12 hours, n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  NCS,Day 14, 12 hours, n=6,6,24,6,14 | 0 | 0 | 2 | 0 | 0
  NCS,Day 14, 24hours, n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  NCS,Day 14, 24hours, n=6,6,24,6,14 | 1 | 0 | 1 | 0 | 0
  NCS,Day 14, 48 hours, n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  NCS,Day 14, 48 hours, n=6,6,24,6,14 | 1 | 0 | 3 | 0 | 1
  NCS,Day 14, 72 hours, n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  NCS,Day 14, 72 hours, n=6,6,24,6,14 | 1 | 0 | 1 | 0 | 1
  NCS,Day 14, 96 hours, n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  NCS,Day 14, 96 hours, n=6,6,24,6,14 | 0 | 0 | 1 | 0 | 2
  NCS, FU (Day 28), n=6,6,24,6,14: number analyzed (Participants) | 6 | 6 | 24 | 6 | 14
  NCS, FU (Day 28), n=6,6,24,6,14 | 0 | 1 | 2 | 0 | 0

41. Secondary Outcome: Part 1: Area Under the Plasma Concentration Time Curve (AUC) From Zero to 24 Hour (AUC[0-24]) of GSK3640254
Description: Blood samples were collected at indicated time points and PK analysis was performed. PK parameters were determined by non-compartmental methods with Phoenix WinNonlin. Results are presented treatment wise.
Time Frame: Pre-dose and 0.5,1,1.5,2,2.5,3,3.5,4,4.5,5,6,8,12,24 hours post-dose
Population: PK Population. The PK Population include all participants who undergo plasma PK sampling and have evaluable PK parameters estimated during the single dose phase of the study Part 1. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: Hour*microgram per milliliter
Arm/Group | Part 1: GSK3640254 1 mg | Part 1: GSK3640254 3 mg | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 30mg | Part 1: GSK3640254 100 mg | Part 1: GSK3640254 200 mg | Part 1: GSK3640254 400 mg | Part 1: GSK3640254 700 mg
Number analyzed (Participants) | 4 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Hour*microgram per milliliter | 0.056 [0.030 to 0.103] | 0.171 [0.126 to 0.231] | 0.576 [0.454 to 0.730] | 1.546 [1.178 to 2.028] | 4.177 [2.161 to 8.074] | 7.334 [5.415 to 9.933] | 21.666 [12.599 to 37.259] | 20.743 [13.296 to 32.362]

42. Secondary Outcome: Part 1: AUC From Zero to Time of Last Sample Taken (AUC[0-Tlast]) of GSK3640254
Description: as for outcome 41
Time Frame: Pre-dose and 0.5,1,1.5,2,2.5,3,3.5,4,4.5,5,6,8,12, 24, 48, 72 and 96 hours post-dose
Population: PK Population. The PK Population include all participants who undergo plasma PK sampling and have evaluable PK parameters estimated during the single dose phase of the study Part 1.
Measure: Geometric Mean (95% Confidence Interval); unit: Hour*microgram per milliliter
Arm/Group | Part 1: GSK3640254 1 mg | Part 1: GSK3640254 3 mg | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 30mg | Part 1: GSK3640254 100 mg | Part 1: GSK3640254 200 mg | Part 1: GSK3640254 400 mg | Part 1: GSK3640254 700 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Hour*microgram per milliliter | 0.020 [0.005 to 0.080] | 0.184 [0.120 to 0.282] | 1.082 [0.875 to 1.338] | 2.816 [2.148 to 3.692] | 8.060 [4.228 to 15.367] | 14.068 [9.545 to 20.735] | 40.238 [24.234 to 66.812] | 37.626 [23.290 to 60.786]

43. Secondary Outcome: Part 1: AUC From Time Zero (Pre-dose) Extrapolated to Infinite Time (AUC[0-inf]) of GSK3640254
Description: as for outcome 41
Time Frame: Pre-dose and 0.5,1,1.5,2,2.5,3,3.5,4,4.5,5,6,8,12, 24, 48, 72 and 96 hours post-dose
Population: as for outcome 41
Measure: Geometric Mean (95% Confidence Interval); unit: Hour*microgram per milliliter
Arm/Group | Part 1: GSK3640254 1 mg | Part 1: GSK3640254 3 mg | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 30mg | Part 1: GSK3640254 100 mg | Part 1: GSK3640254 200 mg | Part 1: GSK3640254 400 mg | Part 1: GSK3640254 700 mg
Number analyzed (Participants) | 3 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Hour*microgram per milliliter | 0.057 [0.022 to 0.145] | 0.329 [0.232 to 0.467] | 1.227 [1.008 to 1.493] | 2.992 [2.281 to 3.924] | 8.539 [4.511 to 16.165] | 14.952 [9.880 to 22.629] | 42.989 [26.047 to 70.953] | 39.692 [24.094 to 65.389]

44. Secondary Outcome: Part 1: Apparent Terminal Phase Half-life (T1/2) of GSK3640254
Description: Blood samples were collected at indicated time points and PK analysis was performed. PK parameters were determined by non-compartmental methods with Phoenix WinNonlin. Most of the concentrations were below limit of quantification (BLQ) at this dose group this value and/ or %AUC extrapolated was >20% for all participants so this value should be used with caution. Results are presented treatment wise.
Time Frame: Pre-dose and 0.5,1,1.5,2,2.5,3,3.5,4,4.5,5,6,8,12, 24, 48, 72 and 96 hours post-dose
Population: as for outcome 41
Measure: Geometric Mean (95% Confidence Interval); unit: Hour
Arm/Group | Part 1: GSK3640254 1 mg | Part 1: GSK3640254 3 mg | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 30mg | Part 1: GSK3640254 100 mg | Part 1: GSK3640254 200 mg | Part 1: GSK3640254 400 mg | Part 1: GSK3640254 700 mg
Number analyzed (Participants) | 3 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Hour | 7.886 [3.427 to 18.145] | 20.486 [16.450 to 25.514] | 25.332 [20.741 to 30.938] | 21.221 [17.557 to 25.650] | 22.838 [20.268 to 25.734] | 22.620 [18.069 to 28.316] | 23.737 [19.747 to 28.533] | 20.761 [16.171 to 26.654]

45. Secondary Outcome: Part 1: Apparent Oral Clearance (CL/F) of GSK3640254
Description: as for outcome 41
Time Frame: Pre-dose and 0.5,1,1.5,2,2.5,3,3.5,4,4.5,5,6,8,12, 24, 48, 72 and 96 hours post-dose
Population: PK Population. The PK Population include all participants who undergo plasma PK sampling and have evaluable PK parameters estimated during the single dose phase of the study Part 1. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Measure: Geometric Mean (95% Confidence Interval); unit: Liters/hour
Arm/Group | Part 1: GSK3640254 1 mg | Part 1: GSK3640254 3 mg | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 30mg | Part 1: GSK3640254 100 mg | Part 1: GSK3640254 200 mg | Part 1: GSK3640254 400 mg | Part 1: GSK3640254 700 mg
Number analyzed (Participants) | 3 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Liters/hour | 17.685 [6.889 to 45.399] | 9.119 [6.428 to 12.937] | 8.152 [6.697 to 9.922] | 10.027 [7.645 to 13.150] | 11.711 [6.186 to 22.168] | 13.376 [8.838 to 20.244] | 9.305 [5.638 to 15.357] | 17.636 [10.705 to 29.053]

46. Secondary Outcome: Part 1: Maximum Observed Concentration (Cmax), Concentration of GSK3640254 at 24 Hours (C24) and Last Quantifiable Concentration (Clast) of GSK3640254
Description: Blood samples were collected at indicated time points and PK analysis was performed. PK parameters were determined by non-compartmental methods with Phoenix WinNonlin.
Time Frame: Pre-dose and 0.5,1,1.5,2,2.5,3,3.5,4,4.5,5,6,8,12, 24, 48, 72 and 96 hours post-dose
Population: as for outcome 42
Measure: Geometric Mean (95% Confidence Interval); unit: Micrograms per milliliter
Arm/Group | Part 1: GSK3640254 1 mg | Part 1: GSK3640254 3 mg | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 30mg | Part 1: GSK3640254 100 mg | Part 1: GSK3640254 200 mg | Part 1: GSK3640254 400 mg | Part 1: GSK3640254 700 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Micrograms per milliliter
  Cmax | 0.005 [0.004 to 0.006] | 0.014 [0.010 to 0.019] | 0.047 [0.034 to 0.064] | 0.130 [0.104 to 0.162] | 0.372 [0.190 to 0.730] | 0.579 [0.438 to 0.765] | 1.881 [1.150 to 3.077] | 1.724 [1.137 to 2.614]
  C24 | 0.001 [0.000 to 0.005] | 0.005 [0.004 to 0.007] | 0.017 [0.013 to 0.023] | 0.043 [0.031 to 0.062] | 0.126 [0.061 to 0.261] | 0.245 [0.153 to 0.392] | 0.610 [0.356 to 1.046] | 0.579 [0.348 to 0.963]
  Clast | 0.004 [0.003 to 0.005] | 0.005 [0.004 to 0.006] | 0.004 [0.003 to 0.005] | 0.005 [0.004 to 0.008] | 0.014 [0.008 to 0.026] | 0.024 [0.010 to 0.054] | 0.072 [0.043 to 0.120] | 0.054 [0.022 to 0.128]

47. Secondary Outcome: Part 1: Time of Occurrence of Cmax (Tmax), Lag Time (Tlag), and Time to Reach Clast (Tlast) of GSK3640254
Description: as for outcome 41
Time Frame: Pre-dose and 0.5,1,1.5,2,2.5,3,3.5,4,4.5,5,6,8,12, 24, 48, 72 and 96 hours post-dose
Population: as for outcome 42
Measure: Median (Full Range); unit: Hour
Arm/Group | Part 1: GSK3640254 1 mg | Part 1: GSK3640254 3 mg | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 30mg | Part 1: GSK3640254 100 mg | Part 1: GSK3640254 200 mg | Part 1: GSK3640254 400 mg | Part 1: GSK3640254 700 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Hour
  Tmax | 3.500 [2.500 to 6.000] | 4.500 [2.000 to 5.000] | 3.500 [2.500 to 5.000] | 4.000 [2.500 to 5.000] | 3.750 [2.000 to 5.000] | 3.000 [1.983 to 4.000] | 3.250 [2.000 to 6.000] | 3.250 [2.000 to 4.500]
  Tlag | 2.000 [1.500 to 4.500] | 1.250 [0.500 to 3.000] | 0.750 [0.500 to 2.000] | 0.500 [0.500 to 0.517] | 0.750 [0.000 to 1.000] | 0.500 [0.500 to 0.500] | 0.500 [0.000 to 0.500] | 0.500 [0.000 to 0.517]
  Tlast | 6.017 [4.500 to 48.000] | 24.017 [24.000 to 48.017] | 72.008 [72.000 to 96.083] | 96.000 [72.033 to 96.000] | 96.000 [95.317 to 96.017] | 95.667 [95.667 to 96.000] | 95.667 [95.483 to 96.100] | 95.542 [95.250 to 96.000]

48. Secondary Outcome: Part 2: AUC(0-24) of GSK3640254: Day 1
Description: as for outcome 41
Time Frame: Pre-dose and 0.5,1,1.5,2,2.5,3,3.5,4,4.5,5,6,8,12 and 24 hours post-dose on Day 1
Population: PK Population. The PK Population include all participants who undergo plasma PK sampling and have evaluable PK parameters estimated during the repeat dose phase of the study Part 2.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*micrograms per milliliter
Arm/Group | Part 2: GSK3640254 50 mg | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 200 mg + Expansion | Part 2: GSK3640254 320 mg
Number analyzed (Participants) | 6 | 6 | 25 | 7
Hour*micrograms per milliliter | 2.855 (29.621) | 6.801 (22.970) | 8.257 (49.782) | 13.456 (23.743)

49. Secondary Outcome: Part 2: Cmax, C24 of GSK3640254 on Day 1
Description: as for outcome 41
Time Frame: Pre-dose and 0.5,1,1.5,2,2.5,3,3.5,4,4.5,5,6,8,12 hours post-dose on Day 1
Population: as for outcome 48
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Part 2: GSK3640254 50 mg | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 200 mg + Expansion | Part 2: GSK3640254 320 mg
Number analyzed (Participants) | 6 | 6 | 25 | 7
Micrograms per milliliter
  Cmax | 0.215 (24.412) | 0.536 (22.959) | 0.614 (44.354) | 1.044 (29.225)
  C24 | 0.082 (33.583) | 0.207 (22.856) | 0.238 (58.452) | 0.417 (39.681)

50. Secondary Outcome: Part 2: Tmax, Tlag of GSK3640254 on Day 1
Description: Blood samples were collected at indicated timepoints and PK analysis was performed. PK parameters were determined by non-compartmental methods with Phoenix WinNonlin.
Time Frame: Pre-dose and 0.5,1,1.5,2,2.5,3,3.5,4,4.5,5,6,8,12 hours post-dose on Day 1
Population: as for outcome 48
Measure: Median (Full Range); unit: Hour
Arm/Group | Part 2: GSK3640254 50 mg | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 200 mg + Expansion | Part 2: GSK3640254 320 mg
Number analyzed (Participants) | 6 | 6 | 25 | 7
Hour
  Tmax | 3.750 [3.000 to 5.017] | 4.250 [2.000 to 5.000] | 4.000 [1.500 to 5.633] | 4.000 [2.500 to 6.000]
  Tlag | 0.508 [0.500 to 0.550] | 0.500 [0.500 to 0.500] | 0.500 [0.000 to 1.500] | 0.500 [0.000 to 1.000]

51. Secondary Outcome: Part 2: Tmax GSK3640254 on Day 14
Description: as for outcome 41
Time Frame: Pre-dose and 0.5,1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 8, 12, 24, 48, 72 and 96 hours after Day 14 dose
Population: PK Population, The PK Population include all participants who undergo plasma PK sampling and have evaluable PK parameters estimated during the repeat dose phase of the study Part 2. Only those participants with data available at the specified data points were analyzed.
Measure: Median (Full Range); unit: Hour
Arm/Group | Part 2: GSK3640254 50 mg | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 200 mg + Expansion | Part 2: GSK3640254 320 mg
Number analyzed (Participants) | 6 | 6 | 24 | 6
Hour | 3.775 [2.500 to 5.000] | 4.000 [1.500 to 4.500] | 3.750 [1.500 to 5.500] | 4.250 [1.500 to 6.000]

52. Secondary Outcome: Part 2: Cmax of GSK3640254 on Day 14
Description: as for outcome 41
Time Frame: Pre-dose and 0.5,1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 8, 12, 24, 48, 72 and 96 hours after Day 14 dose
Population: as for outcome 51
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Part 2: GSK3640254 50 mg | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 200 mg + Expansion | Part 2: GSK3640254 320 mg
Number analyzed (Participants) | 6 | 6 | 24 | 6
Micrograms per milliliter | 0.414 (31.556) | 1.182 (10.264) | 1.402 (30.839) | 2.156 (20.360)

53. Secondary Outcome: Part 2: AUC From Pre-dose to the End of the Dosing Interval at Steady State (AUC[0-tau]): Day 14
Description: as for outcome 41
Time Frame: Pre-dose and 0.5,1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 8, 12, 24 hours after Day 14 dose
Population: as for outcome 51
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour* micrograms per milliliter
Arm/Group | Part 2: GSK3640254 50 mg | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 200 mg + Expansion | Part 2: GSK3640254 320 mg
Number analyzed (Participants) | 6 | 6 | 24 | 6
hour* micrograms per milliliter | 6.282 (34.010) | 17.506 (13.794) | 21.501 (34.205) | 31.954 (35.380)

54. Secondary Outcome: Part 2: Plasma Trough Concentration (Ctau) of GSK3640254: Day 14
Description: Blood samples were collected at indicated timepoints and PK analysis was performed. PK parameters were determined by non-compartmental methods with Phoenix WinNonlin. The PK parameter name for Part 2 (Day 14) trough concentration was changed using Phoenix WinNonlin 8 from Ct to Ctrough. Day 15 Ctrough values were used for dose proportionality and time to steady-state assessments.
Time Frame: Pre-dose and 0.5,1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 8, 12, 24, 48, 72 and 96 hours after Day 14 dose
Population: PK Population, The PK Population include all participants who undergo plasma PK sampling and have evaluable PK parameters estimated during the repeat dose phase of the study Part 2.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter
Arm/Group | Part 2: GSK3640254 50 mg | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 200 mg + Expansion | Part 2: GSK3640254 320 mg
Number analyzed (Participants) | 6 | 6 | 24 | 6
micrograms per milliliter | 0.186 (35.128) | 0.558 (21.407) | 0.630 (37.814) | 0.980 (41.815)

55. Secondary Outcome: Part 2: T1/2 of GSK3640254: Day 14
Description: as for outcome 41
Time Frame: Pre-dose and 0.5,1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 8, 12, 24, 48, 72 and 96 hours after Day 14 dose
Population: as for outcome 51
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour
Arm/Group | Part 2: GSK3640254 50 mg | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 200 mg + Expansion | Part 2: GSK3640254 320 mg
Number analyzed (Participants) | 6 | 6 | 24 | 6
Hour | 24.847 (5.087) | 28.358 (19.199) | 22.125 (14.515) | 22.350 (12.641)

56. Secondary Outcome: Part 2: CL/F of GSK3640254: Day 14
Description: as for outcome 46
Time Frame: Pre-dose and 0.5,1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 8, 12, 24, 48, 72 and 96 hours after Day 14 dose
Population: as for outcome 51
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour
Arm/Group | Part 2: GSK3640254 50 mg | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 200 mg + Expansion | Part 2: GSK3640254 320 mg
Number analyzed (Participants) | 6 | 6 | 24 | 6
Liter per hour | 7.959 (34.010) | 5.712 (13.794) | 9.302 (34.205) | 10.014 (35.380)

57. Secondary Outcome: Part 1: Dose Proportionality (AUC[0-inf]) Following Single Dose of GSK3640254 on Day 1
Description: Blood samples were collected at indicated time points and PK analysis was performed. Dose proportionality was assessed using the power model. Results are presented treatment wise.
Time Frame: Pre-dose and 0.5,1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 8, 12, 24, 48, 72 and 96 hours post dose
Population: PK Population, The PK Population include all participants who undergo plasma PK sampling and have evaluable PK parameters estimated during the single dose phase of the study Part 1.
Measure: Geometric Mean (95% Confidence Interval); unit: hour*micrograms per mililiter
Arm/Group | Part 1: GSK3640254 1 mg | Part 1: GSK3640254 3 mg | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 30mg | Part 1: GSK3640254 100 mg | Part 1: GSK3640254 200 mg | Part 1: GSK3640254 400 mg | Part 1: GSK3640254 700 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
hour*micrograms per mililiter | 0.057 [0.022 to 0.145] | 0.329 [0.232 to 0.467] | 1.1227 [1.008 to 1.493] | 2.992 [2.281 to 3.924] | 8.539 [4.511 to 16.165] | 14.952 [9.880 to 22.629] | 42.989 [26.047 to 70.953] | 39.692 [24.094 to 65.389]
Statistical Analysis 1: Comparison: Part 1: GSK3640254 1 mg vs Part 1: GSK3640254 3 mg vs Part 1: GSK3640254 10 mg vs Part 1: GSK3640254 30mg vs Part 1: GSK3640254 100 mg vs Part 1: GSK3640254 200 mg vs Part 1: GSK3640254 400 mg vs Part 1: GSK3640254 700 mg; Test type: Other; Power model = 0.9476, 90% CI 2-sided [0.8982 to 0.9971] — The statistical model (power model) is based on the PK parameters (AUC0-inf) from all active doses in Part 1

58. Secondary Outcome: Part 1: Dose Proportionality (AUC0-24) Following Single Dose of GSK3640254 on Day 1
Description: as for outcome 57
Time Frame: Pre-dose and 0.5,1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 8, 12, 24 hours post dose
Population: as for outcome 57
Measure: Geometric Mean (95% Confidence Interval); unit: hour*micrograms per mililiter
Arm/Group | Part 1: GSK3640254 1 mg | Part 1: GSK3640254 3 mg | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 30mg | Part 1: GSK3640254 100 mg | Part 1: GSK3640254 200 mg | Part 1: GSK3640254 400 mg | Part 1: GSK3640254 700 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
hour*micrograms per mililiter | 0.056 [0.030 to 0.103] | 0.171 [0.126 to 0.231] | 0.576 [0.454 to 0.730] | 1.546 [1.178 to 2.028] | 4.177 [2.161 to 8.074] | 7.334 [5.415 to 9.933] | 21.666 [12.599 to 37.259] | 20.743 [13.296 to 32.362]
Statistical Analysis 1: Comparison: Part 1: GSK3640254 1 mg vs Part 1: GSK3640254 3 mg vs Part 1: GSK3640254 10 mg vs Part 1: GSK3640254 30mg vs Part 1: GSK3640254 100 mg vs Part 1: GSK3640254 200 mg vs Part 1: GSK3640254 400 mg vs Part 1: GSK3640254 700 mg; Test type: Other; Power model = 0.9280, 90% CI 2-sided [0.8877 to 0.9683] — The statistical model (power model) is based on the PK parameters (AUC0-24) from all active doses in Part 1

59. Secondary Outcome: Part 1: Dose Proportionality for Cmax Following Single Dose of GSK3640254 on Day 1
Description: as for outcome 57
Time Frame: Pre-dose and 0.5,1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 8, 12, 24, 48, 72 and 96 hours post dose
Population: as for outcome 57
Measure: Geometric Mean (95% Confidence Interval); unit: Micrograms per mililiter
Arm/Group | Part 1: GSK3640254 1 mg | Part 1: GSK3640254 3 mg | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 30mg | Part 1: GSK3640254 100 mg | Part 1: GSK3640254 200 mg | Part 1: GSK3640254 400 mg | Part 1: GSK3640254 700 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Micrograms per mililiter | 0.005 [0.004 to 0.006] | 0.014 [0.010 to 0.019] | 0.047 [0.034 to 0.064] | 0.130 [0.104 to 0.162] | 0.372 [0.190 to 0.730] | 0.579 [0.438 to 0.765] | 1.881 [1.150 to 3.077] | 1.724 [1.137 to 2.614]
Statistical Analysis 1: Comparison: Part 1: GSK3640254 1 mg vs Part 1: GSK3640254 3 mg vs Part 1: GSK3640254 10 mg vs Part 1: GSK3640254 30mg vs Part 1: GSK3640254 100 mg vs Part 1: GSK3640254 200 mg vs Part 1: GSK3640254 400 mg vs Part 1: GSK3640254 700 mg; Test type: Other; Power Model = 0.9352, 90% CI 2-sided [0.8970 to 0.9734] — The statistical model (power model) is based on the PK parameters (Cmax) from all active doses in Part 1

60. Secondary Outcome: Part 2: Dose Proportionality (AUC0-tau) Following Repeated Dose of GSK3640254 on Day 14
Description: as for outcome 57
Time Frame: Pre-dose and 0.5,1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 8, 12, 24, 48, 72 and 96 hours after Day 14 dose
Population: as for outcome 51
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*microgram per milliliter
Arm/Group | Part 2: GSK3640254 50 mg | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 200 mg + Expansion | Part 2: GSK3640254 320 mg
Number analyzed (Participants) | 6 | 6 | 24 | 6
hour*microgram per milliliter | 6.282 (34.010) | 17.506 (13.794) | 21.501 (34.205) | 31.954 (35.380)
Statistical Analysis 1: Comparison: Part 2: GSK3640254 50 mg vs Part 2: GSK3640254 100 mg vs Part 2: GSK3640254 200 mg + Expansion vs Part 2: GSK3640254 320 mg; Test type: Other; Power model = 0.7968, 90% CI 2-sided [0.6424 to 0.9512] — The statistical model (power model) is based on the PK parameters (AUC0-tau) from all active doses in Part 1

61. Secondary Outcome: Part 2: Dose Proportionality (Ctrough) Following Repeated Dose of GSK3640254 on Day 14
Description: as for outcome 57
Time Frame: Pre-dose and 0.5,1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 8, 12, 24, 48, 72 and 96 hours after Day 14 dose
Population: as for outcome 51
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Part 2: GSK3640254 50 mg | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 200 mg + Expansion | Part 2: GSK3640254 320 mg
Number analyzed (Participants) | 6 | 6 | 24 | 6
Micrograms per milliliter | 0.205 (33.414) | 0.593 (16.359) | 0.615 (74.191) | 1.255 (37.220)
Statistical Analysis 1: Comparison: Part 2: GSK3640254 50 mg vs Part 2: GSK3640254 100 mg vs Part 2: GSK3640254 200 mg + Expansion vs Part 2: GSK3640254 320 mg; Test type: Other; Power model = 0.7890, 90% CI 2-sided [0.6149 to 0.9631] — The statistical model (power model) is based on the PK parameters (Ctrough) from all active doses in Part 2

62. Secondary Outcome: Part 2: Dose Proportionality (Cmax) Following Repeated Dose of GSK3640254 on Day 14
Description: as for outcome 57
Time Frame: Pre-dose and 0.5,1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 8, 12, 24, 48, 72 and 96 hours after Day 14 dose
Population: as for outcome 51
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | Part 2: GSK3640254 50 mg | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 200 mg + Expansion | Part 2: GSK3640254 320 mg
Number analyzed (Participants) | 6 | 6 | 24 | 6
Microgram per milliliter | 0.414 (31.556) | 1.182 (10.264) | 1.402 (30.839) | 2.156 (20.360)
Statistical Analysis 1: Comparison: Part 2: GSK3640254 50 mg vs Part 2: GSK3640254 100 mg vs Part 2: GSK3640254 200 mg + Expansion vs Part 2: GSK3640254 320 mg; Test type: Other; Power model = 0.7955, 90% CI 2-sided [0.6562 to 0.9349] — The statistical model (power model) is based on the PK parameters (Cmax) from all active doses in Part 2

63. Secondary Outcome: Part 2: Accumulation Ratio of AUC(0-tau) (R [AUC{0-TAU}]) From Day 1 to Day 14
Description: Blood samples were collected at indicated time points and PK analysis was performed. PK parameters were determined by non-compartmental methods with Phoenix WinNonlin. The accumulation ratio was estimated by calculating the ratio of the geometric least squares (GLS) means of PK parameters between Day 14 and Day 1, and the corresponding 90% CI for each dose. Ratio and 90% confidence interval is presented. Results are presented treatment wise.
Time Frame: Pre-dose and 0.5,1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 8, 12, 24, 48, 72 and 96 hours after Day 14 dose
Population: as for outcome 54
Measure: Number (90% Confidence Interval); unit: Ratio of AUC(0-tau)
Arm/Group | Part 2: GSK3640254 50 mg | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 200 mg + Expansion | Part 2: GSK3640254 320 mg
Number analyzed (Participants) | 6 | 6 | 25 | 7
Ratio of AUC(0-tau) | 2.2005 [1.9116 to 2.5330] | 2.5739 [2.2067 to 3.0022] | 2.6167 [2.3460 to 2.9185] | 2.3634 [1.7579 to 3.1774]

64. Secondary Outcome: Part 2: Accumulation Ratio of Cmax (R [CMAX]) From Day 1 to Day 14
Description: as for outcome 63
Time Frame: Pre-dose and 0.5,1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 8, 12, 24, 48, 72 and 96 hours after Day 14 dose
Population: as for outcome 54
Measure: Number (90% Confidence Interval); unit: Ratio of Cmax
Arm/Group | Part 2: GSK3640254 50 mg | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 200 mg + Expansion | Part 2: GSK3640254 320 mg
Number analyzed (Participants) | 6 | 6 | 25 | 7
Ratio of Cmax | 1.9276 [1.6283 to 2.2818] | 2.2069 [1.8360 to 2.6528] | 2.2994 [2.0872 to 2.5331] | 2.0650 [1.6064 to 2.6545]

65. Secondary Outcome: Part 2: Accumulation Ratio of C(Tau) (R[CTAU]) From Day 2 to Day 15
Description: Blood samples were collected at indicated time points and PK analysis was performed. PK parameters were determined by non-compartmental methods with Phoenix WinNonlin. The accumulation ratio was estimated by calculating the ratio of the geometric least squares (GLS) means of PK parameters between Day 15 and Day 2, and the corresponding 90% CI for each dose. Ratio and 90% confidence interval is presented. Results are presented treatment wise.
Time Frame: Pre-dose and 0.5,1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 8, 12, 24, 48, 72 and 96 hours after Day 15 dose
Population: as for outcome 54
Measure: Number (90% Confidence Interval); unit: Ratio of Ctau
Arm/Group | Part 2: GSK3640254 50 mg | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 200 mg + Expansion | Part 2: GSK3640254 320 mg
Number analyzed (Participants) | 6 | 6 | 25 | 7
Ratio of Ctau | 2.1408 [1.9402 to 2.3621] | 2.5847 [2.1437 to 3.1165] | 2.5335 [2.2133 to 2.9001] | 2.1666 [1.4908 to 3.1488]

66. Secondary Outcome: Part 2: Pre-dose Concentration of GSK3640254 on Day 2 to Day 14
Description: as for outcome 41
Time Frame: Pre-dose on Days 2,3,4,6,8,10,12 and 14
Population: as for outcome 48
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter
Arm/Group | Part 2: GSK3640254 50 mg | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 200 mg + Expansion | Part 2: GSK3640254 320 mg
Number analyzed (Participants) | 6 | 6 | 25 | 7
Nanogram per milliliter
  Day 2 Predose | 90.20 (25.312) | 221.55 (55.722) | 283.37 (137.243) | 476.58 (197.909)
  Day 3 Predose | 155.93 (41.869) | 449.82 (68.287) | 517.96 (239.825) | 753.02 (174.186)
  Day 4 Predose | 196.25 (55.807) | 524.87 (120.723) | 667.45 (295.479) | 926.40 (235.884)
  Day 6 Predose | 214.64 (75.891) | 550.48 (125.873) | 701.98 (349.091) | 969.06 (225.600)
  Day 8 Predose | 230.50 (77.819) | 595.26 (151.167) | 712.79 (342.941) | 936.45 (278.866)
  Day 10 Predose | 218.97 (74.858) | 604.52 (137.121) | 802.81 (272.000) | 1051.91 (375.261)
  Day 12 predose | 221.10 (75.744) | 628.86 (114.448) | 726.13 (300.263) | 1182.80 (354.948)
  Day 14 predose | 214.16 (66.980) | 599.45 (97.262) | 706.76 (299.450) | 1324.29 (470.703)

67. Secondary Outcome: Part 2: Dose Proportionality (Cmax) Following Repeated Dose of GSK3640254 at Day 1
Description: as for outcome 57
Time Frame: Pre-dose and 0.5,1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 8, 12, 24, 48, 72 and 96 hours post dose
Population: as for outcome 51
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | Part 2: GSK3640254 50 mg | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 200 mg + Expansion | Part 2: GSK3640254 320 mg
Number analyzed (Participants) | 6 | 6 | 25 | 7
Microgram per milliliter | 0.215 (24.412) | 0.536 (22.959) | 0.614 (44.354) | 1.044 (29.225)
Statistical Analysis 1: Comparison: Part 2: GSK3640254 50 mg vs Part 2: GSK3640254 100 mg vs Part 2: GSK3640254 200 mg + Expansion vs Part 2: GSK3640254 320 mg; Test type: Other; Power model = 0.7370, 90% CI 2-sided [0.5649 to 0.9091] — The statistical model (power model) is based on the PK parameters (Cmax) from all active doses in Part 2

68. Secondary Outcome: Part 2: Dose Proportionality (AUC0-24) Following Repeated Dose of GSK3640254 at Day 1
Description: as for outcome 57
Time Frame: Pre-dose and 0.5,1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 8, 12, 24, 48, 72 and 96 hours post dose
Population: as for outcome 51
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*micrograms per mililiter
Arm/Group | Part 2: GSK3640254 50 mg | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 200 mg + Expansion | Part 2: GSK3640254 320 mg
Number analyzed (Participants) | 6 | 6 | 25 | 7
hour*micrograms per mililiter | 2.855 (29.621) | 6.801 (22.970) | 8.257 (49.782) | 13.456 (23.743)
Statistical Analysis 1: Comparison: Part 2: GSK3640254 50 mg vs Part 2: GSK3640254 100 mg vs Part 2: GSK3640254 200 mg + Expansion vs Part 2: GSK3640254 320 mg; Test type: Other; Power model = 0.7397, 90% CI 2-sided [0.5576 to 0.9218] — The statistical model (power model) is based on the PK parameters (AUC0-24) from all active doses in Part 2

ADVERSE EVENTS:
Time Frame: On-treatment and post-treatment non-serious adverse events and serious adverse events were collected up to Day 15 for Part 1 and Day 28 for Part 2 of the study.
Description: Safety Population was used to collect the adverse events
Groups:
- Part 1:GSK3640254 1 mg: Participants received single dose of GSK3640254 1 mg following a moderate fat meal on Day 1
- Part 1:GSK3640254 3 mg: Participants received single dose of GSK3640254 3 mg following a moderate fat meal on Day 1
- Part 1:GSK3640254 10 mg: Participants received single dose of GSK3640254 10 mg following a moderate fat meal on Day 1
- Part 1:GSK3640254 30 mg: Participants received single dose of GSK3640254 30 mg following a moderate fat meal on Day 1
- Part 1:GSK3640254 100 mg: Participants received single dose of GSK3640254 100 mg following a moderate fat meal on Day 1
- Part 1:GSK3640254 200 mg: Participants received single dose of GSK3640254 200 mg following a moderate fat meal on Day 1
- Part 1:GSK3640254 400 mg: Participants received single dose of GSK3640254 400 mg following a moderate fat meal on Day 1
- Part 1:GSK3640254 700 mg: Participants received single dose of GSK3640254 700 mg following a moderate fat meal on Day 1
- Part 2: Repeated Dose GSK3640254 200mg +Expansion: Participants received repeated dose of GSK3640254 200 mg once daily up to 14 days
Arm/Group | Part 1:GSK3640254 1 mg | Part 1:GSK3640254 3 mg | Part 1:GSK3640254 10 mg | Part 1:GSK3640254 30 mg | Part 1:GSK3640254 100 mg | Part 1:GSK3640254 200 mg | Part 1:GSK3640254 400 mg | Part 1:GSK3640254 700 mg | Part 1: Single Dose Placebo | Part 2: Repeated Dose GSK3640254 50 mg | Part 2: Repeated Dose GSK3640254 100 mg | Part 2: Repeated Dose GSK3640254 200mg +Expansion | Part 2: Repeated Dose GSK3640254 320 mg | Part 2: Repeated Dose Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/16 | 0/6 | 0/6 | 0/25 | 0/7 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/16 | 0/6 | 0/6 | 0/25 | 0/7 | 0/14
Other Adverse Events (participants affected / at risk) | 3/6 | 2/6 | 4/6 | 3/6 | 3/6 | 4/6 | 4/6 | 1/6 | 7/16 | 4/6 | 5/6 | 19/25 | 6/7 | 10/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1:GSK3640254 1 mg (N=6) | Part 1:GSK3640254 3 mg (N=6) | Part 1:GSK3640254 10 mg (N=6) | Part 1:GSK3640254 30 mg (N=6) | Part 1:GSK3640254 100 mg (N=6) | Part 1:GSK3640254 200 mg (N=6) | Part 1:GSK3640254 400 mg (N=6) | Part 1:GSK3640254 700 mg (N=6) | Part 1: Single Dose Placebo (N=16) | Part 2: Repeated Dose GSK3640254 50 mg (N=6) | Part 2: Repeated Dose GSK3640254 100 mg (N=6) | Part 2: Repeated Dose GSK3640254 200mg +Expansion (N=25) | Part 2: Repeated Dose GSK3640254 320 mg (N=7) | Part 2: Repeated Dose Placebo (N=14)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (2) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 3 (5) | 2 (2) | 6 (6)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Faeces pale (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Faeces soft (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 7 (7) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Face injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nightmare (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site bruise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Disturbance in attention (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glossodynia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lip dry (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Catheter site bruise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mass (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eczema nummular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bicuspid aortic valve (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-05-17): https://cdn.clinicaltrials.gov/large-docs/43/NCT03231943/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-08): https://cdn.clinicaltrials.gov/large-docs/43/NCT03231943/SAP_001.pdf